## STATISTICAL ANALYSIS PLAN

Phase 1b Dose-Finding Study of Niraparib, TSR-022, Bevacizumab, and Platinum-Based Doublet Chemotherapy in Combination With TSR-042 in Patients With Advanced or Metastatic Cancer

**Protocol Number:** 3000-01-002

**Protocol Version and Date:** v3.0 August 15, 2018

v2.0 November 15, 2017 (Amendment 1)

v1.0 July 07, 2017 (Original)

**Study Drug Name:** Niraparib, TSR-042, TSR-022, carboplatin-paclitaxel,

carboplatin-pemetrexed, carboplatin-nab-paclitaxel, and

bevacizumab

**Phase:** Phase 1b

**Sponsor:** TESARO, Inc.

Analysis Plan Date: 18 SEP, 2020

**Analysis Plan Version:** Version 1.0

#### **Confidentiality Statement**

All information contained in this document is privileged and confidential to TESARO. Any distribution, copying, or disclosure is strictly prohibited without prior written approval by TESARO.

#### **SPONSOR SIGNATURE PAGE**

**Protocol Title:** Phase 1b Dose-Finding Study of Niraparib, TSR-022, Bevacizumab,

and Platinum-Based Doublet Chemotherapy in Combination With

TSR-042 in Patients With Advanced or Metastatic Cancer

**Protocol Number:** 3000-01-002

**Sponsor:** TESARO, Inc.

1000 Winter Street Waltham MA 02451

By signing this document, I acknowledge that I have read the document and approve of the planned statistical analyses described herein. I agree that the planned statistical analyses are appropriate for this study, are in accordance with the study objectives, and are consistent with the statistical methodology described in the protocol, clinical development plan, and all applicable regulatory guidance and guidelines.

| • | | 4 | L | _ | |
|---|---|---|---|---|---|
| А | ш | т | n | O | r |

PPD Signature:

Lead Statistician Date: 18-SE

**Biostatistics India**,

**GSK** 

Approver:

**PPD**, **PhD** Signature:

Statistician Date: 18-SEP-2020

TESARO, Inc.

PPD , MD Signature:

Medical Director Date: 18-SEP-2020

TESARO, Inc.

## TESARO Inc.

| ٦ | $\Gamma \Delta$ | I | 3 | r 1 | F | $\cap$ | F | $\mathbf{C}$ | $\cap$ | N | П | П | 71 | V. | Г٦ | Γ9 | 3 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | ľ | ١ | Э. | | С. | U | Г | v | ( ) | 1 | | | D. | 1 | | l i | 7 |

| SPO | NSOR SI | GNATURE PAGE | 2 |
|------|----------|---------------------------------|------|
| LIST | Γ OF TAE | BLES INCLUDED IN THE TEXT | 6 |
| LIST | Γ OF FIG | URES INCLUDED IN THE TEXT | 7 |
| ABE | BREVIAT | TONS | 8 |
| 1 | INTROI | DUCTION | . 11 |
| 2 | STUDY | DESIGN OVERVIEW | . 12 |
| 2.1 | Overa | ll Study Design | 12 |
| 2.2 | Sampl | e Size | 17 |
| 2.3 | Rando | mization and Blinding | 17 |
| 3 | STUDY | OBJECTIVES | . 18 |
| 3.1 | Prima | y Objectives | 18 |
| | 3.1.1 | Primary Objectives for Part A | . 18 |
| | 3.1.2 | Primary Objectives for Part B | . 18 |
| | 3.1.3 | Primary Objectives for Part C | . 18 |
| | 3.1.4 | Primary Objectives for Part D. | . 18 |
| | 3.1.5 | Primary Objectives for Part E | . 18 |
| | 3.1.6 | Primary Objectives for Part F | . 19 |
| | 3.1.7 | Primary Objectives for Part G | . 19 |
| | 3.1.8 | Primary Objectives for Part H | . 19 |
| | 3.1.9 | Primary Objectives for Part I | . 19 |
| 3.2 | Secon | dary Objectives | 20 |
| | 3.2.1 | Secondary Objectives for Part A | 20 |
| | 3.2.2 | Secondary Objectives for Part B | 20 |
| | 3.2.3 | Secondary Objectives for Part C | 20 |
| | 3.2.4 | Secondary Objectives for Part D | 20 |
| | 3.2.5 | Secondary Objectives for Part E | 20 |
| | 3.2.6 | Secondary Objectives for Part F | 21 |
| | 3.2.7 | Secondary Objectives for Part G | 21 |
| | 3.2.8 | Secondary Objectives for Part H | 21 |
| | 3.2.9 | Secondary Objectives for Part I | 21 |
| 3.3 | Explo | ratory Objectives | 22 |

| | 3.3.1 | Exploratory Objectives for Part A | 22 |
|---|---|---|---|
| | 3.3.2 | Exploratory Objectives for Part B | 22 |
| | 3.3.3 | Exploratory Objectives for Part C | 22 |
| | 3.3.4 | Exploratory Objectives for Part D | 22 |
| | 3.3.5 | Exploratory Objectives for Part E | 22 |
| | 3.3.6 | Exploratory Objectives for Part F | 23 |
| | 3.3.7 | Exploratory Objectives for Part G | 23 |
| | 3.3.8 | Exploratory Objectives for Part H | 23 |
| | 3.3.9 | Exploratory Objectives for Part I | 23 |
| 4 | STUDY | ENDPOINTS AND EVALUATIONS | 24 |
| 4.1 | Safety | Endpoints and Evaluations | 24 |
| 4.2 | Effica | cy Endpoints and Evaluations | 24 |
| 4.3 | Pharm | acokinetics Endpoints and Evaluations | 24 |
| 4.4 | Immu | nogenicity Endpoints and Evaluations | 25 |
| 4.5 | Bioma | rker Evaluations | 25 |
| 4.6 | Other | Evaluations | 26 |
| 5 | DEFINI | TIONS AND CONVENTIONS FOR DATA HANDLING | 27 |
| 5.1 | Defini | tion of Baseline | 27 |
| 5.2 | First I | Pose Date of Study Treatment | 27 |
| 5.3 | Defini | tion of Treatment Period | 27 |
| 5.4 | Defini | tion of Relative Study Days | 27 |
| 5.5 | Analy | sis Visit Window | 27 |
| 5.6 | Safety | Data Handling | 28 |
| | 5.6.1 | Handling of Unscheduled ECG Measurements | 28 |
| | 5.6.2 | Handling of Partial Dates for AEs | 28 |
| | 5.6.3 | Handling of Partial Dates for Medications | 28 |
| | 5.6.4 | Handling of Partial Dates for Disease History | 29 |
| | 5.6.5 | Handling of Partial Dates for Progression in Prior Treatment | 29 |
| 6 | PLANN | ED ANALYSIS | 30 |
| 6.1 | Chang | ges from Planned Analyses in the Protocol | 30 |
| 6.2 | Interir | n Analysis | 30 |
| 6.3 | Final . | Analyses and Reporting | 30 |

| 7 | ANAL | YSIS POPULATIONS AND APPLICATIONS | 31 |
|-----|-------|-----------------------------------------------------|----|
| 7.1 | All P | atients Population | 31 |
| 7.2 | Safet | y Population | 31 |
| 7.3 | Appl | ication of Analysis Populations | 31 |
| 8 | STATI | STICAL CONSIDERATIONS | 33 |
| 8.1 | Gene | ral Statistical Procedures | 33 |
| 8.2 | Enro | llment and Disposition | 34 |
| | 8.2.1 | Patients Enrollment | 34 |
| | 8.2.2 | Patients Disposition | 34 |
| | 8.2.3 | Protocol Deviations | 34 |
| 8.3 | Dem | ographics and Baseline Characteristics | 35 |
| | 8.3.1 | Demographics, Baseline and Disease Characteristics | 35 |
| | 8.3.2 | Medical History | 35 |
| | 8.3.3 | Prior Anticancer Treatment | 36 |
| | 8.3.4 | Prior and Concomitant Medication/Procedures | 36 |
| | 8.3.5 | HBsAg and HCV Ribonucleic Acid Testing at Baseline | 37 |
| 8.4 | Safet | y Analysis | 37 |
| | 8.4.1 | Adverse Events | 37 |
| | 8.4.2 | Study Drug Exposure | 39 |
| | 8.4.3 | Clinical Laboratory Tests | 45 |
| | 8.4.4 | Vital Signs | 46 |
| | 8.4.5 | Physical Examination Findings | 46 |
| | 8.4.6 | ECOG performance status | 46 |
| | 8.4.7 | Electrocardiogram (ECG) | 46 |
| 8.5 | Effic | acy Analysis | 47 |
| | 8.5.1 | Best Overall Response when confirmation is required | 47 |
| | 8.5.2 | Objective Response Rate | 49 |
| | 8.5.3 | Duration of Response | 49 |
| | 8.5.4 | Disease Control Rate | 50 |
| | 8.5.5 | Progression Free Survival | 50 |
| 9 | APPEN | NDIX: Immune Related Adverse Events | 52 |
| 10 | PLAN | NED STATISTICAL TABLES, FIGURES AND LISTINGS | 56 |

# TESARO Inc. Protocol No: 3000-01-002

# LIST OF TABLES INCLUDED IN THE TEXT

| Table 1: PK Parameters | 25 |
|-----------------------------------------------------------|----|
| Table 2: Application of Populations on Tables and Figures | |
| Table 3: Extent of Study Drug Exposure | |
| Table 4: Censoring Rules Used for DOR Analysis | |
| Table 5: Censoring Rules Used for PFS Analysis | |

| TESARO Inc. | Statistical Analysis Plan |
|-----------------------------------|---------------------------|
| Protocol No: 3000-01-002 | <b>Dated:18SEP2020</b> |
| LIST OF FIGURES INCLUDED IN THE T | EXT |

| Figure 1: Study Design | . 14 |
|------------------------|------|
|------------------------|------|

TESARO Inc.
Protocol No: 3000-01-002

# **ABBREVIATIONS**

| Abbreviation | Explanation |
|------------------|---------------------------------------------------------|
| ADA | Anti-Drug Antibody |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area Under the Plasma or Serum Concentration-Time Curve |
| BE | Biomarker Evaluation |
| BLQQ | Below the Limit of Quantitation |
| BMI | Body Mass Index |
| BOR | Best Overall Response |
| BRCA | Breast Cancer Gene |
| BRCAmut | BRCA Mutation |
| CBC | Complete Blood Count |
| CI | Confidence Interval |
| CL | Clearance After Intravenous Administration |
| CL/F | Clearance After Oral Administration |
| C <sub>max</sub> | Maximum Observed Plasma or Serum Concentration |
| C <sub>min</sub> | Minimum Observed Plasma or Serum Concentration |
| CR | Complete Response |
| CRF | Case Report Form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| Ctrough | Trough plasma concentration |
| CV | Coefficient of Variation |
| DCR | Disease Control Rate |
| DLT | Dose Limiting Toxicity |
| DOR | Duration of Response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronical Case Report Form |
| ЕОТ | End of Treatment |

| FFPE | Formalin-Fixed Paraffin Embedded |
|-------------|-------------------------------------------------------------|
| FT3 | Free Triiodothyronine |
| FT4 | Free Thyroxine |
| gBRCAmut | Germline BRCA Mutation |
| HBsAg | Hepatitis B Surface Antigen |
| HCV | Hepatitis C Virus |
| ID | Identification |
| KM | Kaplan-Meier |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min | Minimum |
| NE | Not Evaluated |
| NSCLC | Non-Small Cell Lung Cancer |
| ORR | Objective Response Rate |
| PD | Progressive Disease |
| PD-L1 | Programmed Death-Ligand 1 |
| PDV | Protocol Deviation |
| PFS | Progression-Free Survival |
| PK | Pharmacokinetic(S) |
| РО | Orally |
| PR | Partial Response |
| PT | Preferred Term |
| Q3W | Every 3 Weeks |
| Q6W | Every 6 Weeks |
| QTcF | Corrected QT Interval Calculated Using Fridericia's Formula |
| RECIST v1.1 | Response Evaluation Criteria in Solid Tumors Version 1.1 |
| Rel | Relative Study |
| RP2D | Recommended Phase 2 Dose |
| SAE | Serious Adverse Event |
| SD | Stable Disease |
| SOC | System Organ Class |
| STD | Standard Deviation |

TESARO Inc.

| Т3 | Triiodothyronine |
|--------|---------------------------------------------------------|
| TEAE | Treatment-Emergent Adverse Event |
| TSH | Thyroid-Stimulating Hormone |
| uBOR | Unconfirmed Best Overall Response |
| uDCR | Unconfirmed Disease Control Rate |
| uDOR | Unconfirmed Duration of Response |
| uORR | Unconfirmed Objective Response Rate |
| Vz | Volume of Distribution After Intravenous Administration |
| Vz/F | Volume of Distribution After Oral Administration |
| WHO | World Health Organization |
| WHO-DD | World Health Organization Drug Dictionary |

#### 1 INTRODUCTION

This statistical analysis plan is designed to outline the statistical methods in evaluating the safety and preliminary efficacy of niraparib or niraparib/bevacizumab in combination with TSR-042 treatment and confirming the safety and tolerability of carboplatin-paclitaxel, carboplatin-paclitaxel/bevacizumab, carboplatin-pemetrexed and TSR-022/carboplatin-pemetrexed in combination with TSR-042 treatment in patients with advanced or metastatic cancer for TESARO study protocol 3000-01-002. Parts G, H and I specified in the study design were not initiated and therefore not included in this SAP.

This document has been prepared based on Study Protocol version 3.0 dated 15 August 2018 and Case Report Form (CRF) dated 12 JUN 2020. Details will be described in this analysis plan to ensure that the data listings, summary tables and figures which will be produced, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives.

#### 2 STUDY DESIGN OVERVIEW

#### 2.1 Overall Study Design

This is a multicenter, open-label, 9-part Phase 1b study evaluating the safety and preliminary efficacy of niraparib or niraparib/bevacizumab in combination with TSR-042 treatment and confirming the safety and tolerability of carboplatin-paclitaxel, carboplatin-paclitaxel, bevacizumab, carboplatin-pemetrexed, TSR-022/carboplatin-paclitaxel, and TSR-022/carboplatin-paclitaxel in combination with TSR-042 treatment in patients with advanced or metastatic cancer.

- Part A (dose finding—TSR-042 and niraparib combination treatment): all comers, defined as patients with previously treated advanced or metastatic cancer
- Part B (safety and tolerability evaluation—TSR-042 and carboplatin-paclitaxel combination treatment): patients with advanced or metastatic cancer for which treatment with carboplatin and paclitaxel is indicated (e.g., including, but not limited to, non-small cell lung cancer [NSCLC], ovarian cancer, and cervical cancer)
- Part C (dose finding—TSR-042, niraparib and bevacizumab combination treatment): all comers, defined as patients with previously treated advanced or metastatic cancer
- Part D (safety and tolerability evaluation—TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment): in patients in whom carboplatin-paclitaxel and bevacizumab is considered a reasonable therapy
- Part E (safety and tolerability evaluation—TSR-042 and carboplatin-pemetrexed combination treatment): as first-line treatment in patients with advanced or metastatic non-squamous NSCLC
- Part F (safety and tolerability evaluation—TSR-042, TSR-022, and carboplatinpemetrexed combination treatment): as first-line treatment in patients with advanced or metastatic non-squamous NSCLC
- Part G (safety and tolerability evaluation—TSR-042 and carboplatin—nab-paclitaxel combination treatment): as first-line treatment in patients with advanced or metastatic NSCLC
- Part H (safety and tolerability evaluation—TSR-042, TSR-022, and carboplatin-nabpaclitaxel combination treatment): as first-line treatment in patients with advanced or metastatic NSCLC
- Part I (safety and tolerability evaluation—TSR-042, TSR-022, and carboplatin-paclitaxel combination treatment): as first-line treatment in patients with advanced or metastatic NSCLC

Don't A will be a dose finding evaluation conducted in all compare (12 to 24 notions) to determine

Part A will be a dose-finding evaluation conducted in all comers (12 to 24 patients) to determine the RP2D of niraparib in combination with TSR-042.

Part B will evaluate the safety and tolerability of TSR-042 and carboplatin-paclitaxel combination treatment in approximately 12 patients with advanced or metastatic cancer for which carboplatin-paclitaxel is indicated.

Part C will be a dose-finding evaluation conducted in all comers (6 to 24 patients) to determine the RP2D of niraparib and bevacizumab in combination with TSR-042.

Part D will evaluate the safety and tolerability of TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment in 6 to 12 patients in whom carboplatin-paclitaxel and bevacizumab combination treatment is considered a reasonable therapy.

Part E will evaluate the safety and tolerability of TSR-042 and carboplatin-pemetrexed combination treatment as first-line treatment in 6 to 12 patients with advanced or metastatic non-squamous NSCLC.

Part F will evaluate the safety and tolerability of TSR-042, TSR-022, and carboplatin-pemetrexed combination treatment as first-line treatment in 6 to 24 patients with advanced or metastatic non-squamous NSCLC.

Part G will evaluate the safety and tolerability of TSR-042 and carboplatin – nab-paclitaxel combination treatment as first-line treatment in 6 to 12 patients with advanced or metastatic NSCLC.

Part H will evaluate the safety and tolerability of TSR-042, TSR-022, and carboplatin – nab-paclitaxel combination treatment as first-line treatment in 6 to 24 patients with advanced or metastatic NSCLC.

Part I will evaluate the safety and tolerability of TSR-042, TSR-022, and carboplatin-paclitaxel combination treatment as first-line treatment in 6 to 24 patients with advanced or metastatic NSCLC

Enrollment of patients into Parts A, B, D, E, G, and I will occur concurrently. Part C will be initiated after dose level 1 (niraparib 200 mg) in Part A is determined to be safe. Part F will be initiated after TSR-042 and carboplatin-pemetrexed combination treatment in Part E is determined to be safe. Part H will be initiated after TSR-042 and carboplatin-nab-paclitaxel combination treatment in Part G is determined to be safe.

The study design of nine parts is presented graphically in Figure 1. The study schedule of events for each part are be found in Table 17-34 in the protocol.

TESARO Inc.

Protocol No: 3000-01-002 Dated:18SEP2020

Figure 1: Study Design

Part A (6 + 6): TSR-042 + Niraparib Dose Finding



#### Part B: TSR-042 + Carboplatin-Paclitaxel Safety and Tolerability



#### Part C (6 + 6): TSR-042 + Niraparib + Bevacizumab Dose Finding



#### Part D (6 + 6): TSR-042 + Carboplatin-Paclitaxel + Bevacizumab Safety and Tolerability




#### Part E: TSR-042 + Pemetrexed + Carboplatin Safety and Tolerability



#### Part F: TSR-042 + TSR-022 + Pemetrexed + Carboplatin Safety and Tolerability



#### Part G: TSR-042 + Carboplatin + Nab-Paclitaxel Safety and Tolerability



#### Part H: TSR-042 + TSR-022 + Carboplatin + Nab-Paclitaxel Safety and Tolerability



#### Part I: TSR-042 + TSR-022 + Carboplatin-Paclitaxel Safety and Tolerability



Abbreviations: AE = adverse event; AUC = area under the plasma or serum concentration-time curve; D1 = Day 1; D21 = Day 21; DLT = dose-limiting toxicity; PK = pharmacokinetics; Q1W = every week; Q3W = every 3 weeks; Q6W = every 6 weeks; RP2D = recommended Phase 2 dose.

- In addition to receiving niraparib (Part A), carboplatin-paclitaxel (Part B), niraparib and bevacizumab (Part C), carboplatin-paclitaxel and bevacizumab (Part D), carboplatin-pemetrexed (Part E), carboplatin-pemetrexed and TSR-022 (Part F), carboplatin-nab-paclitaxel (Part G), TSR-022 and carboplatin-nab-paclitaxel (Part H), and TSR-022 and carboplatin-paclitaxel (Part I) at the specified regimen, all patients will be administered TSR-042 at 500 mg on Day 1 of every cycle (Q3W) for 4 cycles. Beginning on Day 1 of Cycle 5, TSR-042 will be administered to patients in Parts A, B, C, and D at 1,000 mg on Day 1 of every other cycle (Q6W) until the patient discontinues study treatment. Patients in Parts E, F, G, H, and I will continue to receive 500 mg on Day 1 of every cycle (Q3W) throughout the study.
- b The RP2D for TSR-042 and niraparib combination treatment (Part A); TSR-042 and carboplatin-paclitaxel combination treatment (Part B); TSR-042, niraparib, and bevacizumab combination treatment (Part C); TSR-042, carboplatin-paclitaxel, and bevacizumab combination treatment (Part D); TSR-042 and carboplatin-pemetrexed (Part E); TSR-042, carboplatin-pemetrexed, and TSR-022 (Part F); TSR-042 and carboplatin-nab-paclitaxel (Part G); TSR-042, TSR-022, and carboplatin-

nab-paclitaxel (Part H); and TSR-042, TSR-022, and carboplatinpaclitaxel (Part I) will be determined or confirmed based on an evaluation of multiple endpoints, which may include the DLT rate in first and subsequent cycles of combination treatment, the rate of dose modifications for non-DLT AEs, the ability to manage toxicities, PK, niraparib dose intensity, and signs of clinical efficacy.

- c 12 to 24 patients will be enrolled in Part A to determine the RP2D for TSR-042 and niraparib combination treatment.
- d Initially, dose level 1 in Part C will enroll 6 to 12 patients to determine the RP2D for TSR-042, niraparib, and bevacizumab combination treatment. Dose level 2 is optional.
- e 900 mg of TSR-022 is the highest dose tested in dose escalation in combination with TSR-042 that provides maximal pharmacodynamic effect; this dose may be lowered to dose level -1 (300 mg) if needed. Based on available safety information, the Sponsor may decide to test additional dose levels.

## 2.2 Sample Size

- Part A: approximately 12 to 24 patients will be enrolled.
- Part B: approximately 12 patients will be enrolled.
- Part C: approximately 6 to 24 patients may be enrolled.
- Part D: approximately 6 to 12 patients will be enrolled.
- Part E: approximately 6 to 12 patients will be enrolled.
- Part F: approximately 6 to 24 patients will be enrolled.
- Part G: approximately 6 to 12 patients will be enrolled.
- Part H: approximately 6 to 24 patients will be enrolled.
- Part I: approximately 6 to 24 patients will be enrolled.

## 2.3 Randomization and Blinding

This is an open-label Phase 1b study. Patients will not be randomized to study treatment.

#### 3 STUDY OBJECTIVES

## 3.1 Primary Objectives

## 3.1.1 Primary Objectives for Part A

- To evaluate DLTs of TSR-042 and niraparib combination treatment during the first cycle of treatment in patients with advanced or metastatic cancer and to establish a RP2D
- To evaluate the safety and tolerability of TSR-042 and niraparib combination treatment

## 3.1.2 Primary Objectives for Part B

- To evaluate DLTs of TSR-042 and carboplatin-paclitaxel combination treatment during the first cycle of treatment in patients with advanced or metastatic cancer and to confirm an RP2D
- To evaluate the safety and tolerability of TSR-042 and carboplatin-paclitaxel combination treatment

## 3.1.3 Primary Objectives for Part C

- To evaluate DLTs of TSR-042, niraparib, and bevacizumab combination treatment during the first cycle of treatment in patients with advanced or metastatic cancer and to establish an RP2D
- To evaluate the safety and tolerability of TSR-042, niraparib, and bevacizumab combination treatment

#### 3.1.4 Primary Objectives for Part D

- To evaluate DLTs of TSR-042, carboplatin-paclitaxel, and bevacizumab combination treatment during the first cycle of treatment in patients in whom carboplatin-paclitaxel and bevacizumab combination treatment is a reasonable therapy, and to confirm an RP2D
- To evaluate the safety and tolerability of TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

## 3.1.5 Primary Objectives for Part E

- To evaluate DLTs of TSR-042 and carboplatin-pemetrexed combination treatment during the first cycle of treatment, as first-line treatment in patients with advanced or metastatic non-squamous NSCLC, and to confirm an RP2D
- To evaluate the safety and tolerability of TSR-042 and carboplatin-pemetrexed combination treatment

#### 3.1.6 Primary Objectives for Part F

• To evaluate DLTs of TSR-042, TSR-022, and carboplatin-pemetrexed combination treatment during the first cycle of treatment, as first-line treatment in patients with advanced or metastatic non-squamous NSCLC, and to confirm an RP2D

• To evaluate the safety and tolerability of TSR-042, TSR-022, and carboplatin-pemetrexed combination treatment

#### 3.1.7 Primary Objectives for Part G

- To evaluate DLTs of TSR-042 and carboplatin nab-paclitaxel combination treatment during the first cycle of treatment, as first-line treatment in patients with advanced or metastatic NSCLC, and to confirm an RP2D
- To evaluate the safety and tolerability of TSR-042 and carboplatin nab-paclitaxel combination treatment

## 3.1.8 Primary Objectives for Part H

- To evaluate DLTs of TSR-042, TSR-022, and carboplatin nab-paclitaxel combination treatment during the first cycle of treatment, as first-line treatment in patients with advanced or metastatic NSCLC, and to confirm an RP2D
- To evaluate the safety and tolerability of TSR-042, TSR-022, and carboplatin nab-paclitaxel combination treatment

#### 3.1.9 Primary Objectives for Part I

- To evaluate DLTs of TSR-042, TSR-022, and carboplatin-paclitaxel combination treatment during the first cycle of treatment, as first-line treatment in patients with advanced or metastatic NSCLC, and to confirm an RP2D
- To evaluate the safety and tolerability of TSR-042, TSR-022, and carboplatinpaclitaxel combination treatment

#### 3.2 Secondary Objectives

## 3.2.1 Secondary Objectives for Part A

• To evaluate measures of clinical benefit as assessed by the Investigators, including objective response rate (ORR), duration of response (DOR), disease control rate (DCR), and PFS by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)

- To evaluate the PK of niraparib, its major metabolite M1, and TSR-042 during TSR-042 and niraparib combination treatment
- To evaluate ADAs of TSR-042 during TSR-042 and niraparib combination treatment

#### 3.2.2 Secondary Objectives for Part B

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of TSR-042 during TSR-042 and carboplatin-paclitaxel combination treatment
- To evaluate ADAs of TSR-042 during TSR-042 and carboplatin-paclitaxel combination treatment

#### 3.2.3 Secondary Objectives for Part C

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of niraparib, its major metabolite M1, and TSR-042 during TSR-042, niraparib and bevacizumab combination treatment
- To evaluate ADAs of TSR-042 during TSR-042, niraparib and bevacizumab combination treatment

#### 3.2.4 Secondary Objectives for Part D

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of TSR-042 during TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment
- To evaluate ADAs of TSR-042 during TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

#### 3.2.5 Secondary Objectives for Part E

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of TSR-042 during TSR-042 and carboplatin-pemetrexed combination treatment

 To evaluate ADAs of TSR-042 during TSR-042 and carboplatin-pemetrexed combination treatment

## 3.2.6 Secondary Objectives for Part F

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of TSR-042 and TSR-022 during TSR-042, TSR-022, and carboplatinpemetrexed combination treatment
- To evaluate ADAs of TSR-042 and TSR-022 during TSR-042, TSR-022, and carboplatinpemetrexed combination treatment

#### 3.2.7 Secondary Objectives for Part G

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of TSR-042 during TSR-042 and carboplatin nab-paclitaxel combination treatment
- To evaluate ADAs of TSR-042 during TSR-042 and carboplatin nab-paclitaxel combination treatment

#### 3.2.8 Secondary Objectives for Part H

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of TSR-042 and TSR-022 during TSR-042, TSR-022, and carboplatin nab-paclitaxel combination treatment
- To evaluate ADAs of TSR-042 and TSR-022 during TSR-042, TSR-022, and carboplatin nab-paclitaxel combination treatment

#### 3.2.9 Secondary Objectives for Part I

- To evaluate measures of clinical benefit as assessed by the Investigators, including ORR, DOR, DCR, and PFS by RECIST v1.1
- To evaluate the PK of TSR-042 and TSR-022 during TSR-042, TSR-022, and carboplatin-paclitaxel combination treatment
- To evaluate ADAs of TSR-042 and TSR-022 during TSR-042, TSR-022, and carboplatin-paclitaxel combination treatment

#### 3.3 Exploratory Objectives

## 3.3.1 Exploratory Objectives for Part A

• To explore biomarkers that may be predictive of benefit from TSR-042 and niraparib combination treatment based on the pretreatment biomarker profile

• To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042 and niraparib combination treatment and correlate with clinical benefit

#### 3.3.2 Exploratory Objectives for Part B

- To explore biomarkers that may be predictive of benefit from TSR-042 and carboplatinpaclitaxel combination treatment based on the pretreatment biomarker profile
- To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042 and carboplatin-paclitaxel combination treatment and correlate with clinical benefit

## 3.3.3 Exploratory Objectives for Part C

- To explore biomarkers that may be predictive of benefit from TSR-042, niraparib and bevacizumab combination treatment based on the pretreatment biomarker profile
- To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042, niraparib and bevacizumab combination treatment and correlate with clinical benefit

#### 3.3.4 Exploratory Objectives for Part D

- To explore biomarkers that may be predictive of benefit from TSR-042, carboplatinpaclitaxel and bevacizumab combination treatment based on the pretreatment biomarker profile
- To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment and correlate with clinical benefit

#### 3.3.5 Exploratory Objectives for Part E

- To explore biomarkers that may be predictive of benefit from TSR-042 and carboplatinpemetrexed combination treatment based on the pretreatment biomarker profile
- To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042 and carboplatin-pemetrexed combination treatment and correlate with clinical benefit

#### 3.3.6 Exploratory Objectives for Part F

• To explore biomarkers that may be predictive of benefit from TSR-042, TSR-022, and carboplatin-pemetrexed combination treatment based on the pretreatment biomarker profile

 To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042, TSR-022, and carboplatin-pemetrexed treatment and correlate with clinical benefit

## 3.3.7 Exploratory Objectives for Part G

- To explore biomarkers that may be predictive of benefit from TSR-042 and carboplatinnab-paclitaxel combination treatment based on the pretreatment biomarker profile
- To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042 and carboplatin-nab-paclitaxel combination treatment and correlate with clinical benefit

## 3.3.8 Exploratory Objectives for Part H

- To explore biomarkers that may be predictive of benefit from TSR-042, TSR-022, and carboplatin-nab-paclitaxel combination treatment based on the pretreatment biomarker profile
- To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042, TSR-022, and carboplatin-nab-paclitaxel treatment and correlate with clinical benefit

#### 3.3.9 Exploratory Objectives for Part I

- To explore biomarkers that may be predictive of benefit from TSR-042, TSR-022, and carboplatin-paclitaxel combination treatment based on the pretreatment biomarker profile
- To explore changes in biomarkers (e.g., immune cells and immune proteins) in the blood following TSR-042, TSR-022, and carboplatin-paclitaxel treatment and correlate with clinical benefit

## 4 STUDY ENDPOINTS AND EVALUATIONS

## 4.1 Safety Endpoints and Evaluations

The safety evaluations include:

- Dose-limiting toxicities (DLTs)
- Treatment emergent adverse events (TEAEs)
- Adverse Events of Special Interest (AESI)
- Clinical laboratory assessments
  - Hematology (CBC)
  - Serum chemistry
  - Coagulation factors
  - Serum/urine pregnancy testing
  - Urinalysis
  - Thyroid function including TSH, T3 or FT3, and FT4 or equivalent
- Physical examination findings
- Vital signs including height (at screening only) and weight
- ECOG performance status
- ECG
- Concomitant medications

## 4.2 Efficacy Endpoints and Evaluations

For each part, tumor response to treatment will be evaluated according to RECIST v1.1 per Investigation assessment.

The efficacy endpoints include:

- ORR (confirmed)
- DOR (confirmed)
- DCR (confirmed)
- PFS

The definition of ORR, DOR, DCR and PFS is described in Section 8.5.

#### 4.3 Pharmacokinetics Endpoints and Evaluations

Plasma and serum samples for PK determination will be collected from all patients. For Part A and Part C, plasma will be analyzed using liquid chromatography with mass spectrometry detection for niraparib and its major metabolite M1. The serum will be analyzed for TSR-042 using enzymelinked immunosorbent assay (ELISA). For Part B, Part D, and Part E to Part I serum samples will be analyzed for TSR-042 and TSR-022 using ELISA. The plasma samples will be analyzed for

carboplatin using inductively coupled plasma mass spectrometry, and for paclitaxel and pemetrexed using liquid chromatography tandem-mass spectrometry, if appropriate.

The plasma and serum PK parameters based on concentration-time data will be evaluated by non-compartmental analysis using WinNonlin version 6.2.1 or higher.

#### PK evaluations include:

- Plasma or serum concentrations
- PK parameters listed in Table 1 (but not limited to)

**Table 1: PK Parameters** 

| PK Parameter | Definition |
|---|---|
| AUC | Area under the plasma or serum concentration |
| AUCss | Area under the plasma or serum concentration at steady state |
| Cmin | Minimum observed plasma or serum concentration |
| Cmin, ss | Minimum observed plasma or serum concentration at steady state |
| Cmax | Maximum observed plasma or serum concentration |
| Cmax, ss | Maximum observed plasma or serum concentration at steady state |
| CL/F | Clearance after oral administration |
| CL | Clearance after IV administration |
| Vz/F | Volume of distribution after oral administration |
| Vz | Volume of distribution after IV administration |

#### 4.4 Immunogenicity Endpoints and Evaluations

Serum samples for the determination of TSR-042 and TRS-022 ADAs will be the same blood collections as those for the TSR-042 and TSR-022 PK assessments. ADAs will be analyzed in a tiered approach using electrochemiluminescence (i.e., screening, confirmation, titer, and neutralizing antibody assay). Minimally, ADAs will be analyzed in predose samples from all cycles collected; additional samples for ADA determination will be collected upon treatment discontinuation at a post-treatment and safety follow-up visit (i.e., approximately 90 days after the last dose of TSR-042 and TSR-022).

#### 4.5 Biomarker Evaluations

FFPE tumor archival tissue samples (mandatory (if available) for Parts F, H and I, optional for Parts A, B, C, D, E and G) and blood samples will be assessed for biomarkers that may correlate with clinical benefits from study treatments include, but not limited to,

- Germline *BRCA* mutation (g*BRCA*mut)
- Homologous recombination deficiency (HRD) status
- Phenotype and molecular profile of circulating immune cells
- Expression of PD-L1 on tumor cells
- Circulating cytokines or chemokines prior to and during treatment

#### 4.6 Other Evaluations

- Demographics and baseline characteristics
- Medical history including prior blood disorders history
- Prior anticancer treatment
  - Prior anticancer treatment for primary cancer
  - Previous radiotherapy
  - Previous cancer related surgery
- Previous and concomitant medications/procedures
  - Prior non-anticancer medications
  - Concomitant medications
  - Pemetrexed supplemental medications
  - Concomitant procedures
  - Prior and concomitant transfusions and growth factors
- HBsAg and HCV ribonucleic acid testing at baseline
- Subsequent anticancer treatment for primary cancer

## 5 DEFINITIONS AND CONVENTIONS FOR DATA HANDLING

#### **5.1** Definition of Baseline

For all evaluations unless otherwise noted, baseline is defined as the most recent non-missing measurement prior to or on the first administration of study drug. Baseline can be the same date as first dose, given the measurement is expected prior to first dose when only date information is available.

#### **5.2** First Dose Date of Study Treatment

The first dose date of study treatment is defined as the earliest dose date of study drugs in the treatment regimen.

#### 5.3 Definition of Treatment Period

Treatment period is defined as the (Minimum (start date of new anti-cancer therapy, last dose of study treatment +90) – First Dose date of study treatment )+1.

#### 5.4 Definition of Relative Study Days

Unless otherwise noted, relative study days (Rel Days) of an evaluation are defined as number of days relative to the first dose date of study drug which is designated as Day 1, and the preceding day is Day -1, the day before that is Day -2, etc.

Relative study days are calculated as following:

- If an evaluation date is before first dose date of study drug, then
  - Relative study days = first dose date of study drug an evaluation date
- If an evaluation date is on or after first dose date of study drug, then

Relative study days = first dose date of study drug - an evaluation date + 1

Relative study days take negative values if evaluation date occurs prior to first dose date and take positive values if evaluation date occurs on or after first dose date of study drug.

#### 5.5 Analysis Visit Window

For safety parameters as described in Section 4.1 excluding clinical laboratory data, measurements collected from unscheduled visits will not be included in the by-visit summary tables but will be included in the listings. Early termination visits for safety measurements will not be mapped to any scheduled post-baseline visit but will be used as the last assessment during treatment period.

#### 5.6 Safety Data Handling

For all safety data, only observed data will be used for analyses, and missing data will not be imputed.

#### **5.6.1** Handling of Unscheduled ECG Measurements

Unscheduled ECG measurements will not be used in computing the descriptive statistics for change from baseline at each post-baseline time point. However, they will be used in assessing the minimum and maximum of all visits and in the analysis of notable post-baseline abnormal ECG results.

#### 5.6.2 Handling of Partial Dates for AEs

When determining the treatment emergent AE, partial dates will be handled as follows.

- If the day of the month is missing, the onset day will be set to the first day of the month unless it is the same month and year as first dose date. In this case, the onset date will be assumed to be the first date of treatment.
- If the onset day and month are both missing, the day and month will be assumed to be January 1, unless the event occurred in the same year as the study treatment. In this case, the event onset will be coded to the day of treatment to conservatively report the event as treatment-emergent.
- A missing onset date will be coded as the day of treatment. If the resulting onset date is after a reported date of resolution, the onset date will be set equal to the date of resolution.
- Imputation of partial dates is used only to determine whether an event is treatmentemergent; data listings will present the partial date as recorded in the eCRF.

#### **5.6.3** Handling of Partial Dates for Medications

Incomplete prior/concomitant medication dates will be imputed as follows:

#### Start Date:

- If the medication start date is missing completely, then the medication start date will be imputed as the first dose date of study treatment.
- If imputed start date greater than stop date and prior to first dose, then will be imputed as stop date
- If the day of medication start date is missing, but the month and year are equal to the first dose date of study treatment, then the medication start date will be replaced by the first dose date of study treatment.
- If both the day and month of medication start date are missing but the start year is equal to the first dose date of study treatment, then the medication date will be replaced by the first dose date of study treatment.

• In all other cases the missing medication day or missing medication month will be replaced by 1.

#### Stop Date:

- Incomplete stop date will be replaced by the last day of the month (if day is missing only), if not resulting in a date later than the date of patient's death. In the latter case the date of death will be used to impute the incomplete stop date.
- If 'day' and 'month' are missing, and 'year' is not missing, then impute as December 31<sup>st</sup> (or date of study discontinuation/completion if earlier than December 31<sup>st</sup>).

In all other cases the incomplete medication stop date will not be imputed.

## 5.6.4 Handling of Partial Dates for Disease History

Incomplete dates for disease history (e.g. initial diagnosis date; date of documented, locally advanced, metastatic disease diagnosis; date of treatment initiation) will be imputed as follows:

- If the day is missing, it will be imputed to the 1st day of the month.
- If both day and month are missing, the month and day will be imputed as January 1st. If the date is completely missing, no imputation will be performed.

#### 5.6.5 Handling of Partial Dates for Progression in Prior Treatment

Incomplete dates for progression in prior treatment will be imputed as follows:

- 1. If progression date is partial missing day only, use imputed progression date (imputing missing day = 15th)
- 2. If progression date is partial missing both day and month, do the following:
- a. if next regimen start date is not missing/partial AND year (next regimen start date) = year of progression, progression date= next regimen start date
- b. if next regimen start date is not missing/partial, and year (next regimen start date) > year of progression, progression date= 15 Dec (year of progression)
- 3. Else if progression date = missing and next regimen start date is not missing/partial, PD date= Next regimen start date
- 4. Else, progression date = current regimen end date

#### 6 PLANNED ANALYSIS

#### 6.1 Changes from Planned Analyses in the Protocol

In order to capture immune-related adverse events that occur long after the completion of immunotherapy treatment, analyses of AEs will be performed for those events that are considered treatment-emergent where treatment-emergent is defined as any AE with onset beginning at the day of first administration of study treatment throughout the treatment period until 90 days after the last dose of study treatment, instead of 30 days after the last dose of study treatment as specified in the protocol.

Parts G, H and I as defined in the protocol is not included in the analysis as these parts were not initiated.

Data from parts E and F will be only listed due to small sample size.

#### **6.2** Interim Analysis

A 2-stage 6 + 6 scheme is used for dose finding in Part A and Part C. Part C will be initiated after dose level 1 (niraparib 200 mg) if Part A is determined to be safe. Part F will be initiated after TSR-042 and carboplatin-pemetrexed combination treatment in Part E is determined to be safe. Part H will be initiated after TSR-042 and carboplatin-nab-paclitaxel combination treatment in Part G is determined to be safe.

So, interim safety will be evaluated after completion of dose level 1 for Part A, and then for Part C. Safety will also be evaluated after completion of Part E and G.

Similarly, preliminary safety will be evaluated after completion of dose level 2 in Part A before the start of dose level 2 study in Part C, after completion of Part E before starting Part F, and after completion of Part G before starting Part H.

#### 6.3 Final Analyses and Reporting

All final planned analyses per protocol and this analysis plan will be performed only after database freeze.

## 7 ANALYSIS POPULATIONS AND APPLICATIONS

## 7.1 All Patients Population

All Patients Population includes all patients who sign an informed consent form.

#### 7.2 Safety Population

Safety Population includes all patients who receive any amount of study drug.

All safety endpoints will be assessed in the safety population, except DLT assessment which will include only those patients completing the first cycle of therapy, unless the patient discontinued study treatment due to a DLT.

## 7.3 Application of Analysis Populations

Unless otherwise noted, the analysis populations that will be used for creating the summary table(s) of each type is provided in Table 2Table 2. Populations used for listing can be found in Section 9 (Planned Statistical Tables, Figures and Listings).

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

**Table 2: Application of Populations on Tables and Figures** 

| Туре | All | Safety |
|-------------------------------------------------|-----|--------|
| Enrollment | X | X |
| Disposition | | X |
| Demographics and baseline characteristics | | X |
| Protocol deviations | | X |
| Medical and disease history | | X |
| Prior therapies/surgeries | | X |
| Prior and concomitant medications or procedures | | X |
| Efficacy evaluations | | X |
| Safety evaluations | | X |
| Treatment exposure | | X |

#### 8 STATISTICAL CONSIDERATIONS

All analyses described in this plan are considered a priori analyses in that they have been defined prior to freezing the database. All other analyses, if any, designed subsequently to locking the database, will be considered post hoc analyses and will be described as exploratory analyses in the Clinical Study Report.

All summaries and statistical analysis will be performed by SAS v9.4 or later.

#### 8.1 General Statistical Procedures

Frequency distributions for categorical variables will be provided as number of patients with a response in the category and the percentages of the total number of patients in that column. Percentages will be based on number of patients in the given population as noted. Percentages will be reported to one decimal place.

A 2-sided 90% exact binomial (Clopper-Pearson) confidence interval (CI) for categorical variables without multiplicity adjustment will be provided where appropriate for efficacy analysis.

The descriptive statistics for continuous variables will be number of patients, mean, standard deviation (STD), median, minimum (Min) and maximum (Max). Mean and median will be reported to 1 more decimal place than the raw data, while the standard deviation (STD) will be reported to 2 more decimal places than the raw data. Minimum and maximum will be reported the same as the original data.

Time-to-event analyses will be performed using Kaplan-Meier methods.

Otherwise stated, all statistical summary will be performed for Part A, B, C & D.

Listings will be ordered by study Part, patient ID and visit for available data unless otherwise specified in the text. Listings that contain an evaluation date will also contain relative study day (Rel days) which is defined as number of days relative to the first dose date of study drug (see Section 5.2 for details).

Analysis visit windows and safety data handling (partial dates of AEs and medications) are described in Section 5.5 to Section 5.6.

TSR-042 is fixed dose regimen (i.e. 4 x 500 mg Q3W followed by 1000 mg Q6W), the data will be summarized by patient ID and visit without distinguishing TSR-042 dose levels.

#### 8.2 Enrollment and Disposition

#### 8.2.1 Patients Enrollment

Patients enrollment will be summarized for all patients, and safety population. The number of patients in each analysis population will be presented for PartsA -D

Enrollment information will be provided in a data listing for All Patients Population and safety population.

## **8.2.2** Patients Disposition

In this study, each part consists a combination of several study drugs. The Treatment regimen is considered discontinued if patients discontinued all study drugs in the regimen.

Patients' discontinuation from treatment and primary reasons will be tabulated by study drug using Safety Population.

Patients' discontinuation from study and primary reasons will be tabulated for Safety Population.

Discontinued patients from treatment and from study will be provided in a data listing for Safety Population.

#### **8.2.3** Protocol Deviations

Important or significant protocol deviations (PDVs) will be assessed by TESARO and GSK personnel following Protocol Deviation Guideline outlined in Clinical Management Plan.

- A PDV is classified as important if there is the potential to impact the completeness, accuracy, and/or reliability of the study data, or affect a patient's rights, safety, or wellbeing.
- A PDV is classified as significant if it is confirmed to adversely impact the completeness, accuracy, and/or reliability of the study data, or affect a patient's rights, safety, or wellbeing.

If a reported PDV does not meet classification criteria for importance or significance, the PDV will be reported as a protocol deviation without a classification.

All PDVs will be identified and finalized prior to database freeze

Number and percentage of patients with a significant or important PDV will be tabulated by type of deviation for Safety Population.

All protocol deviations will be listed for Safety Population.

## 8.3 Demographics and Baseline Characteristics

#### 8.3.1 Demographics, Baseline and Disease Characteristics

Demographic and baseline (see Section 5.1 for baseline definition) characteristics will be tabulated using descriptive statistics for Safety Population for each part. The following variables will be included in the tables:

- The demographic data are:
  - Age (years) as (date of screening date of birth) / 365.25 if date of birth is reported, or age as reported on the eCRF will be used
  - Age category (18 to < 65, 65 to < 74; and  $\ge 75$ )
  - Sex
  - Race
  - Ethnicity
- Baseline characteristics include:
  - Height (cm)
  - Weight (kg)
  - BMI (body mass index, kg/m<sup>2</sup>, calculated as weight (kg) / height (m)<sup>2</sup>)
  - BSA (m<sup>2</sup>, calculated as ([height (cm) × weight (kg)] / 3600)<sup>0.5</sup>)
  - ECOG performance status
- Primary Cancer History include:
  - Primary tumor site at first diagnosis
  - Cancer stage at first and most recent diagnosis
  - Time from first diagnosis to the date of first dose of study treatment (months),
     calculated as (date of first dose of the treatment date of first diagnosis)/30.4375

Conversions for height and weight are as follows:

```
Height (cm) = Height (inches) x 2.54
Weight (kg) = Weight (lb) x 0.4536
```

Demographics, baseline characteristics and primary cancer history will be listed for Safety Population.

## **8.3.2** Medical History

The medical history will be coded using version 23.0 of Medical Dictionary for Regulatory Activities (MedDRA) dictionary.

The frequency count and percentage of patients experiencing any medical conditions will be tabulated by system organ classifications (SOC) and preferred term (PT) of MedDRA for Safety

Population. If a PT or SOC was reported more than once for a patient, the patient would only be counted once in the incidence for that SOC or PT.

Patients' history of blood disorder will be summarized by count and percentage for Safety Population.

A data listing of medical history and prior blood disorders history will be provided for Safety Population.

#### **8.3.3** Prior Anticancer Treatment

Prior anticancer treatment will be tabulated for each Part and overall for Safety Population. The following variables will be included in the tables:

- Number of regimens
- Reason for administration of last treatment
- Reason for discontinuation of last treatment
- Time from end of last treatment to the date of first dose of study treatment (months), defined as (date of first dose of the treatment stop date of last treatment)/30.4375
- Best response during last treatment
- Any surgeries related to cancer
- Any radiotherapy prior to informed consent

Prior anticancer treatment for primary cancer, prior and concomitant radiotherapy, and previous surgery history will be provided for Safety Population.

#### **8.3.4** Prior and Concomitant Medication/Procedures

All medications as documented by the investigator will be coded using Anatomical Therapeutic Chemical (ATC) classification based on the World Health Organization (WHO) Drug Dictionary (WHO-DD Sept 2018).

Prior non-anticancer medications are defined as any medications, other than study drugs, medications for cancer treatment and pre-medications for study treatment, which ended prior to the first dose date of study treatment.

Concomitant medications are medications other than study treatments, being taken on or after the initial study treatment dosing date through 90 days after the last dose or until the start of subsequent antitumor therapy.

The count and percentage of patients who took prior and concomitant medications will be provided by WHO Drug ATC level 3 and preferred term (PT) for Safety Population. For the summary tables, if a patient has taken a prior or concomitant medication more than once, the patient will be counted only once for the medication.
Patients' prior transfusion and growth factor will be summarized by count and percentage.

Prior and concomitant medication, pemetrexed supplemental medications, concomitant procedures, prior and concomitant transfusions and growth factors will be listed for Safety Population.

### 8.3.5 HBsAg and HCV Ribonucleic Acid Testing at Baseline

The testing results will be listed for Safety Population.

### 8.4 Safety Analysis

#### 8.4.1 Adverse Events

AEs will be coded using MedDRA v23.0 and will be classified by SOC and PT of MedDRA. Severity of AEs will be assessed by investigators according to CTCAE (v4.03).

A treatment-emergent AE (TEAE) will be defined as any new AE that begins, or any preexisting condition that worsens in severity during the treatment period (see Section 5.3 for definition of treatment period).

TEAEs are classified as Related or Unrelated to study drugs by the Investigator. Any TEAEs for which the relationship to study drug is missing will be considered as related to study drugs.

The following types of summaries will be provided by study drug. The summary will be sorted by decreasing frequency of PT (number of patients in total) within SOC which is sorted alphabetically.

- Overview of TEAEs
- DLT by SOC and PT
- TEAEs by SOC and PT
- TEAEs by PT in decreasing frequency
- Immune Related TEAE by PT
  - Preferred term and SOC for Immune Related Adverse events are defined in APPENDIX
  - Immune Related TEAE by PT will summarize incidence of Grade 2 and above events as overall, TSR-042 related events, Grade 3 and above events, TSR-042 related Grade 3 and above, SAE, TSR-042 related SAE and events leading to TSR-042 discontinuation
- Drug-Related TEAEs by PT in descending frequency
  - Niraparib-related TEAEs by PT in descending frequency
  - TSR-042-related TEAEs by PT in descending frequency

- TSR-022-related TEAEs by PT in descending frequency
- Bevacizumab-related TEAEs by PT in descending frequency
- Carboplatin-related TEAEs by PT in descending frequency
- Paclitaxel -related TEAEs by PT in descending frequency
- Drug-related TEAEs by SOC and PT
  - Niraparib-related TEAEs by SOC and PT
  - TSR-042-related TEAEs by SOC and PT
  - TSR-022-related TEAEs by SOC and PT
  - Bevacizumab-related TEAEs by SOC and PT
  - Carboplatin-related TEAEs by SOC and PT
  - Paclitaxel -related TEAEs by SOC and PT
- TEAEs by SOC, PT and Maximum CTCAE toxicity grade  $\geq 3$
- Drug-related TEAEs by SOC, PT and Maximum CTCAE grade  $\geq 3$ 
  - Niraparib-related TEAEs by SOC, PT and Maximum CTCAE grade ≥ 3
  - TSR-042-related TEAEs by SOC, PT and Maximum CTCAE grade ≥ 3
  - TSR-022-related TEAEs by SOC, PT and Maximum CTCAE grade ≥ 3
  - Bevacizumab-related TEAEs by SOC, PT and Maximum CTCAE grade ≥ 3
  - Carboplatin-related TEAEs by SOC, PT and Maximum CTCAE grade  $\geq 3$
  - Paclitaxel-related TEAEs by SOC, PT and Maximum CTCAE grade ≥ 3
- Serious AEs by SOC and PT
- Drug-related serious AEs by SOC and PT
  - Niraparib-related Serious AEs by SOC and PT
  - TSR-042-related Serious AEs by SOC and PT
  - TSR-022-related Serious AEs by SOC and PT
  - Bevacizumab-related Serious AEs by SOC and PT
  - Carboplatin-related Serious AEs by SOC and PT
  - Paclitaxel -related Serious AEs by SOC and PT
- TEAEs leading to study drug discontinuation by SOC and PT
  - TEAEs leading to niraparib discontinuation
  - TEAEs leading to TSR-042 discontinuation
  - TEAEs leading to TSR-022 discontinuation
  - TEAEs leading to bevacizumab discontinuation
  - TEAEs leading to carboplatin discontinuation
  - TEAEs leading to paclitaxel discontinuation
- Drug-related TEAEs leading to study drug discontinuation by SOC and PT
  - Drug-related TEAEs leading to niraparib discontinuation
  - Drug-related TEAEs leading to TSR-042 discontinuation
  - Drug-related TEAEs leading to TSR-022 discontinuation
  - Drug-related TEAEs leading to bevacizumab discontinuation

- Drug-related TEAEs leading to carboplatin discontinuation
- Drug-related TEAEs leading to paclitaxel discontinuation
- TEAEs leading to niraparib reduction or interruption by SOC and PT
- TEAEs leading to study drug interruption by SOC and PT
  - TEAEs leading to TSR-042 interruption
  - TEAEs leading to TSR-022 interruption
  - TEAEs leading to bevacizumab interruption
  - TEAEs leading to carboplatin interruption
  - TEAEs leading to paclitaxel interruption
- AEs of special interest (AESIs) by SOC and PT
- Death and primary reasons causing death

If a SOC or PT was reported more than once for a patient, the patient would only be counted once in the incidence for that SOC or PT.

In tabulation by severity (i.e., CTCAE grade),

- For a given preferred term, only the most severe preferred term for each patient will be included.
- For a given system organ class, only the most severe system organ class for each patient will be included.

The following tables presented as listings will be provided:

- Deaths
- Serious AEs
- TEAEs leading to drug reduction or interruption.
- TEAEs leading to treatment discontinuation

COVID19 assessments and symptom assessments for subjects with COVID19 Adverse events will be listed.

AEs will be listed for All Safety Population.

#### 8.4.2 Study Drug Exposure

Study drug will be summarized using descriptive statistics for Safety Population including:

- Duration of drug exposure
- Number of treatment cycles (Cycle 1, Cycle 2, etc.)
- Actual dose intensity (exclude Carboplatin)
- Relative dose intensity (exclude Carboplatin)
- Number of patients with dose interruptions

• Number of patients with Niraparib dose reduction

Duration of exposure and dose intensity will be calculated as described in

Table 3 for each drug. Dose intensity for Carboplatin will not be included due to unit conversion issue between AUC and mg/m<sup>2</sup>.

For each study treatment, swimmer plots displaying the duration of treatment for each patient will be presented by including indicators:

- Primary tumor type
- Treatment status (ongoing or discontinued)
- Response at each tumor assessment

Details of study treatment exposure will be listed for Safety Population.

**Table 3: Extent of Study Drug Exposure** 

| Parameter | Niraparib | TSR-042 | TSR-022 | Paclitaxel | Bevacizumab | Carboplatin |
|---|---|---|---|---|---|---|
| Dosing | Dose level 1: | Part A to D: 500mg Q3W for | Dose level 1: | 175mg/m <sup>2</sup> | 15mg/kg | AUC of 5 or 6 |
| schedule per protocol | 200mg daily | first 4 cycles, | 900mg Q3W | Q3W | Q3W | Q3W |
| protocor | Dose level2: | 1,000mg Q6W on and after | Dose level -1: | | | |
| | 300mg daily | Day 1 Cycle 5 | 300mg Q3W | | | |
| | | <b>Part E to I:</b> 500mg Q3W | | | | |
| Intended dose (unit) | (mg/day) | (mg/day) | (mg/day) | (mg/m <sup>2</sup><br>/day) | (mg/kg /day) | |
| (unit) | Dose level 1: | Part A to D: | 900/21 | /day) | 15/21 | |
| | 200/1 | First 4 Cycles: 500/21 | | 175/21 | | |
| | Dose level2: 300/1 | On and after Cycle 5: 1000/42 | | | | |
| | | Part E to I: | | | | |
| | | 500/21 | | | | |
| Duration of | (day) | (day) | (day) | (day) | (day) | (day) |
| Treatment (unit) | Last dose | Part A to Part D: First 4 | Last dose date - | Last dose | Last dose date | Last dose date |
| (unit) | date - Start | cycles: | Start dose date | date - Start | - Start dose | - Start dose |
| | dose date +1 | Last dose date prior to cycle 5 – | +21 | dose date + | date + 21 | date + 21 |
| | | Start dose date + 21 | | 21 | | |
| | | After cycle 5: | | | | |
| | | Last dose date – First Dose | | | | |
| | | Date at or after Cycle 5 + 42 | | | | |

| Parameter | Niraparib | TSR-042 | TSR-022 | Paclitaxel | Bevacizumab | Carboplatin |
|---|---|---|---|---|---|---|
| | | Part E to Part F: Last dose date prior to cycle 5 – Start dose date + 21 Note: First 4 cycles: Last dose date prior to cycle 5 – Start dose date + 21. If the subject died less than 21 days after last dose date then duration = death date – start dose date +1. After cycle 5: Last dose date – First Dose Date at or after Cycle 5 + 42. If the subject died less than 42 days after last dose date then duration = death date – start dose date + 1. | | | | |
| Actual | (mg) | (mg) | (mg) | (mg/m²) | (mg/kg) | |
| Cumulative<br>Dose (unit) | Sum of the doses administered to a patient during the treatment period [1] For Niraparib, the sum of the doses consumed (mg) is the total number of capsules consumed multiplyin mg. The total number of capsules consumed is the sum of the number of capsules dispensed less the sum of of capsules returned by the patient during the study. Unused capsules not returned will be assumed to have consumed. [2] For TSR-042, it is calculated separately for the first 4 cycles and cycles after cycle 5 for Part A to Part D | | | n of the number ave been art D. | | |
| | (mg/day) | nat do not have kits actual cumulation (mg/day) | (mg/day) | (mg/m <sup>2</sup> /day) | uration of the drug (mg/kg/day) | taken. |

TESARO Inc.


Statistical Analysis Plan
Dated:18SEP2020

| Parameter | Niraparib | TSR-042 | TSR-022 | Paclitaxel | Bevacizumab | Carboplatin |
|---|---|---|---|---|---|---|
| Actual Dose<br>Intensity<br>(unit) | Actual Cumulative Dose / Duration of treatment For TSR-042, calculated separately for the first 4 cycles and cycles at or after cycle 5 for Part A to Part D. | | | | | |
| Relative Dose<br>Intensity (%) | | Actual Dose Intensity/Intended Dose | | | | |
| | For TSR-042, c | alculated separately for the first 4 | cycles and cycles at | or after cycle 3 | 5 for Part A to Part | D. |

### **8.4.3** Clinical Laboratory Tests

All laboratory parameters collected at each center's local laboratory will be normalized by converting values in original units to values in SI units and classified as normal, low, or high based on normal ranges supplied by the local laboratories and upon employing standardization.

For hematology, coagulation, serum chemistry and thyroid function laboratory parameters which are normalized in SI units, descriptive summary tables for observed values and changes from baseline will be provided by visit for Safety Population.

The laboratory test results will be categorized according to NCI CTCAE v4.03 toxicity grades. Shift tables from baseline toxicity to maximum post-baseline toxicity grade will be provided for Alkaline phosphatase increased, Alanine aminotransferase increased, Aspartate aminotransferase increased, Blood bilirubin increased, Hypoalbuminemia, Creatinine increased, Hypocalcemia, Hypercalcemia, Hypomagnesemia, Hypermagnesemia, Hypokalemia, Hyperkalemia, Hyponatremia, Hypernatremia, Anemia, White blood cell decreased, Platelet count decreased, Lymphocyte count decreased, Neutrophil count decreased applicable hematology and chemistry laboratory parameter in Safety Population.

Continuous urinalysis laboratory parameters at each visit will be summarized using descriptive statistics. The categorical urinalysis parameters will be summarized using frequency table.

Summary of liver function tests will include the following categories. The number and percentage of patients with each of the following during the treatment period will be summarized by treatment group: Patients with maximum elevations in categories of < 3xULN,  $\ge 3xULN$  to <5xULN,  $\ge 5xULN$  to <10xULN,  $\ge 10xULN$  to <20xULN, and  $\ge 20xULN$  under treatment

- o AST and ALT, separately
- Any combinations of elevation categories under treatment of either ALT or AST
- Patient with normal values at baseline and any maximum elevations of TBL under treatment <1.5xULN, ≥1.5xULN to <2xULN, ≥2x ULN
- Patients with normal values at baseline and any maximum elevations of ALP under treatment <1.5xULN, ≥1.5xULN to <2xULN, ≥2x ULN
- Concurrent ALT  $\geq$  3×ULN and TBL  $\geq$  2×ULN Concurrent AST  $\geq$  3×ULN and TBL  $\geq$  2×ULNConcurrent (ALT or AST)  $\geq$  3×ULN and TBL  $\geq$  2×ULN
- Concurrent (ALT or AST)  $\geq 3 \times ULN$  and TBL  $\geq 2 \times ULN$  and ALP  $\geq 2 \times ULN$
- Potential Hy's law: Concurrent (ALT or AST)  $\geq 3 \times$  ULN and TBL  $\geq 2 \times$  ULN and ALP <  $2 \times$  ULN

Concurrent measurements are defined as measurements that occur on the same date.

Separate listings will be provided for all laboratory tests including pregnancy testing for Safety Population.

In general, all by visit summaries of clinical laboratory parameters will only be summarized up to and including month 6 and at the treatment discontinuation visit. The maximum and minimum calculations will use all post-baseline data, including any unscheduled assessments.

Unscheduled measurements will not be used in computing the descriptive statistics for change from baseline at each post-baseline time point. However, they will be used in assessing the minimum and maximum of all visits and in the analysis of notable post-baseline results (for example shift tables).

## 8.4.4 Vital Signs

A patient-detailed listing of vital signs (including systolic and diastolic blood pressure (mmHg), pulse (bmp), temperature (°C)), height (cm) and weight (kg)) will be provided for Safety Population.

Conversion of temperature is as following:

Temperature (°C) = (Temperature (°F) 
$$-32$$
) x  $5/9$ 

## 8.4.5 Physical Examination Findings

Physical examination will be listed for Safety Population.

### **8.4.6** ECOG performance status

The ECOG shift from baseline score to worst (highest) post-baseline score during the on-treatment period will be summarized for Safety Population.

Listings will be provided for Safety Population.

## 8.4.7 Electrocardiogram (ECG)

The following analyses will be performed on Safety Population for each applicable ECG parameters (HR, RR, PR, QRS, QT and QTcF) measured during the on-treatment period (see Section 5.3 for definition).

- For each of continuous ECG parameters, descriptive statistics at baseline, at each post-baseline time point and changes from baseline at each post-baseline time point. If there are multiple measurements at a time point, the average of the replicate measurements should be taken at each time point.
- Frequency (number and percentage) of patients with notable ECG values according to the following categories:
  - QTcF increase from baseline > 30 ms, > 60 ms


- QTcF > 450 ms, > 480 ms, > 500 ms
- HR  $\leq$  50 bpm and decrease from baseline  $\geq$  20 bpm
- HR  $\geq$  120 bpm and increase from baseline  $\geq$  20 bpm
- $PR \ge 220 \text{ ms}$  and increase from baseline  $\ge 20 \text{ ms}$
- QRS  $\geq$  120 ms

Patients with notable ECG interval values and qualitative ECG abnormalities will be listed for each patient and time point and the corresponding notable values and abnormality findings will be included in the listings.

Listing will be presented for Safety Population.

## 8.5 Efficacy Analysis

RECIST v1.1 will be used by the Investigator as the primary measure for assessment of tumor response, date of disease progression. Tumor response assessment is performed every 12 weeks  $(84 \pm 10 \text{ days})$  from the date of the first dose of study treatment until progression while on study treatment, independent of cycle delays or dose interruptions, or at any time when progression of disease is suspected.

The following plots will be provided for Safety Population:

- Spider plots, displaying the percent change from baseline over the period of subject evaluation.
- Waterfall plots, displaying the best percentage change from baseline in the sum of the diameter of all target lesions for each patient with measurable disease at baseline and at least one valid post-baseline assessment.

Detailed tumor time-point response will be listed for Safety Population.

## 8.5.1 Best Overall Response when confirmation is required

To confirm CR or PR response, tumor imaging may be performed at the earliest 4 weeks after the first indication of response or at the next scheduled scan (i.e., 12 weeks later), whichever is clinically indicated. Tumor imaging for confirmation of response occurred less than 4 weeks after the first indication of response of CR or PR may be used for clinical decision, but it will NOT be used for determination of BOR

Statistical Analysis Plan **Dated:18SEP2020** 

TESARO Inc.

Table 4

| Overall response first time point | Overall response subsequent time point | Best overall response |
|---|---|---|
| CR | CR | CR |
| CR | PR | SD provided minimum criteria* for SD duration met, otherwise, PD |
| CR | SD | SD provided minimum criteria* for SD duration met, otherwise, PD |
| CR | PD | SD provided minimum criteria* for SD duration met, otherwise, PD |
| CR | NE | SD provided minimum criteria* for SD duration met, otherwise, NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD |
| PR | PD | SD provided minimum criteria* for SD duration met, otherwise, PD |
| PR | NE | SD provided minimum criteria* for SD duration met, otherwise, NE |
| NE | NE | NE |

<sup>\*</sup> The minimum criteria SD duration for this study is defined as 12 weeks minus 10 days (12 x 7 – 10 = 74 days) from date of first dose of study treatment.

Abbreviation: CR = complete response; PR = partial response; SD = stable disease; PD=Progressive disease; NE=Not eveluated

## **8.5.2** Objective Response Rate

Confirmed ORR is defined as the proportion of patients who have achieved confirmed BOR of CR or PR, evaluated using RECIST v1.1 based on Investigator assessment.

Confirmed ORR will be summarized by count and percentage for Safety Population.

## **8.5.3** Duration of Response

DOR is defined as the time from first documentation of overall response leading to a confirmed CR or PR until the time of first documentation of disease progression by RECIST v1.1 or death by any cause.

DOR will be calculated only for patients who responded to the study treatment using the censoring rules specified in Table.

DOR in months is defined as

• (Date of Event or Censoring – Date of first confirmed CR or PR + 1)/30.4375

Due to a small sample size in each Part, DOR will be listed only.

**Table 5: Censoring Rules Used for DOR Analysis** 

| Situation | Date of Event or Censoring | Outcome |
|---|---|---|
| Start of subsequent anti-cancer therapy without a prior documented progression or death | Date of last evaluable radiologic tumor assessment prior to or on the date of initiation of the subsequent anti-cancer therapy | Censored |
| No documented radiologic progression and no subsequent anti-cancer therapy started | Date of last evaluable radiologic tumor assessment | Censored |
| Documented radiologic progression or death after two or more consecutive missing radiologic assessments | Date of last evaluable radiologic tumor assessment before the missed tumor assessments | Censored |
| Documented radiologic progression or death | Earliest date of documented radiologic progression or death | Event |

Table 6: Assessment window to be considered for missing visit information in tumor data is given below

| Target day | Analysis window | | Analysis Visit |
|------------|-----------------|---------|-------------------|
| | Start day | End day | |
| 60 | 1 | 73 | Unscheduled 2.01 |
| 70 | 1 | 73 | Unscheduled 2.02 |
| 83 | 74 | 94 | Week 12 |
| 95 | 95 | 157 | Unscheduled 12.01 |
| 170 | 158 | 178 | Week 24 |

#### 8.5.4 Disease Control Rate

Confirmed DCR is defined as the proportion of patients who have achieved confirmed BOR of CR, PR, or stable disease (SD) per RECIST v1.1.

Confirmed DCR will be summarized using frequency tables for Safety Population.

#### **8.5.5** Progression Free Survival

PFS is defined as the time from the date of the first dose of study treatment to the earlier date of assessment of progression, or death by any cause in the absence of progression by RECIST v1.1.

PFS in months will be calculated as following using the censoring rules specified in Table:

• (Earlier Date of Event or Censoring – First dose date of study treatment + 1) / 30.4375

The Kaplan-Meier (KM) method will be used to estimate the distribution of PFS for Safety Population including the number and percentage of events, number and percentage of censored patients, and the 25th, 50th, and 75th percentiles of times-to-event with 95% CIs. Survival risks at 6 and 12 months will be provided if applicable.

A KM plot will be provided to graphically present the PFS.

**Table 7: Censoring Rules Used for PFS Analysis** 

| Situation | <b>Date of Event or Censoring</b> | Outcome |
|-----------|-----------------------------------|---------|

# TESARO Inc.

| No baseline tumor assessments | First dose date | Censored |
|---|---|---|
| No post-baseline tumor assessments and no death | First dose date | Censored |
| Start of subsequent anti-cancer therapy prior to a documented radiologic progression or death | Date of last evaluable radiologic tumor assessment prior to or on the date of initiation of the subsequent anti-cancer therapy | Censored |
| No documented radiologic progression, no subsequent anti-cancer therapy started, and no death | Date of last evaluable radiologic tumor assessment | Censored |
| Documented radiologic progression or death after two or more consecutive missing radiologic assessments | Date of last evaluable radiologic tumor assessment before the missed tumor assessments | Censored |
| Documented radiologic progression or death | Earliest date of documented radiologic progression or death | Event |

# 9 APPENDIX: Immune Related Adverse Events

| Immune Related Adverse Events - Preferred | Immune Related Adverse Events- System |
|---|---|
| Term(irAE_PT) | Organ Class(irAE_SOC) |
| Pneumonitis | Immune-mediated Pulmonary |
| Sarcoidosis | Immune-mediated Pulmonary |
| Colitis | Immune-mediated Gastrointestinal |
| Diarrhoea | Immune-mediated Gastrointestinal |
| Gastroenteritis | Immune-mediated Gastrointestinal |
| Enteritis | Immune-mediated Gastrointestinal |
| Gastritis | Immune-mediated Gastrointestinal |
| Duodenitis | Immune-mediated Gastrointestinal |
| Autoimmune hepatitis | Immune-mediated hepatic |
| Hepatitis | Immune-mediated hepatic |
| Hepatitis toxic | Immune-mediated hepatic |
| Liver injury | Immune-mediated hepatic |
| Transaminases increased | Immune-mediated hepatic |
| Aspartate aminotransferase increased | Immune-mediated hepatic |
| Alanine aminotransferase increased | Immune-mediated hepatic |
| Blood bilirubin increased | Immune-mediated hepatic |
| Hyperbilirubinaemia | Immune-mediated hepatic |
| Hepatic enzyme increased | Immune-mediated hepatic |
| Hyperthyroidism | Immune-mediated endocrinopathies |
| Hypothyroidism | Immune-mediated endocrinopathies |

| Thyroid disorder | Immune-mediated endocrinopathies |
|---|---|
| Thyroiditis | Immune-mediated endocrinopathies |
| Hypophysitis | Immune-mediated endocrinopathies |
| Hypopituitarism | Immune-mediated endocrinopathies |
| Adrenal insufficiency | Immune-mediated endocrinopathies |
| Secondary adrenocortical insufficiency | Immune-mediated endocrinopathies |
| Type 1 diabetes mellitus | Immune-mediated endocrinopathies |
| Diabetic ketoacidosis | Immune-mediated endocrinopathies |
| Hyperglycaemia | Immune-mediated endocrinopathies |
| Nephritis | Immune-mediated renal |
| Renal impairment | Immune-mediated renal |
| Blood creatinine increased | Immune-mediated renal |
| Rash | Immune-mediated skin adverse reactions |
| Rash maculo-papular | Immune-mediated skin adverse reactions |
| Rash macular | Immune-mediated skin adverse reactions |
| Rash erythematous | Immune-mediated skin adverse reactions |
| Rash papular | Immune-mediated skin adverse reactions |
| Rash pruritic | Immune-mediated skin adverse reactions |
| Rash pustular | Immune-mediated skin adverse reactions |
| Erythema | Immune-mediated skin adverse reactions |
| Exfoliative rash | Immune-mediated skin adverse reactions |
| Dermatitis exfoliative | Immune-mediated skin adverse reactions |
| Autoimmune dermatitis | Immune-mediated skin adverse reactions |
| Pemphigoid | Immune-mediated skin adverse reactions |

| Vitiligo | Immune-mediated skin adverse reactions |
|-------------------------------|----------------------------------------|
| Pruritus | Immune-mediated skin adverse reactions |
| Stevens-Johnson syndrome | Immune-mediated skin adverse reactions |
| Toxic epidermal necrolysis | Immune-mediated skin adverse reactions |
| Pancreatitis | Immune-mediated pancreatitis |
| Pancreatitis acute | Immune-mediated pancreatitis |
| Autoimmune pancreatitis | Immune-mediated pancreatitis |
| Amylase increased | Immune-mediated pancreatitis |
| Lipase increased | Immune-mediated pancreatitis |
| Aplastic anaemia | Immune-mediated hematologic |
| Autoimmune haemolytic Anaemia | Immune-mediated hematologic |
| Haemolytic anaemia | Immune-mediated hematologic |
| Arthritis | Immune-mediated musculoskeletal |
| Myositis | Immune-mediated musculoskeletal |
| Polymyalgia rheumatica | Immune-mediated musculoskeletal |
| Rhabdomyolysis | Immune-mediated musculoskeletal |
| Autoimmune neuropathy | Immune-mediated nervous system |
| Polyneuropathy | Immune-mediated nervous system |
| Neuropathy peripheral | Immune-mediated nervous system |
| Peripheral sensory neuropathy | Immune-mediated nervous system |
| Hypoaesthesia | Immune-mediated nervous system |
| Paraesthesia | Immune-mediated nervous system |
| Facial paresis | Immune-mediated nervous system |
| Dysaesthesia | Immune-mediated nervous system |

| Demyelination | Immune-mediated nervous system |
|-----------------------------------------|--------------------------------|
| Myelitis | Immune-mediated nervous system |
| Encephalitis autoimmune | Immune-mediated nervous system |
| Seizure | Immune-mediated nervous system |
| Guillain-Barre syndrome | Immune-mediated nervous system |
| Motor dysfunction | Immune-mediated nervous system |
| Myasthenia gravis | Immune-mediated nervous system |
| Myasthenic syndrome | Immune-mediated nervous system |
| Iridocyclitis | Immune mediated Ocular |
| Uveitis | Immune mediated Ocular |
| Iritis | Immune mediated Ocular |
| Myocarditis | Immune-mediated cardiovascular |
| Vasculitis | Immune-mediated cardiovascular |
| Pericarditis | Immune-mediated cardiovascular |
| Hypersensitivity | Hypersensitivity |
| Infusion related reaction | Hypersensitivity |
| Anaphylactic reaction | Hypersensitivity |
| Drug hypersensitivity | Hypersensitivity |
| Type I hypersensitivity | Hypersensitivity |
| Haemophagocytic lymphohistiocytosis | Immune-mediated Others |
| Histiocytosis | Immune-mediated Others |
| Histiocytic necrotising lymphadenitis | Immune-mediated Others |
| Systemic inflammatory response syndrome | Immune-mediated Others |
| Vogt-Koyanagi-Harada disease | Immune-mediated Others |

# 10 PLANNED STATISTICAL TABLES, FIGURES AND LISTINGS

# **Programming Specifications**

1. add following footnotes for corresponsing Part(s) included in the summary.

```
Part A-200: TSR-042 and niraparib (200mg) combination treatment
Part A-300: TSR-042 and niraparib (300mg) combination treatment
Part A: TSR-042 and niraparib (300mg/900mg) combination treatment
Part B: TSR-042 and carboplatin-paclitaxel combination treatment
Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment
Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment
Part C: TSR-042, niraparib (200mg/300mg) and bevacizumab combination treatment
Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment
Part E: TSR-042 and carboplatin-pemetrexed combination treatment
Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment
Part F-900: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment
Part F: TSR-042, TSR-022 (300mg/900mg) and carboplatin-pemetrexed combination treatment
```

- 2. Summary tables for adverse events (AEs) will be sorted by decreasing total number of patients of preferred term (PT) within system organ class (SOC) which is sorted alphabetically.
- 3. Listing will be sorted by Part, patient ID and visit.
- 4. Date is presented as MMDDYYY and time is presented as HH:MM:SS.

TESARO Inc.

# TABLE OF CONTENTS

| Table 14.1.1 Overview of Patients Enrollment | 68 |
|---|---|
| Table 14.1.2.1 Patients Disposition for Part A (Safety Population) | 69 |
| Table 14.1.2.2 Patients Disposition for Part B (Safety Population) | 70 |
| Table 14.1.2.3 Patients Disposition for Part C (Safety Population) | 71 |
| Table 14.1.2.4 Patients Disposition for Part D (Safety Population) | 73 |
| Table 14.1.3.1 Protocol Deviation by Category and Severity for Part A (Safety Population) | 74 |
| Table 14.1.3.2 Protocol Deviation by Category and Severity for Part B (Safety Population) | 76 |
| Table 14.1.3.3 Protocol Deviation by Category and Severity for Part C (Safety Population) | 76 |
| Table 14.1.3.4 Protocol Deviation by Category and Severity for Part D (Safety Population) | 76 |
| Table 14.1.4.1 Demographic Characteristics for Part A (Safety Population) | 77 |
| Table 14.1.4.2 Demographic Characteristics for Part B (Safety Population) | 78 |
| Table 14.1.4.3 Demographic Characteristics for Part C (Safety Population) | 78 |
| Table 14.1.4.4 Demographic Characteristics for Part D (Safety Population) | 78 |
| Table 14.1.5.1 Baseline Characteristics for Part A (Safety Population) | 79 |
| Table 14.1.5.2 Baseline Characteristics for Part B (Safety Population) | 80 |
| Table 14.1.5.3 Baseline Characteristics for Part C (Safety Population) | 80 |
| Table 14.1.5.4 Baseline Characteristics for Part D (Safety Population) | 80 |
| Table 14.1.6.1 Primary Cancer History for Part A (Safety Population) | 81 |
| Table 14.1.6.2 Primary Cancer History for Part B (Safety Population) | 82 |
| Table 14.1.6.3 Primary Cancer History for Part C (Safety Population) | 82 |
| Table 14.1.6.4 Primary Cancer History for Part D (Safety Population) | 82 |
| Table 14.1.7.1 Prior Anticancer Treatment for Primary Cancer for Part A (Safety Population) | 83 |
| Table 14.1.7.2 Prior Anticancer Treatment for Primary Cancer for Part B (Safety Population) | 84 |
| Table 14.1.7.3 Prior Anticancer Treatment for Primary Cancer for Part C (Safety Population) | 84 |
| Table 14.1.7.4 Prior Anticancer Treatment for Primary Cancer for Part D (Safety Population) | 84 |
| Table 14.1.8.1 Medical History by System Organ Class and Preferred Term for Part A (Safety Population | |
| Table 14.1.8.2 Medical History by System Organ Class and Preferred Term for Part B (Safety Population | |
| Table 14.1.8.3 Medical History by System Organ Class and Preferred Term for Part C (Safety Population | |
| | 86 |

| Table 14.1.8.4 Medical History by System Organ Class and Preferred Term for Part D (Safety | |
|---|---|
| Table 14.1.9.1 Prior Blood Disorder for Part A (Safety Population) | |
| Table 14.1.9.2 Prior Blood Disorder for Part B (Safety Population) | |
| Table 14.1.9.3 Prior Blood Disorder for Part C (Safety Population) | |
| Table 14.1.9.4 Prior Blood Disorder for Part D (Safety Population) | 88 |
| Table 14.1.10.1 Prior Transfusion and Growth Factor for Part A (Safety Population) | 89 |
| Table 14.1.10.2 Prior Transfusion and Growth Factor for Part B (Safety Population) | 90 |
| Table 14.1.10.3 Prior Transfusion and Growth Factor for Part C (Safety Population) | 90 |
| Table 14.1.10.4 Prior Transfusion and Growth Factor for Part D (Safety Population) | 90 |
| Table 14.1.11.1.1 Prior Non-Anticancer Medication by Anatomical Therapeutic Chemica Preferred Term for Part A (Safety Population) | |
| Table 14.1.11.1.2 Prior Non-Anticancer Medication by Anatomical Therapeutic Chemical Preferred Term for Part B (Safety Population) | |
| Table 14.1.11.1.3 Prior Non-Anticancer Medication by Anatomical Therapeutic Chemical Preferred Term for Part C (Safety Population) | |
| Table 14.1.11.1.4 Prior Non-Anticancer Medication by Anatomical Therapeutic Chemical Preferred Term for Part D (Safety Population) | |
| Table 14.1.11.2.1 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) a Term for Part A (Safety Population) | |
| Table 14.1.11.2.2 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) a Term for Part B (Safety Population) | |
| Table 14.1.11.2.3 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) a Term for Part C (Safety Population) | |
| Table 14.1.11.2.4 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) a Term for Part D (Safety Population) | |
| Table 14.2.1.1.1 Best Overall Response for Part A (Confirmed, Safety Population) | 92 |
| Table 14.2.1.1.2 Best Overall Response for Part B (Confirmed, SafetyPopulation) | 95 |
| Table 14.2.1.1.3 Best Overall Response for Part C (Confirmed, Safety Population) | 95 |
| Table 14.2.1.1.4 Best Overall Response for Part D (Confirmed, Safety Population) | 95 |
| Table 14.2.2.1 Progression Free Survival for Part A (Safety Population) | 96 |
| Table 14.2.2.2 Progression Free Survival for Part B (Safety Population) | 97 |
| Table 14.2.2.3 Progression Free Survival for Part C (Safety Population) | |
| Table 14.2.2.4 Progression Free Survival for Part D (Safety Population) | 97 |

| Figure 14.2.1.1.1 Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part A (Safety Population) |
|---|
| Figure 14.2.1.1.2 Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part B (Safety Population) |
| Figure 14.2.1.1.3 Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part C (SafetyPopulation) |
| Figure 14.2.1.1.4 Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part D (Safety Population) |
| Figure 14.2.1.2.1 Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part A (Safety Population) |
| Figure 14.2.1.2.2 Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part B (Safety Population) |
| Figure 14.2.1.2.3 Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part C (Safety Population) |
| Figure 14.2.1.2.4 Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part D (Safety Population) |
| Figure 14.2.2.1 Kaplan-Meier Plot for Progression Free Survival for Part A (Safety Population)102 |
| Figure 14.2.2.2 Kaplan-Meier Plot for Progression Free Survival for Part B (Safety Population) 102 |
| Figure 14.2.2.3 Kaplan-Meier Plot for Progression Free Survival for Part C (Safety Population) 102 |
| Figure 14.2.2.4 Kaplan-Meier Plot for Progression Free Survival for Part D (Safety Population) 102 |
| Table 14.3.1.1.1 Overall Treatment Emergent Adverse Events Summary for Part A (Safety Population) |
| Table 14.3.1.1.2 Overall Treatment Emergent Adverse Events Summary for Part B (Safety Population) |
| Table 14.3.1.1.3 Overall Treatment Emergent Adverse Events Summary for Part C (Safety Population) |
| Table 14.3.1.1.4 Overall Treatment Emergent Adverse Events Summary for Part D (Safety Population) |
| Table 14.3.1.2.1 Dose-Limiting Toxicity by Preferred Term and Maximum CTCAE Toxicity Grade for Part A ( Safety Population) |
| Table 14.3.1.2.2 Dose-Limiting Toxicity by Preferred Termand Maximum CTCAE Toxicity Grade for Part B (Safety Population) |
| Table 14.3.1.2.3 Dose-Limiting Toxicity by Preferred Termand Maximum CTCAE Toxicity Grade for Part C (Safety Population) |
| Table 14.3.1.2.4 Dose-Limiting Toxicity by Preferred Termand Maximum CTCAE Toxicity Grade for Part D (Safety Population) |

| Table 14.3.1.3.1 Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part A (Safety Population) |
|---|
| Table 14.3.1.3.2 Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part B (Safety Population) |
| Table 14.3.1.3.3 Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part C (Safety Population) |
| Table 14.3.1.3.4 Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.4.1 Treatment Emergent Adverse Events by Preferred Term for Part A (Safety Population) |
| Table 14.3.1.4.2 Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part B (Safety Population) |
| Table 14.3.1.4.3 Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part C (Safety Population) |
| Table 14.3.1.4.4 Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part D (Safety Population) |
| Table 14.3.1.5.1 Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part A (Safety Population) |
| Table 14.3.1.5.2 Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part B Group (Safety Population) |
| Table 14.3.1.5.3.1 Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part C – Result 1 (Safety Population) |
| Table 14.3.1.5.3.2 Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part C - Result 2 (Safety Population) |
| Table 14.3.1.5.4 Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.6.1 Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part A (Safety Population) |
| Table 14.3.1.6.2 Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part B (Safety Population) |
| Table 14.3.1.6.3.1 Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part C – Result 1 (Safety Population) |
| Table 14.3.1.6.3.2 Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part C – Result 2 (Safety Population) |
| Table 14.3.1.6.4 Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part D (Safety Population) |

| Table 14.3.1.7.1 Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade ≥ 3 for Part A (Safety Population) |
|---|
| Table 14.3.1.7.2 Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade ≥ 3 for Part B (Safety Population) |
| Table 14.3.1.7.3 Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade ≥ 3 for Part C (Safety Population) |
| Table 14.3.1.7.4 Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade ≥ 3 for Part D (Safety Population) |
| Table 14.3.1.8.1 Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade ≥ 3 for Part A (Safety Population) |
| Table 14.3.1.8.2 Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade ≥ 3 for Part B (Safety Population)127 |
| Table 14.3.1.8.3.1 Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade ≥ 3 for Part C − Result 1 (Safety Population) |
| Table 14.3.1.8.3.2 Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade ≥ 3 for Part C − Result 2 (Safety Population) |
| Table 14.3.1.8.4 Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade ≥ 3 for Part D (Safety Population) |
| Table 14.3.1.9.1 Serious AEs by System Organ Class and Preferred Term for Part A (Safety Population) |
| Table 14.3.1.9.2 Serious AEs by System Organ Class and Preferred Term for Part B (Safety Population) |
| Table 14.3.1.9.3 Serious AEs by System Organ Class and Preferred Term for Part C (Safety Population) |
| Table 14.3.1.9.4 Serious AEs by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.10.1 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part A (Safety Population) |
| Table 14.3.1.10.2 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part B (Safety Population) |
| Table 14.3.1.10.3.1 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part C – Result 1 (Safety Population) |
| Table 14.3.1.10.3.2 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part C – Result 2 (Safety Population) |
| Table 14.3.1.10.4 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part D (Safety Population) |

TESARO Inc.

| Table 14.3.1.11.1 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part A (Safety Population) |
|---|
| Table 14.3.1.11.2 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part B (Safety Population) |
| Table 14.3.1.11.3 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part C (Safety Population) |
| Table 14.3.1.11.4 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.12.1 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part A (Safety Population) |
| Table 14.3.1.12.2 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part B (Safety Population) |
| Table 14.3.1.12.3.1 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part C – Result 1 (Safety Population) 136 |
| Table 14.3.1.12.3.2 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part C – Result 2 (Safety Population) 136 |
| Table 14.3.1.12.4 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.13.1.1 Treatment Emergent Adverse Events Leading to Niraparib Reduction/Interruption by System Organ Class and Preferred Term for Part A (Safety Population) |
| Table 14.3.1.13.1.2 Treatment Emergent Adverse Events Leading to Niraparib Reduction/Interruption by System Organ Class and Preferred Term for Part C (Safety Population) |
| Table 14.3.1.13.2.1 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part A (Safety Population) |
| Table 14.3.1.13.2.2 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part B (Safety Population) |
| Table 14.3.1.13.2.3 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part C (Safety Population) |
| Table 14.3.1.13.2.4 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.13.3.1 Treatment Emergent Adverse Events Leading to Carboplatin Interruption by System Organ Class and Preferred Term for Part B (Safety Population) |
| Table 14.3.1.13.3.2 Treatment Emergent Adverse Events Leading to Carboplatin Interruption by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.13.4.1 Treatment Emergent Adverse Events Leading to Paclitaxel Interruption by System Organ Class and Preferred Term for Part B (Safety Population) |

| Table 14.3.1.13.4.2 Treatment Emergent Adverse Events Leading to Paclitaxel Interruption by System Organ Class and Preferred Term for Part D (Safety Population) |
|---|
| Table 14.3.1.13.5.1 Treatment Emergent Adverse Events Leading to Bevacizumab Interruption by System Organ Class and Preferred Term for Part C (Safety Population) |
| Table 14.3.1.13.5.2 Treatment Emergent Adverse Events Leading to Bevacizumab Interruption by System Organ Class and Preferred Term for Part D (Safety Population) |
| Table 14.3.1.14.1 Deaths in Part A (Safety Population) |
| Table 14.3.1.14.2 Deaths in Part B (Safety Population) |
| Table 14.3.1.14.3 Deaths in Part C (Safety Population) |
| Table 14.3.1.14.4 Deaths in Part D (Safety Population) |
| Table 14.3.1.15.1 Adverse Events of Special Interest by Preferred Term for Part A (Safety Population)14- |
| Table 14.3.1.15.2 Adverse Events of Special Interest by Preferred Term for Part B (Safety Population)145 |
| Table 14.3.1.15.3 Adverse Events of Special Interest by Preferred Term for Part C (Safety Population)14; |
| Table 14.3.1.15.4 Adverse Events of Special Interest by Preferred Term for Part D (Safety Population)14. |
| Table 14.3.2.2 Listing of Serious Adverse Events (Safety Population) |
| Table 14.3.2.3 Listing of Treatment Emergent Adverse Events Leading to Dose Interruption (Safety Population) |
| Table 14.3.2.4 Listing of Treatment Emergent Adverse Events Leading to Dose Modification (Safety Population) |
| Table 14.3.2.5 Listing of Treatment Emergent Adverse Events Leading to Discontinuation from Treatmen (Safety Population) |
| Table 14.3.4.1 Listing of Abnormal Laboratory Values (Safety Population) |
| Table 14.3.4.2 Listing of Laboratory Values with CTCAE Toxicity Grade ≥ 3 (Safety Population) 149 |
| Table 14.3.4.3 Listing of Clinically Significant Laboratory Values (Safety Population)149 |
| Table 14.3.5.1 Extent of Exposure for Part A (Safety Population) |
| Table 14.3.5.2 Extent of Exposure for Part B (Safety Population) |
| Table 14.3.5.3 Extent of Exposure for Part C (Safety Population) |
| Table 14.3.5.4 Extent of Exposure for Part D (Safety Population) |
| Figure 14.3.5.1 Swimmer Plot of Treatment Duration for Part A (Safety Population) |
| Figure 14.3.5.2 Swimmer Plot of Treatment Duration for Part B (Safety Population) |
| Figure 14.3.5.3 Swimmer Plot of Treatment Duration for Part C (Safety Population) |
| Figure 14.3.5.4 Swimmer Plot of Treatment Duration for Part D (Safety Population)165 |
| Table 14.3.6.1.2 Summary of Actual and Change from Baseline Value for Hematology Parameters for Par B (Safety Population) |

| Table 14.3.6.1.3 Summary of Actual and Change from Baseline Value for Hematology Parameters for Part C (Safety Population) |
|---|
| Table 14.3.6.1.4 Summary of Actual and Change from Baseline Value for Hematology Parameters for Part D (Safety Population) |
| Table 14.3.6.2.1 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part A (Safety Population) |
| Table 14.3.6.2.2 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part B (Safety Population) |
| Table 14.3.6.2.3 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part C (Safety Population) |
| Table 14.3.6.2.4 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part D (Safety Population) |
| Table 14.3.6.3.1 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part A (Safety Population) |
| Table 14.3.6.3.2 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part B (Safety Population) |
| Table 14.3.6.3.3 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part C (Safety Population) |
| Table 14.3.6.3.4 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part D (Safety Population) |
| Table 14.3.6.4.1 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part A (Safety Population) |
| Table 14.3.6.4.2 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part B (Safety Population) |
| Table 14.3.6.4.3 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part C (Safety Population) |
| Table 14.3.6.4.4 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part D (Safety Population) |
| Table 14.3.7.1 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part A (Safety Population) |
| Table 14.3.7.2 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part B (Safety Population) |
| Table 14.3.7.3 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part C (Safety Population) |
| Table 14.3.7.4 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part D (Safety Population) |

| Table 14.3.8.1.1 Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity G for Part A (Safety Population) | |
|---|---|
| Table 14.3.8.1.2 Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity Grad Part B (Safety Population) | |
| Table 14.3.8.1.3 Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity Grad Part C (Safety Population) | |
| Table 14.3.8.1.4 Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity Grad Part D (Safety Population) | |
| Table 14.3.8.2.1 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade Part A (Safety Population) | |
| Table 14.3.8.2.2 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade Part B (Safety Population) | |
| Table 14.3.8.2.3 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade Part C (Safety Population) | |
| Table 14.3.8.2.4 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade Part D (Safety Population) | |
| Table 14.3.9.1.2 Summary of Post-Baseline Liver Function for Part B (Safety Population) | .176 |
| Table 14.3.9.1.3 Summary of Post-Baseline Liver Function for Part C (Safety Population) | .176 |
| Table 14.3.9.1.4 Summary of Post-Baseline Liver Function for Part D (Safety Population) | .176 |
| Table 14.3.10.1.2 Shift of ECOG Performance Status from Baseline to Worst Post-Baseline Score for B (Safety Population) | |
| Table 14.3.10.1.3 Shift of ECOG Performance Status from Baseline to Worst Post-Baseline Score for C (Safety Population) | |
| Table 14.3.10.1.4 Shift of ECOG Performance Status from Baseline to Worst Post-Baseline Score for D (Safety Population) | Part |
| Table 14.3.10.2.1 Notable ECG Values for Part A (Safety Population) | .179 |
| Table 14.3.10.2.2 Notable ECG Values for Part B (Safety Population) | .180 |
| Table 14.3.10.2.3 Notable ECG Values for Part C (Safety Population) | .180 |
| Table 14.3.10.2.4 Notable ECG Values for Part D (Safety Population) | . 180 |
| Listing 16.2.1.2.1 Discontinuation of Treatment Niraparib (Safety Population) | .183 |
| Listing 16.2.1.2.2 Discontinuation of Treatment TSR-042 (Safety Population) | .183 |
| Listing 16.2.1.2.3 Discontinuation of Treatment Bevacizumab (Safety Population) | .183 |
| Listing 16.2.1.2.4 Discontinuation of Carboplatin-Paclitaxel (Safety Population) | .183 |
| Listing 16.2.1.2.5 Discontinuation of Treatment TSR-022 (Safety Population) | .183 |
| Listing 16.2.1.2.6 Discontinuation of Treatment Carboplatin (Safety Population) | .183 |

| Protocol | No: | 3000- | .01_ | 002 |
|--------------|------|---------------|------|-----|
| 1 1 0 10 101 | 11U. | <b>JUUU</b> - | UI- | UUZ |

| Listing 16.2.1.2.7 Discontinuation of Treatment Pemetrexed (Safety Population) | 183 |
|---|---|
| Listing 16.2.1.3 Discontinuation from Study (Safety Population) | 184 |
| Listing 16.2.2 Protocol Deviation by Category and Severity (All Patients Population) | 185 |
| Listing 16.2.3 Patients Excluded Due to Eligibility (All Patients Population) | 186 |
| Listing 16.2.4.1 Demographics (Safety Population) | 187 |
| Listing 16.2.4.2 Medical History (Safety Population) | 188 |
| Listing 16.2.4.3 Surgical History (Safety Population) | 189 |
| Listing 16.2.4.4 Previous Radiotherapy (Safety Population) | 190 |
| Listing 16.2.4.5 Concomitant Radiotherapy (Safety Population) | 191 |
| Listing 16.2.4.6 Prior Transfusions and Growth Factors (Safety Population) | 192 |
| Listing 16.2.4.7 Concomitant Transfusion (Safety Population) | 193 |
| Listing 16.2.4.8 Concomitant Growth Factors (Safety Population) | 194 |
| Listing 16.2.4.9 Prior Blood Disorders (Safety Population) | 195 |
| Listing 16.2.4.10 Prior Anticancer Treatment for Primary Cancer (Safety Population) | 196 |
| Listing 16.2.4.11 Primary Cancer History (Safety Population) | 197 |
| Listing 16.2.4.12 HBsAg and HCV Testing at Baseline (Safety Population) | 198 |
| Listing 16.2.5.1 Prior and Concomitant Medication/Therapy (Safety Population) | 199 |
| Listing 16.2.5.2 Concomitant Procedures (Safety Population) | 200 |
| Listing 16.2.5.3 Niraparib First Dose (Safety Population) | 201 |
| Listing 16.2.5.4 Niraparib Dose Modification (Safety Population) | 202 |
| Listing 16.2.5.5 Niraparib Administration (Safety Population) | 203 |
| Listing 16.2.5.6 | 204 |
| TSR-042 Administration (Safety Population) | 204 |
| Listing 16.2.5.7 Carboplatin Administration (Safety Population) | 205 |
| Listing 16.2.5.8 | 207 |
| Paclitaxel Administration (Safety Population) | 207 |
| Listing 16.2.5.9 Pemetrexed Administration (Safety Population) | 207 |
| Listing 16.2.5.11 Bevacizumab Administration (Safety Population) | 208 |
| Listing 16.2.5.12 TSR-022 Administration (Safety Population) | 209 |
| Listing 16.2.5.14 Pemetrexed Supplemental Medications (Safety Population) | 211 |
| Listing 16.2.6.1 Tumor Target Lesion Assessment (Safety Population) | 212 |
| Listing 16.2.6.2 Tumor Non-Target Lesion Assessment (Safety Population) | 213 |

Table 14.1.1 Overview of Patients Enrollment

| | | All | G C 4 |
|------------|------------|------------------------|----------------------|
| Treatment | Statistics | Patients<br>Population | Safety<br>Population |
| Not Dosed | n | XX | XX |
| Part A | n | XX | XX |
| Part A-200 | n | XX | XX |
| Part A-300 | n | XX | XX |
| Part B | n | XX | XX |
| - | | | |
| Part C | n | XX | XX |
| Part C-200 | n | XX | XX |
| Part C-300 | n | XX | XX |
| Part D | n | XX | XX |
| Part E | n | XX | XX |
| Part F | n | XX | XX |
| Part F-300 | n | XX | XX |
| Part F-900 | n | XX | XX |
| Overall | n | XX | XX |

Source: Listing 16.2.1.1

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment

TESARO Inc.

Protocol No: 3000-01-002 Dated

Table 14.1.2.1
Patients Disposition for Part A (Safety Population)

| Parameter | | a | Part A-200 | Part A-300 | Overall |
|---|---|---|---|---|---|
| Primary Reason for Discontinuations from Study Image: Consent of the Consent of Cons | Parameter | Statistics | (N=XX) | (N=XX) | (N=XX) |
| Withdrawal of consent | Discontinued from Study | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal of consent | Primary Reason for Discontinuations from Study | | | | |
| Lost to follow-up | · | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | Lost to follow-up | ` ' | , | , , | |
| Sponsor decision to terminate study | Death | | | | |
| Investigator decision | Sponsor decision to terminate study | | | | |
| Discontinued from Niraparib Adverse event A | | | | | |
| Primary Reason for Discontinuation from Niraparib Adverse event Risk to patient as judged by investigator and/or sponsor and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 Adverse event Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient prediction from TSR-042 n (%) xx ( | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary Reason for Discontinuation from Niraparib Adverse event Risk to patient as judged by investigator and/or sponsor and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 Adverse event Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient prediction from TSR-042 n (%) xx ( | | | | | |
| Adverse event Risk to patient as judged by investigator and/or sponsor Risk to patient as judged by investigator and/or sponsor Risk to patient as judged by investigator and/or sponsor Risk to patient as judged by investigator Risk to patient as judged by investigator Risk to patient as judged by investigator Risk to patient as judged by investigator Risk to patient sponsor Risk to patient as judged by investigator Risk to patient sponsor Risk to patient sponsor Risk to patient sponsor Risk to patient sponsor decision to terminate study Risk to patient sponsor Risk to patient sponsor Risk to patient sponsor Risk to patient sponsor to protocol as judged by investigator Risk to patient as judged by investigator and/or sponsor Risk to patient sponsor Risk to pa | Discontinued from Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Primary Reason for Discontinuation from TSR-042 Adverse event n (%) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | Primary Reason for Discontinuation from Niraparib | | | | |
| Severe noncompliance to protocol as judged by investigator and/or sponsor | Adverse event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| and/or sponsor Patient request Patient request Patient request Patient becomes pregnancy Patient Patient Patient Patient P | Risk to patient as judged by investigator and/or sponsor | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient request Patient request Patient becomes pregnancy Patient pecusion to terminate study Patient becomes pregnancy Patient request Patient reques | Severe noncompliance to protocol as judged by investigator | | | | |
| Patient becomes pregnancy Sponsor decision to terminate study Sponsor decision to terminate study Disease progression per RECIST 1.1 Disease progression based on clinical criteria by Investigator Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR Other n (%) xx (xx.x) Discontinued from TSR-042 n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Primary Reason for Discontinuation from TSR-042 Adverse event Aisk to patient as judged by investigator and/or sponsor Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) | | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sponsor decision to terminate study Disease progression per RECIST 1.1 Disease progression based on clinical criteria by Investigator Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR Other n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 Primary Reason for Discontinuation from TSR-042 Adverse event n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy xp (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression per RECIST 1.1 Disease progression based on clinical criteria by Investigator Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR Other | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) Other n (%) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Primary Reason for Discontinuation from TSR-042 Adverse event n (%) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | | . , | xx (xx.x) | , , | |
| Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) Other n (%) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Primary Reason for Discontinuation from TSR-042 Adverse event n (%) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) Other n (%) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Primary Reason for Discontinuation from TSR-042 Adverse event n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other n (%) xx (xx.x) xx (xx.x) xx (xx.x) Discontinued from TSR-042 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Primary Reason for Discontinuation from TSR-042 Adverse event n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | | | | | |
| Discontinued from TSR-042 Primary Reason for Discontinuation from TSR-042 Adverse event Risk to patient as judged by investigator and/or sponsor and/or sponsor and/or sponsor n (%) xx (xx.x) Disease progression to terminate study n (%) xx (xx.x) | with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary Reason for Discontinuation from TSR-042 Adverse event n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator n (%) Risk (xx.x) Risk (xx. | Discontinued from TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator and/or sponsor n (%) Risk to patient as judged by investigator n (%) Risk (xx.x) Risk (xx. | Division Division for Division from TCD 042 | | | | |
| Risk to patient as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) | • | m (0/) | () | () | () |
| Severe noncompliance to protocol as judged by investigator and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) | | | | ` ' | . , |
| and/or sponsor n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) xx (xx.x) | | 11 (70) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Patient request n (%) xx (xx.x) xx (xx.x) xx (xx.x) Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) | | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Patient becomes pregnancy n (%) xx (xx.x) xx (xx.x) xx (xx.x) Sponsor decision to terminate study n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) | | | ` ′ | ` ′ | ` ′ |
| Sponsor decision to terminate study Disease progression per RECIST 1.1 Disease progression based on clinical criteria by Investigator Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) | | | | | |
| Disease progression per RECIST 1.1 n (%) xx (xx.x) xx (xx.x) xx (xx.x) Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) | | ` ' | ` / | , , | ` ′ |
| Disease progression based on clinical criteria by Investigator n (%) xx (xx.x) xx (xx.x) xx (xx.x) Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) | | ` ' | ` ′ | ` ′ | . , |
| Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR n (%) xx (xx.x) xx (xx.x) xx (xx.x) | | | ` ' | ` ′ | |
| with study treatment, and have at least 2 cycles beyond initial CR $n$ (%) $xx$ (xx.x) $xx$ (xx.x) $xx$ (xx.x) $xx$ (xx.x) | | (/ ") | () | () | () |
| | | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | ` , | ` ′ | ` ′ |

Source: Listing 16.2.1.2.1 Listing 16.2.1.2.2 Listing 16.2.1.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

TESARO Inc.

Table 14.1.2.2
Patients Disposition for Part B (Safety Population)

| Parameter | Statistics | Part B (N=XX) |
|---|---|---|
| Discontinued from Study | n (%) | xx (xx.x) |
| Primary Reason for Discontinuations from Study | | |
| Withdrawal of consent | n (%) | xx (xx.x) |
| Lost to follow-up | n (%) | xx (xx.x) |
| Death | n (%) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) |
| Investigator decision | n (%) | xx (xx.x) |
| Other | n (%) | xx (xx.x) |
| Discontinued from Carboplatin/Paclitaxel | n (%) | xx (xx.x) |
| Primary Reason for Discontinuation from carboplatin-paclitaxel | | |
| Adverse event | n (%) | xx (xx.x) |
| Risk to patient as judged by investigator and/or sponsor | n (%) | xx (xx.x) |
| Severe noncompliance to protocol as judged by investigator | | |
| and/or sponsor | n (%) | xx (xx.x) |
| Patient request | n (%) | xx(xx.x) |
| Patient becomes pregnancy | n (%) | xx(xx.x) |
| Sponsor decision to terminate study | n (%) | xx(xx.x) |
| Disease progression per RECIST 1.1 | n (%) | xx (xx.x) |
| Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) |
| Confirmed Complete Response, treated for at least 24 weeks | | |
| with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) |
| Other | n (%) | xx (xx.x) |
| Discontinued from TSR-042 | n (%) | xx (xx.x) |
| Primary Reason for Discontinuation from TSR-042 | | |
| Adverse event | n (%) | xx (xx.x) |
| Risk to patient as judged by investigator and/or sponsor<br>Severe noncompliance to protocol as judged by investigator | n (%) | xx (xx.x) |
| and/or sponsor | n (%) | xx (xx.x) |
| Patient request | n (%) | xx (xx.x) |
| Patient becomes pregnancy | n (%) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) |
| Disease progression per RECIST 1.1 | n (%) | xx (xx.x) |
| Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) |
| Confirmed Complete Response, treated for at least 24 weeks | | |
| with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) |
| Other | n (%) | xx (xx.x) |

Source: Listing 16.2.1.2.2 Listing 16.2.1.2.4 Listing 16.2.1.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

TESARO Inc.

Table 14.1.2.3
Patients Disposition for Part C (Safety Population)

| | a | Part C-200 | Part C-300 | Overall |
|---|---|---|---|---|
| Parameter | Statistics | (N=XX) | (N=XX) | (N=XX) |
| Discontinued from Study | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary Reason for Discontinuations from Study | | | | |
| Withdrawal of consent | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator decision | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary Reason for Discontinuation from Niraparib | | | | |
| Adverse event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Risk to patient as judged by investigator and/or sponsor | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Severe noncompliance to protocol as judged by investigator | | | | |
| and/or sponsor | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient request | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient becomes pregnancy | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression per RECIST 1.1 | n (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression based on clinical criteria by Investigator | n (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Confirmed Complete Response, treated for at least 24 weeks | (0/) | ( ) | ( ) | ( ) |
| with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary Reason for Discontinuation from TSR-042 | | | | |
| Adverse event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Risk to patient as judged by investigator and/or sponsor | n (%) | xx(xx.x) | xx (xx.x) | xx (xx.x) |
| Severe noncompliance to protocol as judged by investigator and/or sponsor | n (%) | vv (vv v) | vv (vv v) | vv (vv v) |
| • | | XX (XX.X) | xx (xx.x) | xx (xx.x) |
| Patient request Patient becomes pregnancy | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| * * * | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sponsor decision to terminate study Disease progression per RECIST 1.1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression per RECIST 1.1 Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| , , | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued from Bevacizumab | n (%) | xx (xx.x) | xx (xx.x) | n (%) |

| Primary Reason for Discontinuation from Bevacizumab | | | | |
|---|---|---|---|---|
| Adverse event | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Risk to patient as judged by investigator and/or sponsor | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Severe noncompliance to protocol as judged by investigator | | | | |
| and/or sponsor | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Patient request | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Patient becomes pregnant | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Disease progression per RECIST 1.1 | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Confirmed Complete Response, treated for at least 24 weeks | | | | |
| with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Completed Course | n (%) | xx (xx.x) | xx (xx.x) | n (%) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | n (%) |


Source: Listing 16.2.1.2.1 Listing 16.2.1.2.2 Listing 16.2.1.2.3 Listing 16.2.1.3

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment
TESARO Inc.

Table 14.1.2.4
Patients Disposition for Part D (Safety Population)

| Parameter | Statistics | Part D (N=XX) |
|---|---|---|
| Discontinued from Study | n (%) | xx (xx.x) |
| Primary Reason for Discontinuations from Study | | |
| Withdrawal of consent | n (%) | xx (xx.x) |
| Lost to follow-up | n (%) | xx (xx.x) |
| Death | n (%) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) |
| Investigator decision | n (%) | xx (xx.x) |
| Other | n (%) | xx (xx.x) |
| Discontinued from Carboplatin/Paclitaxel | n (%) | xx (xx.x) |
| Primary Reason for Discontinuation from Carboplatin-paclitaxel | | |
| Adverse event | n (%) | xx (xx.x) |
| Risk to patient as judged by investigator and/or sponsor<br>Severe noncompliance to protocol as judged by investigator | n (%) | xx (xx.x) |
| and/or sponsor | n (%) | xx (xx.x) |
| Patient request | n (%) | xx (xx.x) |
| Patient becomes pregnancy | n (%) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) |
| Disease progression per RECIST 1.1 | n (%) | xx (xx.x) |
| Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) |
| Confirmed Complete Response, treated for at least 24 weeks | | |
| with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) |
| Completed Course | n (%) | xx (xx.x) |
| Other | n (%) | xx (xx.x) |
| Discontinued from TSR-042 | n (%) | xx (xx.x) |
| Primary Reason for Discontinuation from TSR-042 | | |
| Adverse event | n (%) | xx (xx.x) |
| Risk to patient as judged by investigator and/or sponsor<br>Severe noncompliance to protocol as judged by investigator | n (%) | xx (xx.x) |
| and/or sponsor | n (%) | xx (xx.x) |
| Patient request | n (%) | xx (xx.x) |
| Patient becomes pregnancy | n (%) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) |
| Disease progression per RECIST 1.1 | n (%) | xx (xx.x) |
| Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) |
| Confirmed Complete Response, treated for at least 24 weeks with study treatment, and have at least 2 cycles beyond initial CR Other | n (%) | xx (xx.x) |
| Discontinued from Bevacizumab | n (%) | xx (xx.x) |
| Primary Reason for Discontinuation from Bevacizumab | | |
| | n (0/1) | vv (vv v) |
| Adverse event | n (%) | xx (xx.x) |


| and/or sponsor | n (%) | xx (xx.x) |
|---|---|---|
| Patient request | n (%) | xx (xx.x) |
| Patient becomes pregnancy | n (%) | xx (xx.x) |
| Sponsor decision to terminate study | n (%) | xx (xx.x) |
| Disease progression per RECIST 1.1 | n (%) | xx (xx.x) |
| Disease progression based on clinical criteria by Investigator | n (%) | xx (xx.x) |
| Confirmed Complete Response, treated for at least 24 weeks | | |
| with study treatment, and have at least 2 cycles beyond initial CR | n (%) | xx (xx.x) |
| Completed Course | n (%) | xx (xx.x) |
| Other | n (%) | xx (xx.x) |

Source: Listing 16.2.1.2.2 Listing 16.2.1.2.3 Listing 16.2.1.2.4 Listing 16.2.1.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Table 14.1.3.1
Protocol Deviation by Category and Severity for Part A (Safety Population)

| Parameter | Statistics | Part A-200 (N=XX) | Part A-300 (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Patients with any Protocol Deviation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | (0.4) | | | |
| Important Deviation | n (%) | xx (xx.x) | xx (xx.x) | xx(xx.x) |
| Category 1 | n (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Category 2 | n (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Category 3 | n (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| ••• | | | | |
| Significant Deviation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Category 1 | n (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Category 2 | n (%) | xx(xx.x) | xx(xx.x) | xx (xx.x) |
| Category 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.2

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

## Repeat for Table 14.1.3.1 for

Table 14.1.3.2 Protocol Deviation by Category and Severity for Part B (Safety Population)

Table 14.1.3.3 Protocol Deviation by Category and Severity for Part C (Safety Population)

Table 14.1.3.4 Protocol Deviation by Category and Severity for Part D (Safety Population)

Table 14.1.4.1

Demographic Characteristics for Part A (Safety Population)

| Characteristics | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Age (years) | | | | , |
| | n | xx | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Age Category | | | | |
| 18-64 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 65-74 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Liver | | | | |
| ≥ 75 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sex | | | | |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | | |
| Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race | | | | |
| American Indian or Alaska Native | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| White | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.4.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

TESARO Inc. **Protocol No: 3000-01-002** 

Repeat for Table 14.1.4.1 for

Table 14.1.4.2 Demographic Characteristics for Part B (Safety Population)

Table 14.1.4.3 Demographic Characteristics for Part C (Safety Population)

Table 14.1.4.4 Demographic Characteristics for Part D (Safety Population)

Table 14.1.5.1
Baseline Characteristics for Part A (Safety Population)

| Parameter | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Height (cm) | n | xx | xx | xx |
| - , , | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Weight (kg) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| BMI (kg/m²) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| BSA (m²) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| ECOG performance status | | | | |
| 0 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.9 Listing 16.2.10

Note: BMI=Body Mass Index; BSA = Body Surface Area

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Repeat Table 14.1.5.1 for

Table 14.1.5.2 Baseline Characteristics for Part B (Safety Population)

Table 14.1.5.3 Baseline Characteristics for Part C (Safety Population)

Table 14.1.5.4 Baseline Characteristics for Part D (Safety Population)

Table 14.1.6.1 Primary Cancer History for Part A (Safety Population)

| | | Part A-200 | Part A-300 | Overall |
|---|---|---|---|---|
| Parameter | Statistics | (N=XX) | (N=XX) | (N=XX) |
| Primary tumor site at first diagnosis | | | | |
| Brain | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Breast | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Cancer stage at first diagnosis | | | | |
| Stage I | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Stage I A | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Stage I B | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Stage I C | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Stage II | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ••• | | | | |
| Stage III | n (%) | xxx(xx.x) | xxx(xx.x) | xxx (xx.x) |
| Ctage IV | m (0/) | () | | () |
| Stage IV | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Unknown | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Time from first diagnosis to first dose of | | | | |
| study treatment (months) [1] | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Cancer stage at most recent diagnosis | | | | |
| Stage I | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Stage II | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Stage III | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Stage IV | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Unknown | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

<sup>[1]</sup> Time from first diagnosis to first dose of study treatment (months) = (first dose date – first diagnosis

date + 1)/30.4375

TESARO Inc.

Source: Listing 16.2.4.11

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment


Repeat Table 14.1.6.1 for

Table 14.1.6.2 Primary Cancer History for Part B (Safety Population)

Table 14.1.6.3 Primary Cancer History for Part C (Safety Population)

Table 14.1.6.4 Primary Cancer History for Part D (Safety Population)

Table 14.1.7.1
Prior Anticancer Treatment for Primary Cancer for Part A (Safety Population)

| Parameter | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Number of Prior Regimens | n | XX | xx | XX |
| · · | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Reason for administration of last treatment | | | | |
| Neoadjuvant | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adjuvant | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Advanced/Metastatic | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Best Response during last treatment | | | | |
| Complete Response (CR) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Partial Response (PR) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stable Disease (SD) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Progressive Disease (PD) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Evaluable | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for discontinuation of last treatment | | | | |
| Toxicity | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed planned courses | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Disease progression | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time from end of last treatment to first dose | | | | |
| of study treatment (months) [1] | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Prior Surgery Related to Cancer | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Radiotherapy Prior to Informed Content | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> Time from end of last treatment to first dose of study treatment (months) = (first dose date - last date of last treatment + 1)/30.4375.

Source: Listing 16.2.4.3 Listing 16.2.4.4 Listing 16.2.4.10

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

TESARO Inc.


Repeat Table 14.1.7.1 for

Table 14.1.7.2 Prior Anticancer Treatment for Primary Cancer for Part B (Safety Population)

Table 14.1.7.3 Prior Anticancer Treatment for Primary Cancer for Part C (Safety Population)

Table 14.1.7.4 Prior Anticancer Treatment for Primary Cancer for Part D (Safety Population)

Table 14.1.8.1 Medical History by System Organ Class and Preferred Term for Part A (Safety Population)

| System Organ Class | | | | |
|---|---|---|---|---|
| Preferred Term | Statistics | Part A-200 (N=XX) | Part A-300 (N=XX) | Overall (N=XX) |
| SOC 1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PT1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PT2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PT3 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| SOC 2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PT1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx(xx.x) |
| PT2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PT3 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Note: Patients who report multiple occurrences of the same condition (preferred term) are included only once per SOC and preferred term

Source: Listing 16.2.4.2

For programmer: add following footnotes

Repeat Table 14.1.8.1 for

Table 14.1.8.2 Medical History by System Organ Class and Preferred Term for Part B (Safety Population)

Table 14.1.8.3 Medical History by System Organ Class and Preferred Term for Part C (Safety Population)

Table 14.1.8.4 Medical History by System Organ Class and Preferred Term for Part D (Safety Population)

Table 14.1.9.1
Prior Blood Disorder for Part A (Safety Population)

| Event | | | | |
|---|---|---|---|---|
| Grade | Statistic | Part A-200 (N=XX) | Part A-300 (N=XX) | Overall (N=XX) |
| Any blood disorder | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Thrombocytopenia | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Leukopenia | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anemia | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Neutropenia | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 14.2.4.9

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Repeat Table 14.1.9.1 for

Table 14.1.9.2 Prior Blood Disorder for Part B (Safety Population)

Table 14.1.9.3 Prior Blood Disorder for Part C (Safety Population)

Table 14.1.9.4 Prior Blood Disorder for Part D (Safety Population)

Table 14.1.10.1
Prior Transfusion and Growth Factor for Part A (Safety Population)

| Administration Type | Statistic | Part A-200 (N= | =XX) Part A-300 (N= | XX) Overall (N=XX) |
|---|---|---|---|---|
| Transfusion | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Red Blood Cells | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Platelets | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Erythropoietin | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Others | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Growth Factor | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Granulocyte colony stimulating factor granulocyte | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Macrophage colony stim factor | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Others | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.4.6

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

## Repeat Table 14.1.10.1 for

Table 14.1.10.2 Prior Transfusion and Growth Factor for Part B (Safety Population)

Table 14.1.10.3 Prior Transfusion and Growth Factor for Part C (Safety Population)

Table 14.1.10.4 Prior Transfusion and Growth Factor for Part D (Safety Population)

Table 14.1.11.1.1
Prior Non-Anticancer Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part A (Safety Population)

| ATC Level 3 | | | | |
|-----------------------|-----------|------------|------------|------------|
| | | Part A-200 | Part A-300 | Overall |
| Preferred Term | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Any Prior Medications | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ATC Level 3 | | | | |
| PT1 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PT2 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| PT3 | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| ••• | | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.5.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Repeat for Table 14.1.11.1.1

Table 14.1.11.1.2 Prior Non-Anticancer Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part B (Safety Population)

Table 14.1.11.1.3 Prior Non-Anticancer Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part C (Safety Population)

Table 14.1.11.1.4 Prior Non-Anticancer Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part D (Safety Population)

TESARO Inc.

Repeat for Table 14.1.11.1.1

Table 14.1.11.2.1 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part A (Safety Population)

Table 14.1.11.2.2 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part B (Safety Population)

Table 14.1.11.2.3 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part C (Safety Population)

Table 14.1.11.2.4 Concomitant Medication by Anatomical Therapeutic Chemical (ATC) and Preferred Term for Part D (Safety Population)

TESARO Inc.

Table 14.2.1.1.1
Best Overall Response for Part A (Confirmed, Safety Population)

| | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| D. O. U.B. J. DEGIGT 11 | | | | |
| Best Overall Response by RECIST v1.1 | (0/) | | | ( ) |
| Confirmed Complete Response | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Confirmed Partial Response | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Stable Disease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Progressive Disease | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Evaluable | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Done | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Objective Response Rate (ORR) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 90% CI | XX.X, XX.X | XX.X, XX.X | xx.x, xx.x |
| Duration of Response | | | | |
| Median in Months (range) | | x.x(xx.x, xx.x) | x.x(xx.x, xx.x) | x.x(xx.x, xx.x) |
| Response Ongoing | n (%) | XX | XX | XX |
| Disease Control Rate (DCR) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | 90% CI | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |

Objective Response is defined as overall response as confirmed complete response (CR) or partial response (PR) CI: Confidence Interval. Response Ongoing: All responders who have not yet died or progressed (including clinical progression), denominator for percentage is number of responders.

Source: Listing 16.2.6.4 Listing 16.2.6.5.2

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

# TESARO Inc.


Repeat Table 14.2.1.1.1 for

Table 14.2.1.1.2 Best Overall Response for Part B (Confirmed, SafetyPopulation)

Table 14.2.1.1.3 Best Overall Response for Part C (Confirmed, Safety Population)

Table 14.2.1.1.4 Best Overall Response for Part D (Confirmed, Safety Population)

Table 14.2.2.1 Progression Free Survival for Part A (Safety Population)

| Assessment | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Number of Patients | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Events | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Censored Patients | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Progression Free Survival (months) | | | | |
| | 25 Percentile | XX.X | XX.X | XX.X |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | 50 Percentile | XX.X | XX.X | xx.x |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | 75 Percentile | XX.X | XX.X | XX.X |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Survival Distribution Function (SDF) | | | | |
| 6 months | SDF | XX.X | XX.X | XX.X |
| | 95% CI | XX.X, XX.X | xx.x, xx.x | xx.x, xx.x |
| 12 months | SDF | XX.X | xx.x | XX.X |
| | 95% CI | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |

Note: Progression Free Survival is defined as the date of first dose to the date of disease progression or death due to any cause, whichever occurs earlier.

CI: Confidence Interval

Source: Listing 16.2.6.4 Listing 16.2.6.5.2 Listing 16.2.6.16

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Repeat Table 14.2.2.1 for

Table 14.2.2.2 Progression Free Survival for Part B (Safety Population)

Table 14.2.2.3 Progression Free Survival for Part C (Safety Population)

Table 14.2.2.4 Progression Free Survival for Part D (Safety Population)

Figure 14.2.1.1.1
Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part A (Safety Population)

An Example:



Source: Listing 16.2.6.1

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Repeat Figure 14.2.1.1.1 for

Figure 14.2.1.1.2 Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part B (Safety Population)

Figure 14.2.1.1.3 Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part C (SafetyPopulation)

Figure 14.2.1.1.4 Spider Plot of Percentage Change from Baseline in Target Lesion Size Over Time for Part D (Safety Population)

Figure 14.2.1.2.1

Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part A (Safety Population)

An Example:



Source: Listing 16.2.6.1

#### Repeat for

Figure 14.2.1.2.2 Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part B (Safety Population)

Figure 14.2.1.2.3 Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part C (Safety Population)

Figure 14.2.1.2.4 Waterfall Plot of Best Percentage Change from Baseline in Target Lesion Size for Part D (Safety Population)

### For programmer: add following footnotes as applicable to each output

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Figure 14.2.2.1
Kaplan-Meier Plot for Progression Free Survival for Part A (Safety Population)

#### An Example:





This is an example of KM plot with 90% CI. For Part A, KM plot includes PFS curve for Part A-200, Part A-300 and Part A overall. Do similar plot for Part C.

Source: Listing 16.2.6.4 Listing 16.2.6.5.1 Listing 16.2.6.5.2 Listing 16.2.6.16

PROGRAM NAME: DATE: DDMMYYYY

#### Repeat for

Figure 14.2.2.2 Kaplan-Meier Plot for Progression Free Survival for Part B (Safety Population)

Figure 14.2.2.3 Kaplan-Meier Plot for Progression Free Survival for Part C (Safety Population)

Figure 14.2.2.4 Kaplan-Meier Plot for Progression Free Survival for Part D (Safety Population)

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Statistical Analysis Plan **Dated:18SEP2020** 

TESARO Inc. Protocol No: 3000-01-002

Table 14.3.1.1.1 Overall Treatment Emergent Adverse Events Summary for Part A (Safety Population)

| Characteristic | Statistic | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Treatment Emergent Adverse Event (TEAE) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dose-Limiting Toxicities (DLTs) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to both drugs | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CTCAE Grade ≥ 3 TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related CTCAE Grade ≥ 3 TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to both drugs | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AE (SAE) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related SAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to both drugs | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Dose Reduction/Interruption | | | | |
| TEAE Leading to Niraparib Dose Reduction | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Niraparib Dose Interruption | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to TSR-042 Infusion Interruption | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to TSR-042 Infusion Delayed | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Treatment Discontinuation | | | | |
| TEAEs Leading to Niraparib Discontinuation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Leading to TSR-042 Discontinuation TEAE Leading to Discontinuation of Both | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Drugs | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Leading to Death | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

TESARO Inc.


 ${\it Table~14.3.1.1.2}$  Overall Treatment Emergent Adverse Events Summary for Part B (Safety Population)

| Characteristic | Statistic | Part B (N=XX) |
|---|---|---|
| Treatment Emergent Adverse Event (TEAE) | n (%) | xx (xx.x) |
| Dose-Limiting Toxicities (DLTs) | n (%) | xx (xx.x) |
| Related to TEAE | n (%) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx(xx.x) |
| Related to Carboplatin | n (%) | xx(xx.x) |
| Related to Paclitaxel | n (%) | xx (xx.x) |
| CTCAE Grade ≥ 3 TEAE | n (%) | xx (xx.x) |
| Related CTCAE Grade ≥ 3 TEAE | n (%) | xx(xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) |
| Related to Carboplatin | n (%) | xx (xx.x) |
| Related to Paclitaxel | n (%) | xx (xx.x) |
| Serious AE (SAE) | n (%) | xx (xx.x) |
| Related SAE | n (%) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) |
| Related to Carboplatin | n (%) | xx (xx.x) |
| Related to Paclitaxel | n (%) | xx (xx.x) |
| TEAE Leading to Infusion Interruption/Delayed | | |
| TEAE Leading to TSR-042 Infusion Interruption | n (%) | xx (xx.x) |
| TEAE Leading to TSR-042 Infusion Delayed | n (%) | xx (xx.x) |
| TEAE Leading to Carboplatin Infusion Interruption | n (%) | xx (xx.x) |
| TEAE Leading to Carboplatin Infusion Delayed | n (%) | xx (xx.x) |
| TEAE Leading to Paclitaxel Infusion Interruption | n (%) | xx (xx.x) |
| TEAE Leading to Paclitaxel Infusion Delayed | n ( %) | xx (xx.x) |
| TEAE Leading to Treatment Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to TSR-042 Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to Carboplatin Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to Paclitaxel Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to Death | n (%) | xx (xx.x) |

Source: Listing 16.2.7.2

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Statistical Analysis Plan **Dated:18SEP2020** 

TESARO Inc.

Table 14.3.1.1.3

Overall Treatment Emergent Adverse Events Summary for Part C (Safety Population)

| | | Part C-200 | Part C-300 | Overall |
|---|---|---|---|---|
| Characteristic | Statistic | (N=XX) | (N=XX) | (N=XX) |
| Treatment Emergent Adverse Event (TEAE) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Dose-Limiting Toxicities (DLTs) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Bevacizumab | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| CTCAE Grade ≥ 3 TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related CTCAE Grade ≥ 3 TEAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Bevacizumab | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AE (SAE) | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related SAE | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Niraparib | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Related to Bevacizumab | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Dose Reduction/ Interruption | | | | |
| TEAE Leading to Niraparib Dose Reduction | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Niraparib Dose Interruption | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to TSR-042 Infusion Interruption | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to TSR-042 Infusion Delayed | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Bevacizumab Infusion Interruption | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Bevacizumab Infusion Delayed | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAE Leading to Treatment Discontinuation | | | | |
| TEAEs Leading to Niraparib Discontinuation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Leading to TSR-042 Discontinuation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Leading to Bevacizumab Discontinuation | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| TEAEs Leading to Death | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

TESARO Inc.


Table 14.3.1.1.4

Overall Treatment Emergent Adverse Events Summary for Part D (Safety Population)

| Characteristic | Statistic | Part D (N=XX) |
|---|---|---|
| Treatment Emergent Adverse Event (TEAE) | n (%) | xx (xx.x) |
| Dose-Limiting Toxicities (DLTs) | n (%) | xx (xx.x) |
| Related to TEAE | n (%) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) |
| Related to Carboplatin | n (%) | xx (xx.x) |
| Related to Paclitaxel | n (%) | xx (xx.x) |
| Related to Bevacizumab | n (%) | xx (xx.x) |
| CTCAE Grade ≥ 3 TEAE | n (%) | xx (xx.x) |
| Related CTCAE Grade ≥ 3 TEAE | n (%) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) |
| Related to Carboplatin | n (%) | xx (xx.x) |
| Related to Paclitaxel | n (%) | xx (xx.x) |
| Related to Bevacizumab | n (%) | xx (xx.x) |
| Serious AE (SAE) | | |
| Related SAE | n (%) | xx (xx.x) |
| Related to TSR-042 | n (%) | xx (xx.x) |
| Related to Carboplatin | n (%) | xx (xx.x) |
| Related to Paclitaxel | n (%) | xx (xx.x) |
| Related to Bevacizumab | n (%) | xx (xx.x) |
| TEAE Leading to Infusion Interruption/Delayed | | |
| TEAE Leading to TSR-042 Infusion Interruption | n (%) | xx (xx.x) |
| TEAE Leading to TSR-042 Infusion Delayed | n (%) | xx (xx.x) |
| TEAE Leading to Carboplatin Infusion Interruption | n (%) | xx (xx.x) |
| TEAE Leading to Carboplatin Infusion Delayed | n (%) | xx (xx.x) |
| TEAE Leading to Paclitaxel Infusion Interruption | n (%) | xx (xx.x) |
| TEAE Leading to Paclitaxel Infusion Delayed | n (%) | xx (xx.x) |
| TEAE Leading to Bevacizumab Infusion Interruption | n (%) | xx (xx.x) |
| TEAE Leading to Bevacizumab Infusion Delayed | n (%) | xx (xx.x) |
| TEAE Leading to Treatment Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to TSR-042 Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to Carboplatin Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to Paclitaxel Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to Bevacizumab Discontinuation | n (%) | xx (xx.x) |
| TEAEs Leading to Death | n (%) | xx (xx.x) |

Source: Listing 16.2.7.4

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Table 14.3.1.2.1

Dose-Limiting Toxicity by Preferred Term and Maximum CTCAE Toxicity Grade for Part A ( Safety Population)

| Preferred Term | Maximum Statistic CTCAE Co | Part A-200 | Part A-300 | Overall (N-VV) |
|---|---|---|---|---|
| | Statistic CTCAE Gra | | (N=XX) | (N=XX) |
| Any dose-limiting toxicity | n (%) | n (%) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) Grade 1 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 2 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 3 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 4 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 5 | n (%) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) Grade 1 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 2 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 3 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 4 | n (%) | xx (xx.x) | xx (xx.x) |
| | n (%) Grade 5 | n (%) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes
Repeat Table 14.3.1.2.1 for

Table 14.3.1.2.2 Dose-Limiting Toxicity by Preferred Termand Maximum CTCAE Toxicity Grade for Part B (Safety Population)

Table 14.3.1.2.3 Dose-Limiting Toxicity by Preferred Termand Maximum CTCAE Toxicity Grade for Part C (Safety Population)

Table 14.3.1.2.4 Dose-Limiting Toxicity by Preferred Termand Maximum CTCAE Toxicity Grade for Part D (Safety Population)

Table 14.3.1.3.1

Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part A (Safety Population)

| Preferred Term | Statistics | Part A - 200 (N=XX) | Part A - 300 (N=XX) | Overall (N=XX |
|---|---|---|---|---|
| Any treatment emergent adverse event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | | |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Repeat Table 14.3.1.3.1 for

Table 14.3.1.3.2 Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part B (Safety Population)

Table 14.3.1.3.3 Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part C (Safety Population)

Table 14.3.1.3.4 Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part D (Safety Population)

Table 14.3.1.4.1
Treatment Emergent Adverse Events by Preferred Term for Part A (Safety Population)

| Preferred Term | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Any Treatment Emergent Adverse<br>Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1<br>PT 2 | n (%)<br>n (%) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| | ••• | | | |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

# Repeat for

Table 14.3.1.4.2 Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part B (Safety Population)

Table 14.3.1.4.3 Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part C (Safety Population)

Table 14.3.1.4.4 Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part D (Safety Population)

Table 14.3.1.5.1

Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part A (Safety Population)

| System Organ Class | | Part A-20 | 0 (N=XX) | Part A-30 | 0 (N=XX) | Part A | (N=XX) | _ |
|---|---|---|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Related to | Related to | Related to | Overall |
| Preferred Term | Statistics | Niraparib | TSR-042 | Niraparib | TSR-042 | Niraparib | TSR-042 | (N=XX) |
| Any Treatment | | | | | | | | |
| Emergent Adverse | | | | | | | | |
| Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| ••• | | | | | | | | |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part A: TSR-042 and niraparib (200mg/300mg) combination treatment

Table 14.3.1.5.2

Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part B Group (Safety Population)

| System Organ Class | | | Part B (N=XX | K) | |
|---|---|---|---|---|---|
| Preferred Term | Statistics | Related to TSR-042 | Related to<br>Carboplatin | Related to<br>Paclitaxel | Overall (N=XX) |
| Any Treatment Emergent Adverse Events | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | ••• | | | | |

Source: Listing 16.2.7.2

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

 $\label{thm:continuous} Table\ 14.3.1.5.3.1$  Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part C — Result 1 (Safety Population)

| System Organ Class | | F | Part C-200 (N= | =XX) | I | Part C-300 (N= | =XX) |
|---|---|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Related to | Related to | Related to |
| Preferred Term | Statistics | Niraparib | TSR-042 | Bevacizumab | Niraparib | TSR-042 | Bevacizumab |
| Any Treatment | | | | | | | |
| Emergent Adverse Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Table 14.3.1.5.3.2

Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part C - Result 2 (Safety Population)

| System Organ Class | | | Part C (N=X | X) | |
|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Overall |
| Preferred Term | Statistics | Niraparib | TSR-042 | Bevacizumab | (N=XX) |
| Any Treatment Emergent Adverse | | | | | |
| Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | | | |

Source: Listing 16.2.7.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part C: TSR-042, niraparib (200mg/300mg) and bevacizumab combination treatment

Table 14.3.1.5.4

Drug-Related Treatment Emergent Adverse Events by System Organ Class and Preferred Term for Part D (Safety Population)

| System Organ Class | _ | | Part 1 | D (N=XX) | | _ |
|---|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Related to | Overall |
| Preferred Term | Statistics | TSR-042 | Carboplatin | Paclitaxel | Bevacizumab | (N=XX) |
| Any Treatment Emergent Adverse | | | | | | |
| Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | | | | |
| SOC 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | ••• | | | | | |

Source: Listing 16.2.7.4

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Table 14.3.1.6.1

Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part A (Safety Population)

| | | Part A-20 | 0 (N=XX) | Part A-3 | 00 (N=XX) | Part A | (n=XX) | |
|---|---|---|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Related to | Related to | Related to | Overall |
| Preferred Term | Statistics | s Niraparib | TSR-042 | Niraparib | TSR-042 | Niraparib | TSR-042 | (N=XX) |
| Any Treatment Emergent Adverse | | | | | | | | |
| Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

# For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part A: TSR-042 and niraparib (200mg/300mg) combination treatment

Table 14.3.1.6.2

Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part B (Safety Population)

| | | | X) | | |
|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Overall |
| Preferred Term | Statistic | TSR-042 | Carboplatin | Paclitaxel | (N=XX) |
| Any Treatment Emergent Adverse Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.2

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment


TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

Table 14.3.1.6.3.1

Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part C – Result 1 (Safety Population)

| | | P | Part C-200 (N=XX) | | | Part C-300 (N=XX) | |
|---|---|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Related to | Related to | Related to |
| Preferred Term | Statistic | Niraparib | TSR-042 | Bevacizumab | Niraparib | TSR-042 | Bevacizumab |
| Any Treatment Emergent Adverse Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.3

PROGRAM NAME: DATE: DDMMYYYY

# For programmer: add following footnotes

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment


Table 14.3.1.6.3.2

Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part C – Result 2 (Safety Population)

| | | Part C (N=XX) | | | |
|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Overall |
| Preferred Term | Statistic | Niraparib | TSR-042 | Bevacizumab | (N=XX) |
| Any Treatment Emergent Adverse Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part C: TSR-042, niraparib (200mg/300mg) and bevacizumab combination treatment


Table 14.3.1.6.4

Drug-Related Treatment Emergent Adverse Events by Preferred Term in Decreasing Frequency for Part D (Safety Population)

| | | Part D (N=XX) | | | | |
|---|---|---|---|---|---|---|
| | | Related to | Related to | Related to | Related to | Overall |
| Preferred Term | Statistic | TSR-042 | Carboplatin | Paclitaxel | Bevacizumab | (N=XX) |
| Any Treatment Emergent Adverse Event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.4

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment


 $\label{thm:condition} Table~14.3.1.7.1$  Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade  $\geq$  3 for Part A (Safety Population)

| System Organ Class | | | | | |
|---|---|---|---|---|---|
| | | Maximum | Part A-200 | Part A-300 | Overall |
| Preferred Term | Statistics | CTCAE Grades | (N=XX) | (N=XX) | (N=XX) |
| Any Treatment Emergent Adverse Event | n (%) | | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| PT2 | n (%) | Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | n (%) | Grade 5 | xx (xx.x) | xx(xx.x) | xx (xx.x |
| SOC 2 | n (%) | $Grade \ge 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | n (%) | Grade 4 | xx (xx.x) | xx(xx.x) | xx (xx.x |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | ••• | | | | |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Repeat Table 14.3.1.7.1 for

Table 14.3.1.7.2 Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade ≥ 3 for Part B (Safety Population)

Table 14.3.1.7.3 Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade ≥ 3 for Part C (Safety Population)

Table 14.3.1.7.4 Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Maximum CTCAE Toxicity Grade ≥ 3 for Part D (Safety Population)

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

 $\label{eq:thm:condition} Table~14.3.1.8.1$  Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade  $\geq$  3 for Part A (Safety Population)

| System Organ Class | | Maximum | Part A-20 | 00 (N=XX) | Part A-30 | 0 (N=XX) | Part A | (N=XX) | _ |
|---|---|---|---|---|---|---|---|---|---|
| | | CTCAE | Related to | Related to | Related to | Related to | Related to | Related to | Overall |
| Preferred Term | Statistic | Grades | Niraparib | TSR-042 | Niraparib | TSR-042 | Niraparib | TSR-042 | (N=XX) |
| Any Treatment Emergent Adverse Event | n (%) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | $Grade \ge 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | $Grade \ge 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | ••• | | | | | | | | |
| SOC 2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

| System Organ Class | | | | Part B (N=XX | ) | |
|---|---|---|---|---|---|---|
| Preferred Term | Statistic | Maximum<br>CTCAE<br>Grades | Related to<br>TSR-042 | Related to<br>Carboplatin | Related to<br>Paclitaxel | Overall (N=XX) |
| Any Treatment Emergent | | | | | | |
| Adverse Event | n (%) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | ••• | | | | | |

Source: Listing 16.2.7.2

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

Table 14.3.1.8.3.1 Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade  $\geq$  3 for Part C – Result 1 (Safety Population)

| ystem Organ Class | • | Maximum | F | Part C-200 (N | =XX) | 1 | Part C-300 (N | =XX) |
|---|---|---|---|---|---|---|---|---|
| | | CTCAE | Related to | Related to | Related to | Related to | Related to | Related to |
| Preferred Term | Statistic | Grades | Niraparib | TSR-042 | Bevacizumab | Niraparib | TSR-042 | Bevacizumab |
| ny Treatment Emergent Adverse Event | n (%) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| OC 1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | Grade ≥ 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| OC 2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | | , , | ` ′ | ` ' | ` / | | ` , |

...

Source: Listing 16.2.7.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment


Table 14.3.1.8.3.2 Drug-Related Treatment Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum CTCAE Toxicity Grade  $\geq 3$  for Part C – Result 2 (Safety Population)

| System Organ Class | | Maximum | | Part C (N=X | (X) | _ |
|---|---|---|---|---|---|---|
| | | CTCAE | Related to | Related to | Related to | Overall |
| Preferred Term | Statistic | Grades | Niraparib | TSR-042 | Bevacizumab | (N=XX) |
| Any Treatment Emergent | | | | | | |
| Adverse Event | n (%) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | | | | |
| SOC 2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | | | | | | |

Source: Listing 16.2.7.3

PROGRAM NAME:

TESARO Inc.

Statistical Analysis Plan Protocol No: 3000-01-002 Dated:18SEP2020

DATE: DDMMYYYY

For programmer: add following footnotes

Part C: TSR-042, niraparib (200mg/300mg) and bevacizumab combination treatment


 $TESARO\ Inc.$ 


 $\label{eq:total control of the con$ 

| System Organ Class | | Maximum | | Part D | (N=XX) | | |
|---|---|---|---|---|---|---|---|
| , , | | CTCAE | Related to | Related to | Related to | Related to | Overall |
| Preferred Term | Statistic | Grades | TSR-042 | Carboplatin | Paclitaxel | Bevacizumab | (N=XX) |
| Any Treatment | | | | | | | |
| Emergent Adverse | (0./) | | | , | , , | | , , |
| Event | n (%) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 1 | (0/) | Grade ≥ 3 | () | () | () | xx (xx.x) | xx (xx.x) |
| SOC I | n (%) | _ | xx (xx.x) | xx (xx.x) | xx (xx.x) | | , , |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 111 | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | ` , | | , , | , | , , | ` / | ` / |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| ••• | 11 (70) | 31440 | () | () | () | () | () |
| SOC 2 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT1 | n (%) | Grade $\geq 3$ | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | n (%) | Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |


TESARO Inc.

Statistical Analysis Plan Protocol No: 3000-01-002 Dated:18SEP2020

Source: Listing 16.2.7.4

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Confidential Page 132 | 234 Repeat Table 14.3.1.3.1 for

Table 14.3.1.9.1 Serious AEs by System Organ Class and Preferred Term for Part A (Safety Population)

Table 14.3.1.9.2 Serious AEs by System Organ Class and Preferred Term for Part B (Safety Population)

Table 14.3.1.9.3 Serious AEs by System Organ Class and Preferred Term for Part C (Safety Population)

Table 14.3.1.9.4 Serious AEs by System Organ Class and Preferred Term for Part D (Safety Population)

Repeat Table 14.3.1.5.1 for

Table 14.3.1.10.1 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part A (Safety Population)

Repeat Table 14.3.1.5.2 for

Table 14.3.1.10.2 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part B (Safety Population)

Repeat Table 14.3.1.5.3.1 for

Table 14.3.1.10.3.1 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part C – Result 1 (Safety Population)

Repeat Table 14.3.1.5.3.2 for

Table 14.3.1.10.3.2 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part C – Result 2 (Safety Population)

Repeat Table 14.3.1.5.4 for

Table 14.3.1.10.4 Drug-Related Serious AEs by System Organ Class and Preferred Term for Part D (Safety Population)


#### Repeat Table 14.3.1.3.1 for

Table 14.3.1.11.1 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part A (Safety Population)

Table 14.3.1.11.2 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part B (Safety Population)

Table 14.3.1.11.3 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part C (Safety Population)

Table 14.3.1.11.4 Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part D (Safety Population)

TESARO Inc.


Dated:18SEP2020

Repeat Table 14.3.1.5.1 for

Table 14.3.1.12.1 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part A (Safety Population)

Repeat Table 14.3.1.5.2 for

Table 14.3.1.12.2 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part B (Safety Population)

Repeat Table 14.3.1.5.3.1 for

Table 14.3.1.12.3.1 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part C – Result 1 (Safety Population)

Repeat Table 14.3.1.5.3.2 for

Table 14.3.1.12.3.2 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part C – Result 2 (Safety Population)

Repeat Table 14.3.1.5.4 for

Table 14.3.1.12.4 Drug-Related Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class and Preferred Term for Part D (Safety Population)

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

Table 14.3.1.13.1.1

Treatment Emergent Adverse Events Leading to Niraparib Reduction/Interruption by System Organ Class and Preferred Term for Part A (Safety Population)

| Statistics | Part A-200 (N=XX) | Part A-300 (N=XX) | Overall (N=XX) |
|---|---|---|---|
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n (%) | vv (vv v) | vv (vv v) | xx (xx.x) |
| | · · | | xx (xx.x) |
| | | | xx (xx.x) |
| 11 (70) | AA (AA.A) | XX (XX.X) | XX (XX.X) |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | · · | | xx (xx.x) |
| | · · | | xx (xx.x) |
| | . , | , , | , , |
| n (0/s) | vv (vv v) | vv (vv v) | vv (vv v) |
| | · · | · · | xx (xx.x) |
| | · · | | xx (xx.x) |
| n (%) | XX (XX.X) | XX (XX.X) | xx (xx.x) |
| | n (%) n (%) n (%) n (%) n (%) n (%) | n (%) | n (%) xx (xx.x) xx (xx.x) n (%) xx (xx.x) xx (xx.x) |

Source: Listing 16.2.7.1

PROGRAM NAME:

DATE: DDMMYYYY

#### Repeat using proper drugs in the treatment for

Table 14.3.1.13.1.2 Treatment Emergent Adverse Events Leading to Niraparib Reduction/Interruption by System Organ Class and Preferred Term for Part C (Safety Population)

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Protocol No: 3000-01-002

Dated:18SEP2020

Repeat Table 14.3.1.3.1 for

Table 14.3.1.13.2.1 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part A (Safety Population)

Table 14.3.1.13.2.2 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part B (Safety Population)

Table 14.3.1.13.2.3 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part C (Safety Population)

Table 14.3.1.13.2.4 Treatment Emergent Adverse Events Leading to TSR-042 Interruption by System Organ Class and Preferred Term for Part D (Safety Population)

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

Repeat Table 14.3.1.3.1 for

Table 14.3.1.13.3.1 Treatment Emergent Adverse Events Leading to Carboplatin Interruption by System Organ Class and Preferred Term for Part B (Safety Population)

Table 14.3.1.13.3.2 Treatment Emergent Adverse Events Leading to Carboplatin Interruption by System Organ Class and Preferred Term for Part D (Safety Population)


Dated:18SEP2020

Repeat Table 14.3.1.3.1 for

Table 14.3.1.13.4.1 Treatment Emergent Adverse Events Leading to Paclitaxel Interruption by System Organ Class and Preferred Term for Part B (Safety Population)

Table 14.3.1.13.4.2 Treatment Emergent Adverse Events Leading to Paclitaxel Interruption by System Organ Class and Preferred Term for Part D (Safety Population)

Table 14.3.1.13.5.1 Treatment Emergent Adverse Events Leading to Bevacizumab Interruption by System Organ Class and Preferred Term for Part C (Safety Population)

Table 14.3.1.13.5.2 Treatment Emergent Adverse Events Leading to Bevacizumab Interruption by System Organ Class and Preferred Term for Part D (Safety Population)

Statistical Analysis Plan **Dated:18SEP2020** 

TESARO Inc.


Table 14.3.1.14.1
Deaths in Part A (Safety Population)

| Period | Statistic | Part A-200 (N=XX) | Part A-300 (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| During Treatment Period | | | | |
| Deaths | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reasons for Death | | | | |
| Disease Progression | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Follow-up Period | | | | |
| Deaths | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for Death | | | | |
| Disease Progression | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse event | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment


TESARO Inc.

Statistical Analysis Plan Protocol No: 3000-01-002 Dated:18SEP2020

Repeat Table 14.3.1.14.1 for

Table 14.3.1.14.2 Deaths in Part B (Safety Population)

Table 14.3.1.14.3 Deaths in Part C (Safety Population)

Table 14.3.1.14.4 Deaths in Part D (Safety Population)

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

Table 14.3.1.15.1

Adverse Events of Special Interest by Preferred Term for Part A (Safety Population)

| Adverse Event Special Interest Category Preferred Term | Statistic | TRT A-200 (N=XX) | TRT A-300 (N=XX) | Overall (N=XX) |
|---|---|---|---|---|
| Any Adverse Event of Special Interest | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Category 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Category 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 1 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 2 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PT 3 | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Source: Listing 16.2.7.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

TRT A-200: TSR-042 and niraparib (200mg) combination treatment TRT A-300: TSR-042 and niraparib (300mg) combination treatment
Statistical Analysis Plan **Protocol No: 3000-01-002 Dated:18SEP2020** 

Repeat for

Table 14.3.1.15.2 Adverse Events of Special Interest by Preferred Term for Part B (Safety Population)

Table 14.3.1.15.3 Adverse Events of Special Interest by Preferred Term for Part C (Safety Population)

Table 14.3.1.15.4 Adverse Events of Special Interest by Preferred Term for Part D (Safety Population)

Table 14.3.1.16

Overall Summary of Immune Related Treatment Emergent Adverse Events by Preferred Term (Safety Population)

| | | | | TSR-042 | | TSR-042 | Leading to |
|---|---|---|---|---|---|---|---|
| | | TSR-042 | | Related | | Related | TSR-042 |
| Preferred | Term/Overall | Related | >=Grade3 | >=Grade3 | 3 SAE | SAE | Discontinuation |
| Treatment | n (%) | n (%) | n(%) | n(%) | n(%) | n(%) | n (%) |
| Diarrhoea | | | | | | | |
| Part A-200 (N= 16) | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Part A-300 (N= 6) | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Part B (N= 14) | 3 ( 21.43) | 0 | 0 | 0 | 0 | 0 | 0 |
| Part C-200 (N= 6) | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Part C-300 (N= 7) | 1(14.29) | 1(14.29) | 1(14.29) | 1(14.29) | 0 | 0 | 0 |
| Part D (N= 6) | 3 ( 50.00) | 0 | 1(16.67) | 0 | 0 | 0 | 0 |
| Overall (N= 55) | 7 ( 12.73) | 1( 1.82) | 2 ( 3.64) | 1( 1.82) | 0 | 0 | 0 |
| Alanineaminotransferase increased | | | | | | | |
| Part A-200 (N= 16) | 1( 6.25) | 1( 6.25) | 1( 6.25) | 1( 6.25) | 0 | 0 | 0 |
| Part A-300 (N= 6) | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Part B (N= 14) | 2(14.29) | 2(14.29) | 2(14.29) | 2(14.29) | 0 | 0 | 2(14.29) |
| Part C-200 (N= 6) | 1(16.67) | 0 | 0 | 0 | 0 | 0 | 0 |
| Part C-300 (N= 7) | 1(14.29) | 1(14.29) | 1(14.29) | 1(14.29) | 0 | 0 | 0 |
| Part D (N= 6) | 1(16.67) | 0 | 0 | 0 | 0 | 0 | 0 |
| Overall (N= 55) | 6(10.91) | 4 ( 7.27) | 4 ( 7.27) | 4 ( 7.27) | 0 | 0 | 2(3.64) |

TESARO Inc.


Statistical Analysis Plan
Dated:18SEP2020

# Table 14.3.2.1 Patients with Adverse Events with Outcome of Death (Safety Analysis Set)

| | Patient | | | Last Dose | Death | Death<br>within 90<br>Days of<br>Last | |
|---|---|---|---|---|---|---|---|
| Part | ID | Drugs | Date | Date | Date | Treatment | Cause of Death |
| | | | | | DDMM | | |
| | | | | | YYYY | Y/N | |

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

 $Part\ D:\ TSR-042,\ carboplatin-paclitaxel\ and\ bevacizumab\ combination\ treatment$ 

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment

TESARO Inc. Statistical Analysis Plan Protocol No: 3000-01-002 **Dated:18SEP2020** 

Table 14.3.2.2 Listing of Serious Adverse Events (Safety Population)

| | | System Organ Class/ | | | | | Action | |
|---|---|---|---|---|---|---|---|---|
| | | Preferred Term/Verbatim | Start Date/Time | Stop | | Relationship | Taken | 16.2.7. |
| Part | Patient ID | Term | (Rel Days [1]) | Date/Time | Severity | to Drug | [2][3] | 1 |
| | | | DDMMYYYYTH | | | | | |
| Part A - 200 | | | H:MM:SS (days) | | | | | Y/N |
| Part A - 300 | | | | ongoing | | | | |

- [1] Rel Days are calculated as AE date minus first dose date (plus 1 day if AE date is on or after first dose date).
- [2] N=Niraparib, T=TSR-042, C=Carboplatin, PC=Paclitacxel, B=Bevacizumab, PM=Pemetrexed, TT=TSR-022 [3] 1= Dose/Infusion Not Changed; 4= Drug/Infusion Interrupted; 5= Infusion Delayed; 6= Drug Withdrawn; 7= Not Applicable;

PROGRAM NAME: DATE: DDMMYYYY

#### Repeat for

Table 14.3.2.3 Listing of Treatment Emergent Adverse Events Leading to Dose Interruption (Safety Population)

Table 14.3.2.4 Listing of Treatment Emergent Adverse Events Leading to Dose Modification (Safety Population)

Table 14.3.2.5 Listing of Treatment Emergent Adverse Events Leading to Discontinuation from Treatment (Safety Population)

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

Table 14.3.4.1 Listing of Abnormal Laboratory Values (Safety Population)

| Part | Patient ID | Age/Sex | Group | Visit | Visit Date (Rel<br>Days [1]) | Laboratory Test<br>(Unit) | Measurement<br>Date | Result | CTCAE<br>Grade | Normal<br>Range | Clinically<br>Significant |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Chemistry | Baseline | | | DDMMYYYY | | | xx.xx, xx.xx | Y/N |
| | | | | ••• | | | | | | | |
| | | | Hematology | Baseline | | | | | | | |
| | | | | ••• | | | | | | | |
| | | | Coagulation | Baseline | | | | | | | |
| | | | | ••• | | | | | | | |
| | | | Chemistry | Baseline | | | | | | | |
| | | | | ••• | | | | | | | |

[1] Rel Days are calculated as visit date minus first dose date (plus 1 day if visit date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

#### Repeat for

Table 14.3.4.2 Listing of Laboratory Values with CTCAE Toxicity Grade ≥ 3 (Safety Population)

Table 14.3.4.3 Listing of Clinically Significant Laboratory Values (Safety Population)

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

TESARO Inc.

Table 14.3.5.1 Extent of Exposure for Part A (Safety Population)

| Study Drug Parameters | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall<br>(N=XX) |
|---|---|---|---|---|
| Niraparib | Statistics . | (11 1111) | (11 111) | (11112) |
| Duration of Exposure (days) | n | XX | XX | XX |
| Duranon of Empound (augu) | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | 1,1111, 1,1421 | M, M | AA, AA | <i>m</i> , <i>m</i> |
| Number of Treatment Cycles | | | | |
| 1 Cycle | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Actual Cumulative Dose (mg) | n | XX | XX | XX |
| retain Camalative Bose (mg) | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | ivini, iviax | AA, AA | AA, AA | AA, AA |
| Actual Dose Intensity (mg/day) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Relative Dose Intensity (%) | n | xx | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| Number of patients with dose interruptions | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Number of patients with dose reduction | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| TSR-042 | | | | |
| Duration of Treatment (day) | n | XX | XX | XX |
| . • , | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Number of Treatment Cycles | | | | |
| 1 Cycle | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | n (70) | MAX (MAM) | AM (MAX) | MAX (MAIA) |
| Actual Dose Intensity (mg/day) | | | | |
| < 5 <sup>th</sup> Cycle | n | vv | vv | XX |
| \ J Cyclc | Mean (STD) | xx<br>xx.x (xx.xx) | xx<br>xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | | | |
| | Min, Max | XX.X | XX.X | XX.X |
| | wiii, wiax | xx, xx | xx, xx | XX, XX |
| | Confidentia | 1 | Pa | ge 150 234 |


| $\geq 5^{\text{th}}$ Cycle | n | XX | XX | XX |
|---|---|---|---|---|
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Relative dose Intensity (%) | | | | |
| < 5 <sup>th</sup> Cycle | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| ≥ 5 <sup>th</sup> Cycle | n | XX | xx | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Source: Listing 16.2.5.4 Listing 16.2.5.5 Listing 16.2.5.6

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

TESARO Inc.

Table 14.3.5.2 Extent of Exposure for Part B (Safety Population)

| G. I. D. | | |
|--------------------------------------------|------------|---------------|
| Study Drug Parameters | Statistics | Part B (N=XX) |
| TSR-042 | Statistics | Tand (IV-AA) |
| Duration of Treatment (day) | n | XX |
| Butunon of Treatment (auy) | Mean (STD) | xx.x (xx.xx) |
| | Median | xx.x |
| | Min, Max | XX, XX |
| Number of Treatment Cycles | | |
| 1 Cycle | n (%) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) |
| ••• | | |
| Actual Cumulative Dose (mg) | | |
| < 5th Cycle | n | XX |
| | Mean(STD) | xx.x (xx.xx) |
| | Median | XX.X |
| A set of | Min,Max | xx, xx |
| ≥ 5 <sup>th</sup> Cycle | n | XX |
| | Mean(STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx, xx |
| Actual Dose Intensity (mg/day) | | |
| < 5 <sup>th</sup> Cycle | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| > 5th C 1 | | |
| ≥ 5 <sup>th</sup> Cycle | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| Relative dose Intensity (%) | | |
| < 5 <sup>th</sup> Cycle | n | XX |
| . J. Cyclo | Mean (STD) | xx.x (xx.xx) |
| | Median | ` ´ |
| | Min, Max | XX.X |
| | wiiii, wax | XX, XX |
| ≥ 5 <sup>th</sup> Cycle | n | XX |
| · | Mean (STD) | xx.x (xx.xx) |
| | Median | xx.x |
| | Min, Max | xx, xx |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) |
| Paclitaxel | | |
| Duration of Treatment (day) | n | XX |
| ·-···································· | | |


| | Mean (STD) | xx.x (xx.xx) |
|--------------------------------------------|------------|--------------|
| | Median | XX.X |
| | Min, Max | XX, XX |
| Number of Treatment Cycles | | |
| 1 Cycle | n (%) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) |
| Actual Dose Intensity (mg/m2/day) | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| Relative dose Intensity (%) | n | XX |
| • · | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) |
| Carboplatin | | |
| Duration of Treatment (day) | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| Number of Treatment Cycles | | |
| 1 Cycle | n (%) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) |

Source: Listing 16.2.5.6 Listing 16.2.5.7 Listing 16.2.5.8

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Table 14.3.5.3 Extent of Exposure for Part C (Safety Population)

| | | Part C-200 | Part C-300 | Overall |
|---|---|---|---|---|
| Parameters | Statistics | (N=XX) | (N=XX) | (N=XX) |
| Niraparib | | | | |
| Duration of Exposure (day) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| Number of Treatment Cycles | | | | |
| 1 Cycle | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Actual Cumulative Dose (mg) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| Actual Dose Intensity (mg/day) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | xx.x | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Relative Dose Intensity (%) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Min, Max | xx, xx | xx, xx | XX, XX |
| Number of patients with dose interruptions | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Number of patients with dose reduction | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

| Protocol | No: | 3000- | 01-002 |
|----------|-----|-------|--------|
|----------|-----|-------|--------|

| TSR-042 | | | | |
|---|---|---|---|---|
| Duration of Treatment (day) | n<br>Mean (STD) | xx<br>xx.x (xx.xx) | xx<br>xx.x (xx.xx) | xx<br>xx.x (xx.xx) |
| | Median<br>Min, Max | XX.X<br>XX, XX | xx.x<br>xx, xx | XX.X<br>XX, XX |
| Number of Treatment Cycles | | | | |
| 1 Cycle | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Actual Cumulative Dose(mg) | | | | |
| < 5 <sup>th</sup> Cycle | n | XX | XX | n |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | Mean (STD) |
| | Median | XX.X | XX.X | Median |
| S of h G 1 | Min, Max | XX, XX | xx, xx | Min, Max |
| $\geq 5^{\text{th}}$ Cycle | n<br>M (CTD) | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median<br>Min May | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | xx, xx |
| Actual Dose Intensity (mg/day) | | | | |
| < 5 <sup>th</sup> Cycle | n | XX | XX | n |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | Mean (STD) |
| | Median | XX.X | XX.X | Median |
| | Min, Max | XX, XX | XX, XX | Min, Max |
| ≥ 5 <sup>th</sup> Cycle | n | xx | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Relative dose Intensity (%) | | | | |
| < 5 <sup>th</sup> Cycle | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Min, Max | XX, XX | xx, xx | xx, xx |
| | , | , | , | * |

| ≥ 5 <sup>th</sup> Cycle | n | XX | xx | XX |
|---|---|---|---|---|
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | xx.x |
| | Min, Max | xx, xx | XX, XX | xx, xx |
| Number of patients with dose interruptions | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Bevacizumab | | | | |
| Duration of Treatment (day) | n | xx | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Number of Treatment Cycles | | | | |
| 1 Cycle | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Actual Cumulative Dose (mg) | n | XX | XX | XX |
| Treatment of Desc (mg) | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | xx.x | xx.x |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Actual Dose Intensity (mg/kg/day) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | XX.X | XX.X | XX.X |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| Relative dose Intensity (%) | n | XX | XX | XX |
| | Mean (STD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | Median | xx.x | XX.X | XX.X |
| | Min, Max | xx, xx | xx, xx | xx, xx |
| Number of patients with dose interruptions | n (%) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Statistical Analysis Plan Protocol No: 3000-01-002 Dated:18SEP2020

Source: Listing 16.2.5.4 Listing 16.2.5.5 Listing 16.2.5.6

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Table 14.3.5.4 Extent of Exposure for Part D (Safety Population)

| Parameters | Statistics | Part D (N=XX) |
|--------------------------------|------------|---------------|
| TSR-042 | | , |
| Duration of Treatment (day) | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx, xx |
| Number of Treatment Cycles | | |
| 1 Cycle | n (%) | xxx(xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) |
| Actual Cumulative Dose(mg) | | |
| < 5 <sup>th</sup> Cycle | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx, xx |
| ≥ 5 <sup>th</sup> Cycle | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| Actual Dose Intensity (mg/day) | | |
| < 5 <sup>th</sup> Cycle | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| ≥ 5 <sup>th</sup> Cycle | n | XX |
| 3 | Mean (STD) | xx.x (xx.xx) |
| | Median | xx.x |
| | Min, Max | xx, xx |
| Relative dose Intensity (%) | | |
| < 5 <sup>th</sup> Cycle | n | XX |
| - | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Wicaian | AA.A |

| | Min, Max | xx, xx |
|--------------------------------------------|------------|--------------|
| ≥ 5 <sup>th</sup> Cycle | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx, xx |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) |
| Paclitaxel | | |
| Duration of Treatment (day) | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx, xx |
| Number of Treatment Cycles | | |
| 1 Cycle | n (%) | xxx (xx.x) |
| 2 Cycles | n (%) | xxx (xx.x) |
| Actual Cumulative Dose (mg) | n | XX |
| ( 0) | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | XX, XX |
| Actual Dose Intensity (mg/m²/day) | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx, xx |
| Relative dose Intensity (%) | n | XX |
| | Mean (STD) | xx.x (xx.xx) |
| | Median | XX.X |
| | Min, Max | xx, xx |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) |
| Carboplatin | | |

| Duration of Treatment (day) | n<br>Mean (STD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
|---|---|---|
| Number of Treatment Cycles 1 Cycle 2 Cycles | n (%)<br>n (%) | xxx (xx.x)<br>xxx (xx.x) |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) |
| Bevacizumab | | |
| Duration of Treatment (day) | n<br>Mean (STD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| Number of Treatment Cycles 1 Cycle 2 Cycles | n (%)<br>n (%) | xxx (xx.x)<br>xxx (xx.x) |
| Actual Cumulative Dose (mg) | n<br>Mean (STD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| Actual Dose Intensity (mg/kg/day) | n<br>Mean (STD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| Relative dose Intensity (%) | n<br>Mean (STD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx, xx |
| Number of patients with Dose Interruptions | n (%) | xxx (xx.x) |

Statistical Analysis Plan Protocol No: 3000-01-002 Dated:18SEP2020

Source: Listing 16.2.5.6 Listing 16.2.5.7 Listing 16.2.5.8 Listing 16.2.5.11

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment


TESARO Inc.


Statistical Analysis Plan
Dated:18SEP2020

Figure 14.3.5.1
Swimmer Plot of Treatment Duration for Part A (Safety Population)



This is an example of swimmer plot. Add indicators to the plot: primary tumor type, treatment on-going or discontinued and response at each tumor assessment. Source: Listing 16.2.6.1

PROGRAM NAME: DATE: DDMMYYYY

Programming Notes for Programmers

Include subjid and dose level in Y-axis. Label should be Subject (Dose level) Y-axis label should be "Duration of exposure (weeks)"

| TES | ARC | Inc. |
|------|--------|------|
| ILD. | $\sim$ | me. |


| * | End of Treatment | |
|---|------------------|---------------|
| • | PR | |
| A | SD | |
| A | PD | in the figure |

Include the following indicators in the figure. Legend should be placed in the bottom right corner of the figure

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Statistical Analysis Plan **Dated:18SEP2020** 


Statistical Analysis Plan **Dated:18SEP2020** 

Repeat Figure 14.3.5.1 for

Figure 14.3.5.2 Swimmer Plot of Treatment Duration for Part B (Safety Population)

Figure 14.3.5.3 Swimmer Plot of Treatment Duration for Part C (Safety Population)

Figure 14.3.5.4 Swimmer Plot of Treatment Duration for Part D (Safety Population)

TESARO Inc.

Table 14.3.6.1.1 Summary of Actual and Change from Baseline Value for Hematology Parameters for Part A (Safety Population)

| | | Actual/Chan | | PARTA-200 | PART | A-300 Overall |
|---|---|---|---|---|---|---|
| Parameter | Visit | ge | Statistics | (N=16) | (N=6) | (N=22) |
| Hemoglobin (g/L) | Baseline | Actual | n | 16 | 6 | 22 |
| | | | Mean (STD) | 121.6 (13.36) | 134.0 (8.72) | 125.0 (13.32) |
| | | | Median | 123.0 | 132.0 | 126.5 |
| | | | Min, Max | 93, 146 | 126, 151 | 93, 151 |
| | CYCLE 1 DAY 8 | Actual | n | 16 | 5 | 21 |
| | | | Mean (STD) | 120.8 (12.87) | 133.8 (7.95) | 123.9 (13.01) |
| | | | Median | 122.0 | 131.0 | 127.0 |
| | | | Min, Max | 100, 145 | 127, 147 | 100, 147 |
| | | Change | n | 16 | 5 | 21 |
| | | | Mean (STD) | -0.9 (6.70) | -0.4 (4.83) | -0.8 (6.20) |
| | | | Median | -1.0 | -1.0 | -1.0 |
| | | | Min, Max | <b>-9,</b> 16 | <b>-6,</b> 5 | <b>-9,</b> 16 |
| | CYCLE 1 DAY 15 | Actual | n | 13 | 6 | 19 |
| | | | Mean (STD) | 119.8 (12.77) | 127.0 (7.18) | 122.1 (11.60) |
| | | | Median | 124.0 | 127.5 | 125.0 |
| | | | Min, Max | 93, 139 | 115, 137 | 93, 139 |
| | | Change | n | 13 | 6 | 19 |
| | | | Mean (STD) | -2.5 (9.32) | -7.0 (10.68) | -3.9 (9.71) |
| | | | Median | -5.0 | -5.5 | -5.0 |
| | | | Min, Max | -18, 16 | -23, 6 | -23, 16 |

# Statistical Analysis Plan **Dated:18SEP2020**

Repeat Table 14.3.6.1.1 for

Table 14.3.6.1.2 Summary of Actual and Change from Baseline Value for Hematology Parameters for Part B (Safety Population)

Table 14.3.6.1.3 Summary of Actual and Change from Baseline Value for Hematology Parameters for Part C (Safety Population)

Table 14.3.6.1.4 Summary of Actual and Change from Baseline Value for Hematology Parameters for Part D (Safety Population)

# Statistical Analysis Plan **Dated:18SEP2020**

Repeat Table 14.3.6.1.1 for

Table 14.3.6.2.1 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part A (Safety Population)

Table 14.3.6.2.2 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part B (Safety Population)

Table 14.3.6.2.3 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part C (Safety Population)

Table 14.3.6.2.4 Summary of Actual and Change from Baseline Value for Chemistry Parameters for Part D (Safety Population)


Statistical Analysis Plan **Dated:18SEP2020** 

Repeat Table 14.3.6.1.1 for

Table 14.3.6.3.1 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part A (Safety Population)

Table 14.3.6.3.2 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part B (Safety Population)

Table 14.3.6.3.3 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part C (Safety Population)

Table 14.3.6.3.4 Summary of Actual and Change from Baseline Value for Coagulation Parameters for Part D (Safety Population)

Repeat Table 14.3.6.1.1 for

Table 14.3.6.4.1 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part A (Safety Population)

Table 14.3.6.4.2 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part B (Safety Population)

Table 14.3.6.4.3 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part C (Safety Population)

Table 14.3.6.4.4 Summary of Actual and Change from Baseline Value for Thyroid Function Parameters for Part D (Safety Population)


Statistical Analysis Plan **Dated:18SEP2020** 

Repeat Table 14.3.6.1.1 for

Table 14.3.7.1 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part A (Safety Population)

Table 14.3.7.2 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part B (Safety Population)

Table 14.3.7.3 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part C (Safety Population)

Table 14.3.7.4 Summary of Actual and Change from Baseline Value for ECG Continuous Parameters for Part D (Safety Population)

Programming Notes for programmers:

Add Timepoint column after Visit to capture the timepoints PREDOSE and 2 HOURS POST DOSE

TESARO Inc.


Statistical Analysis Plan

Dated:18SEP2020

Table 14.3.8.1.1
Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part A (Safety Population)

| Hemoglobin (Anemia) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| (MICHEA) | | | Post-Baseline Maximum CTCAE Grade | | | | | | | |
| Treatment Group | Statistics | Baseline<br>CTCAE Grade | Missing | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 | Overall |
| Part A-200 (N=16) | n (%) | Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Grade 0 | 0 | 1 (6.3) | 3 (18.8) | 1 (6.3) | 2 (12.5) | 0 | 0 | 7 (43.8) |
| | n (%) | Grade 1 | 0 | 0 | 4 (25.0) | 3 (18.8) | 1 (6.3) | 0 | 0 | 8 (50.0) |
| | n (%) | Grade 2 | 0 | 0 | 0 | 0 | 1 (6.3) | 0 | 0 | 1 (6.3) |
| | n (%) | Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Overall | 0 | 1 (6.3) | 7 (43.8) | 4 (25.0) | 4 (25.0) | 0 | 0 | 16<br>(100.0) |
| Part A-300 (N=6) | n (%) | Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Grade 0 | 0 | 1 (16.7) | 0 | 2 (33.3) | 0 | 0 | 0 | 3 (50.0) |
| | n (%) | Grade 1 | 0 | 0 | 2 (33.3) | 1 (16.7) | 0 | 0 | 0 | 3 (50.0) |
| | n (%) | Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Overall | 0 | 1 (16.7) | 2 (33.3) | 3 (50.0) | 0 | 0 | 0 | 6 (100.0) |

. . .

Note: Percentages are based on number of patients who has grades present at both baseline and post-baseline in safety population for each study treatment.

Source: Listing 16.2.8.1

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Repeat Table 14.3.8.1.1 for

Table 14.3.8.1.2 Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part B (Safety Population)

Table 14.3.8.1.3 Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part C (Safety Population)

Table 14.3.8.1.4 Shift of Hematology Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part D (Safety Population)


# Statistical Analysis Plan **Dated:18SEP2020**

Repeat Table 14.3.8.1.1 for

Table 14.3.8.2.1 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part A (Safety Population)

Table 14.3.8.2.2 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part B (Safety Population)

Table 14.3.8.2.3 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part C (Safety Population)

Table 14.3.8.2.4 Shift of Chemistry Parameters from Baseline to Worst Post-Baseline Toxicity Grade for Part D (Safety Population)

TESARO Inc.

Table 14.3.9.1.1

Summary of Post-Baseline Liver Function for Part A (Safety Population)

| Maximum | Elevation | under | PART | A-200 PART | A-300 Overall |
|---|---|---|---|---|---|
| treatment | | Statistics | (N=16) | (N=6) | (N=22) |
| ALT | | | | | |
| <3 x ULN | | n (%) | 15( 93.8) | 6(100.0) | 21( 95.5) |
| 3 x ULN =< < 5 | x ULN | n (%) | 0 | 0 | 0 |
| 5 x ULN =< < 10 | ) x ULN | n (%) | 0 | 0 | 0 |
| 10 x ULN =< < 2 | 20 x ULN | n (%) | 0 | 0 | 0 |
| >= 20 x ULN | | n(%) | 1(6.3) | 0 | 1 ( 4.5) |
| AST | | | | | |
| <3 x ULN | | n (%) | 14( 87.5) | 5 ( 83.3) | 19( 86.4) |
| 3 x ULN =< < 5 | x ULN | n(%) | 1(6.3) | 0 | 1( 4.5) |
| 5 x ULN =< < 10 | ) x ULN | n(%) | 0 | 1(16.7) | 1( 4.5) |
| 10 x ULN =< < 2 | 20 x ULN | n(%) | 0 | 0 | 0 |
| >= 20 x ULN | | n(%) | 1(6.3) | 0 | 1 ( 4.5) |
| ALT or AST | | | | | |
| <3 x ULN | | n (%) | 13( 81.3) | 5 ( 83.3) | 18( 81.8) |
| 3 x ULN =< < 5 | x ULN | n (%) | 1(6.3) | 0 | 1( 4.5) |
| 5 x ULN =< < 10 | ) x ULN | n (%) | 0 | 1(16.7) | 1( 4.5) |
| 10 x ULN =< < 2 | 20 x ULN | n (%) | 0 | 0 | 0 |
| >= 20 x ULN | | n(%) | 1(6.3) | 0 | 1 ( 4.5) |
| Total Bilirubin Level | _ (TBL) | | | | |
| < 1.5 x ULN | | n(%) | 15( 93.8) | 5 ( 83.3) | 20( 90.9) |
| 1.5 x ULN =< < | 2 x ULN | n(%) | 1(6.3) | 0 | 1( 4.5) |
| >= 2 x ULN | | n(%) | 0 | 1(16.7) | 1 ( 4.5) |
| Alkaline Phosphatase | (ALP) | | | | |
| < 1.5 x ULN | | n (웅) | 11( 68.8) | 4 ( 66.7) | 15 ( 68.2) |
| 1.5 x ULN =< < | 2 x ULN | n(%) | 0 | 0 | 0 |
| >= 2 x ULN | | n (%) | 5 ( 31.3) | 2(33.3) | 7 ( 31.8) |

| TESARO Inc. Protocol No: 3 | 3000-01-002 | 2 | | | | | Statistical Analysis Plan <b>Dated:18SEP2020</b> |
|---|---|---|---|---|---|---|---|
| Concurrent TBL >=2×ULN | ALT | | >=3×ULN | and n (%) | 0 | 0 | 0 |
| Concurrent TBL >=2×ULN | AST | | >=3×ULN | and n (%) | 0 | 1(16.7) | 1( 4.5) |
| Concurrent TBL >=2×ULN | (ALT | or AST | ) >=3×ULN | and n(%) | 0 | 1(16.7) | 1( 4.5) |
| Concurrent TBL >=2×ULN an | • | or AST<br>×ULN | ) >=3×ULN | and n (%) | 0 | 1(16.7) | 1( 4.5) |
| Potential<br>Concurrent | (ALT | Hy's | AST) | law: n(%)<br>>=3×ULN | 0 | 0 | 0 |

## Repeat for

and TBL  $>=2 \times ULN$  and ALP  $<2 \times ULN$ 

Table 14.3.9.1.2 Summary of Post-Baseline Liver Function for Part B (Safety Population)

Table 14.3.9.1.3 Summary of Post-Baseline Liver Function for Part C (Safety Population)

Table 14.3.9.1.4 Summary of Post-Baseline Liver Function for Part D (Safety Population)

Table 14.3.10.1.1

Shift of ECOG Performance Status from Baseline to Worst Post-Baseline Score for Part A (Safety Population)

| | Worst Post-Baseline ECOG Score | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Part | Statist | Baseline<br>ECOG<br>cics Score | 0 | 1 | 2 | 3 | 4 | 5 | Missing | Overall |
| Part A-200 (N=16) | n (%) | 0 | 3 ( 18.8) | 4 ( 25.0) | 0 | 0 | 0 | 0 | 1(6.3) | 8 ( 50.0) |
| | n(%) | 1 | 0 | 5 ( 31.3) | 1(6.3) | 0 | 0 | 0 | 2(12.5) | 8 ( 50.0) |
| | n(%) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n(%) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n(%) | Overall | 3 ( 18.8) | 9(56.3) | 1(6.3) | 0 | 0 | 0 | 3 ( 18.8) | 16(100.0) |
| Part A-300 (N=6) | n (%) | 0 | 1(16.7) | 1(16.7) | 1(16.7) | 0 | 0 | 0 | 0 | 3 ( 50.0) |
| | n(%) | 1 | 0 | 3 ( 50.0) | 0 | 0 | 0 | 0 | 0 | 3 ( 50.0) |
| | n(%) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n(%) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n(%) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | Overall | 1(16.7) | 4 ( 66.7) | 1(16.7) | 0 | 0 | 0 | 0 | 6(100.0) |
| Overall (N=22) | n (%) | 0 | 4 ( 18.2) | 5( 22.7) | 1( 4.5) | 0 | 0 | 0 | 1( 4.5) | 11(50.0) |
| | n(%) | 1 | 0 | 8 ( 36.4) | 1(4.5) | 0 | 0 | 0 | 2( 9.1) | 11( 50.0) |
| | n (%) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n (%) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| | n(%) | Overall | 4 ( 18.2) | 13( 59.1) | 2( 9.1) | 0 | 0 | 0 | 3 ( 13.6) | 22(100.0) |


Repeat Table 14.3.10.1.1 for

Table 14.3.10.1.2 Shift of ECOG Performance Status from Baseline to Worst Post-Baseline Score for Part B (Safety Population)

Table 14.3.10.1.3 Shift of ECOG Performance Status from Baseline to Worst Post-Baseline Score for Part C (Safety Population)

Table 14.3.10.1.4 Shift of ECOG Performance Status from Baseline to Worst Post-Baseline Score for Part D (Safety Population)

TESARO Inc.

Table 14.3.10.2.1 Notable ECG Values for Part A (Safety Population)

| Visit | Parameter | Statistics | Part A-200<br>(N=XX) | Part A-300<br>(N=XX) | Overall (N=XX) |
|---|---|---|---|---|---|
| Cycle 1 Day 1 | Number of Patients | n | XX | xx | |
| | QTcF increase from baseline | | | | |
| | >30 ms | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | >60 ms | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | QTcF | | | | |
| | > 450 ms | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 480 ms | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | > 500 ms | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | HR HR $\leq 50$ bpm and decrease from baseline $\geq 20$ | | | | |
| | bpm $HR \ge 120 \text{ bpm and increase from baseline} \ge 20$ | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | bpm | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | PR | | | | |
| | $PR \geq 220 \text{ ms}$ and increase from baseline $\geq 20 \text{ ms}$ | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | QRS $\geq$ 120 ms | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Cycle 2 Day 1 | Number of Patients | n | XX | xx | |
| | QTcF increase from baseline | | | | |
| | >30 ms | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Percentage is calculated using the number of patients at visit as denominator

Source: Listing 16.2.12.2 Listing 16.2.12.3

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

## Repeat for

Table 14.3.10.2.2 Notable ECG Values for Part B (Safety Population)

Table 14.3.10.2.3 Notable ECG Values for Part C (Safety Population)

Table 14.3.10.2.4 Notable ECG Values for Part D (Safety Population)
Listing 16.2.1.1
Patient Enrollment (All Patients Population)

| | | | | Informed | Drug | Date of |
|---|---|---|---|---|---|---|
| Part | Patient ID | AAP | SP | Consent Date | Received | First Dose |
| Not Dosed | PPD | Y | N | PPD | | |
| | | Y | N | | | |
| Part A-200 | | Y | Y | | TSR-042/Niraparib | PPD |
| | | Y | Y | | TSR-042/Niraparib | |
| | | Y | Y | | TSR-042/Niraparib | |
| | | Y | Y | | TSR-042/Niraparib | |
| | | Y | Y | | TSR-042/Niraparib | |

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment


Listing 16.2.1.2.1 Discontinuation of Treatment Niraparib (Safety Population)

| Part | Patient<br>ID | Date of Discontinuation | First Dose<br>Date | Last Dose<br>Date | Number of Days<br>on Treatment [1] | Discontinuation<br>Reasons | Other<br>Reasons |
|---|---|---|---|---|---|---|---|
| 1 411 | ID | Discontinuation | DDMMY | DDMMY | on Treatment [1] | Reasons | ICCasons |
| Part A -200 | | DDMMYYYY | YYY | YYY | | | |
| Part A-300 | | | | | | | |
| Part C-200 | | | | | | | |
| Part C-300 | | | | | | | |

<sup>[1]</sup> Days on treatment = Last dose date - first dose date + 1

PROGRAM NAME: DATE: DDMMYYYY

Repeat using proper treatment and study drug for

Listing 16.2.1.2.2 Discontinuation of Treatment TSR-042 (Safety Population)

Listing 16.2.1.2.3 Discontinuation of Treatment Bevacizumab (Safety Population)

Listing 16.2.1.2.4 Discontinuation of Carboplatin-Paclitaxel (Safety Population)

Listing 16.2.1.2.5 Discontinuation of Treatment TSR-022 (Safety Population)

Listing 16.2.1.2.6 Discontinuation of Treatment Carboplatin (Safety Population)

Listing 16.2.1.2.7 Discontinuation of Treatment Pemetrexed (Safety Population)

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Listing 16.2.1.3
Discontinuation from Study (Safety Population)

| Part | Patient ID | Discontinuation<br>Date | Reasons for Discontinuation | Other Reasons for Discontinuation | Death<br>Date | Cause of Death | Other Death<br>Cause | Autopsy<br>performed |
|---|---|---|---|---|---|---|---|---|
| Part A-200 | | DDMMYYYY | DDMMYYYY | | | | | Y/N |
| Part A-300 | | | | | | | | |
| Part B | | | | | | | | |
| Part C-200 | | | | | | | | |
| Part C-300 | | | | | | | | |
| Part D | | | | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Listing 16.2.2
Protocol Deviation by Category and Severity (All Patients Population)

| Part | Patient ID | Date of Protocol<br>Deviation | Protocol Deviation<br>Category | Protocol Deviation<br>Severity | Description of<br>Protocol Deviation |
|---|---|---|---|---|---|
| Part A-200 | | DDMMYYYY | | | |
| Part A-300 | | | | | |
| Part B | | | | | |
| Part C-200 | | | | | |
| Part C-300 | | | | | |
| Part D | | | | | |
| ••• | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

TESARO Inc.

Listing 16.2.3
Patients Excluded Due to Eligibility (All Patients Population)

| | | | | | | Failed | d Criteria |
|---|---|---|---|---|---|---|---|
| Patient ID | SAFFL | Initial Protocol<br>Version | Current<br>Protocol<br>Version | Visit Date | Meet all<br>Eligibility<br>Criteria? | Criterion Type | Criterion Number |
| • | | | | DDMMYYYY | Y | | |
| | | | | DDMMYYYY | N | Exclusion | EXCL 5 |
| | | | | <br>DDMMYYYY | N | Inclusion | INCL 1 |
| | | | | ••• | | | |
| | | | | ••• | | | |

PROGRAM NAME: DATE: DDMMYYYY

## Listing 16.2.4.1 Demographics (Safety Population)

| | D : ID | Age | pd 11 | D. | |
|---|---|---|---|---|---|
| Part | Patient ID | (Years) S | Sex Ethnicity | Race | Specify Other Race |
| Part A-200 | | | | | |
| Part A-300 | | | | | |
| Part B | | | | | |
| Part C-200 | | | | | |
| Part C-300 | | | | | |
| Part D | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

# Listing 16.2.4.2 Medical History (Safety Population)

| Part | Patient ID | Condition | System Organ<br>Class/Preferred Term | Start date (Rel<br>Days [1]) | Condition Ongoing at Study Entry | Stop date |
|---|---|---|---|---|---|---|
| | | | | DDMMYYYY | | |
| Part A-200 | | | | (days) | Y/N | DDMMYYYY |
| Part A-300 | | | | Unknown | | Unknown |
| Part B | | | | | | |
| Part C-200 | | | | | | |
| Part C-300 | | | | | | |
| Part D | | | | | | |
| ••• | | | | | | |

<sup>[1]</sup> Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date)

## PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

# Listing 16.2.4.3 Surgical History (Safety Population)

| Part | Patient ID | Major Surgeries Reported | Surgery | Surgery Date (Rel Days [1]) | Cancer Related |
|---|---|---|---|---|---|
| Part A-200 | | Y/N | | DDMMYYYY (days) | Y/N |
| Part A-300 | | | | | |
| Part B | | | | | |
| Part C-200 | | | | | |
| Part C-300 | | | | | |
| Part D | | | | | |
| ••• | | | | | |

<sup>[1]</sup> Rel Days are calculated as surgery date minus first dose date (plus 1 day if surgery date is on or after first dose date)

## PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment


# Listing 16.2.4.4 Previous Radiotherapy (Safety Population)

| Part | Patient ID | Radiotherapy Prior to<br>Informed Consent | Site or Region | Start Date (Rel Days [1]) | End Date | Total<br>Grays |
|---|---|---|---|---|---|---|
| Part A-200 | | Y/N | | DDMMYYYY (days) | DDMMYYYY | |
| Part A-300 | | 1/11 | | DDIMIT I I I (days) | 22 | |
| Part B | | | | | | |
| Part C-200 | | | | | | |
| Part C-300 | | | | | | |
| Part D | | | | | | |

<sup>[1]</sup> Rel Days = first dose date - start date

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

# Listing 16.2.4.5 Concomitant Radiotherapy (Safety Population)

| Part | Patient ID | Was the site a target or non-target lesion? | Lesion Number | Start Date (Rel<br>Days [1]) | End Date | Total<br>Grays |
|---|---|---|---|---|---|---|
| Part A-200 | | Y/N | | DDMMYYYY<br>(days) | DDMMY<br>YYY | |
| Part A-300 | | | | | | |
| Part B | | | | | | |
| Part C-200 | | | | | | |
| Part C-300 | | | | | | |
| Part D | | | | | | |
| ••• | | | | | | |

[1] Rel Days are calculated as start date minus first dose date (plus 1 day if radiotherapy start date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.4.6
Prior Transfusions and Growth Factors (Safety Population)

| Part | Patient<br>ID | Received Transfusions or Growth Factors | Type of Administration | Specify<br>Other | Total<br>Units | Start Date (Rel<br>Days [1]) | Stop Date |
|---|---|---|---|---|---|---|---|
| 1 411 | ID. | or Growth ructors | 1 Idiiiiiisti dii oli | Other | Cinto | DDMMYYYY | Stop Bute |
| Part A-200 | | Y/N | | | | (days) | DDMMYYYY |
| Part A-300 | | | | | | | |
| Part B | | | | | | | |
| Part C-200 | | | | | | | |
| Part C-300 | | | | | | | |
| Part D | | | | | | | |

[1] Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date).

# PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

## Listing 16.2.4.7 Concomitant Transfusion (Safety Population)

| Part | Patient<br>ID | Transfusions within 14 days prior to first dose and/or during the study | Type of Administration | Specify<br>Other | Total<br>Units | Start Date (Rel<br>Days [1]) | End Date |
|---|---|---|---|---|---|---|---|
| Part A-200<br>Part A-300<br>Part B<br>Part C-200<br>Part C-300<br>Part D | | Y/N | | | | DDMMYYYY<br>(days) | DDMM<br>YYYY |

[1] Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date).

# PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.4.8
Concomitant Growth Factors (Safety Population)

| Part | Patient<br>ID | Growth factor given within 14 days prior to first dose and/or during the study | Type of<br>Administration | Specify<br>Other | Dose | Units | Start Date<br>(Rel Days [1]) | End Date |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | DDMMYYY | DDMM |
| Part A-200 | | Y/N | | | | | Y (days) | YYYY |
| Part A-300 | | | | | | | | |
| Part B | | | | | | | | |
| Part C-200 | | | | | | | | |
| Part C-300 | | | | | | | | |
| Part D | | | | | | | | |

<sup>[1]</sup> Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date).

# PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Listing 16.2.4.9
Prior Blood Disorders (Safety Population)

| | | Prior History of Thrombocytopenia, | | CTCAE | Start Date (Rel | |
|---|---|---|---|---|---|---|
| Part | Patient ID | Leukopenia, Anemia or Neutropenia | Event | Grade | Days [1]) | End Date |
| | | | | | DDMMYYYY | DDMMYYY |
| Part A-200 | | Y/N | | | (days) | Y |
| Part A-300 | | | | | | |
| Part B | | | | | | |
| Part C-200 | | | | | | |
| Part C-300 | | | | | | |
| Part D | | | | | | |

[1] Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.4.10
Prior Anticancer Treatment for Primary Cancer (Safety Population)

| Part | Patient<br>ID | Regimen<br>Number | Agent<br>Name | Specify<br>Other | Start<br>Date | End<br>Date | Best<br>Response | SDate of Progression or Recurrence | Reason for Discontinuation | Specify if<br>Toxicity or Other |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | DDMM | | | | | |
| Part A-200 | | | | | YYYY | | | | | |
| Part A-300 | | | | | | | | | | |
| Part B | | | | | | | | | | |
| Part C-200 | | | | | | | | | | |
| Part C-300 | | | | | | | | | | |
| Part D | | | | | | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

# Listing 16.2.4.11 Primary Cancer History (Safety Population)

| Part | Patient<br>ID | Date of First<br>Diagnosis (Rel<br>Days [1]) | Tumor Site at<br>First Diagnosis | Cancer Stage<br>First Diagnosis | Tumor Site Most<br>Recent Diagnosis | Cancer Stage<br>Most Recent<br>Diagnosis |
|---|---|---|---|---|---|---|
| Part A-200 | | DDMMYYYY | | | | |
| Part A-300 | | | | | | |
| Part B | | | | | | |
| Part C-200 | | | | | | |
| Part C-300 | | | | | | |
| Part D | | | | | | |

[1] Rel Days are calculated as first diagnosis date minus first dose date (plus 1 day if first diagnosis date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Listing 16.2.4.12
HBsAg and HCV Testing at Baseline (Safety Population)

| | | | Test Date (Rel | | |
|------------|------------|-----------|----------------|-------|-----|
| Part | Patient ID | Test Name | Days [1]) | HBsAg | HCV |
| | | | DDMMYYYY | | |
| Part A-200 | | | (days) | | |
| Part A-300 | | | | | |
| Part B | | | | | |
| Part C-200 | | | | | |
| Part C-300 | | | | | |
| Part D | | | | | |

[1] Rel Days are calculated as test date minus first dose date (plus 1 day if test date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

# Listing 16.2.5.1 Prior and Concomitant Medication/Therapy (Safety Population)

| Part | Patient<br>ID | ATC/Generic<br>Name/Verbatim<br>Name | Non-<br>Anticancer | Indication | Dose per administration | Dose<br>Unit | Frequency | Route of<br>Administration | Start Date (Rel<br>Days [1]) | End<br>Date | Ongoing |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Part A-200 | | | Y/N | | | | | | | | Y/N |
| Part A-300 | | | | | | | | | | | |
| Part B | | | | | | | | | | | |
| Part C-200 | | | | | | | | | | | |

<sup>[1]</sup> Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

## Listing 16.2.5.2 Concomitant Procedures (Safety Population)

| | Patient | Procedure | Start Date (Rel | | | | |
|---|---|---|---|---|---|---|---|
| Part | ID | Performed | Days [1]) | Procedure | Results/Findings | AE/SAE | Indication |
| Part A-200 | | Y/N | | | | | |
| Part A-300 | | | | | | | |
| Part B | | | | | | | |
| Part C-200 | | | | | | | |
| Part C-300 | | | | | | | |
| Part D | | | | | | | |

<sup>[1]</sup> Rel Days are calculated as procedure date minus first dose date (plus 1 day if procedure date is on or after first dose date)

## PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.5.3 Niraparib First Dose (Safety Population)

| Part | Patient<br>ID | Taken at<br>C1D1 | Dose date | Time | Kit<br>Number<br>Assigned | No. of Pills dispensed | Dose<br>prescribed<br>(mg) | Full Dose<br>Consumed | Dose<br>Consumed<br>(mg) | Reason<br>Not<br>Consumed |
|---|---|---|---|---|---|---|---|---|---|---|
| Part A-200 | | Y/N | DDMMYYYY | HH:MM:SS | | | | | | |
| Part A-300 | | | | | | | | | | |
| Part C-200 | | | | | | | | | | |
| Part C-300 | | | | | | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Listing 16.2.5.4 Niraparib Dose Modification (Safety Population)

| Part | Patient ID | Dose Modified or<br>Missed | Start date (Rel Days [1]) | Stop<br>date | No. of Pills<br>Not Taken | Action<br>Taken | Dose | Unit | Reason for<br>Modification | Other Reason for Modification |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | DDMMYYYY | | | | | | | |
| A-200 | | Y/N | (days) | | | | | | | |
| A-300 | | | | | | | | | | |
| C-200 | | | | | | | | | | |
| C-300 | | | | | | | | | | |

[1] Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Listing 16.2.5.5 Niraparib Administration (Safety Population)

| | | | | | | | At this | Cycle | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Nirapar<br>ib | | | Niraparib | | | Dose | Date | | Time<br>e Dose | Full | Dose | Reason |
| Part | Patient<br>ID | Wieit | Kit<br>Return | Kit No<br>Returned | . Pills | Dose | Kit No<br>Disp. | . Pills Disp. | | Administer<br>(Rel Days | | Adminis<br>tered | Dose<br>Consumed | | d Modific<br>ation |
| | 10 | VISIC | recuin | Necariica | rcmain | 01.0011 | DIOP. | DISP. | ea (mg) | (NCI Days | [±]/ | CCICA | CONSUMCA | (mg) | 401011 |
| A-200 | PPD | C2D1 | Y | P1000041 | 30 | Y | P100004 | 3 72 | 200 | PPD | (22) | 10:26 | Y | 200 | |
| A-200 | | C3D1 | Y | P1000043 | 32 | Y | P100004 | 4 72 | 200 | | (43) | 13:05 | Y | 200 | |
| A-200 | | C4D1 | Y | P1000044 | 30 | Y | P100006 | 1 72 | 200 | | (64) | 11:53 | Y | 200 | |
| A-200 | | C5D1 | Y | P1000061 | 30 | Y | P100006 | 2 72 | 200 | | (85) | 12:37 | Y | 200 | |
| A-200 | | C6D1 | Y | P1000062 | 32 | Y | P100006 | 3 72 | 200 | | (107) | 11:26 | Y | 200 | |

[1] Rel Days are calculated as administration date minus first dose date (plus 1 day if administration date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

# For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment


Listing 16.2.5.6
TSR-042 Administration (Safety Population)

| | | | | | Delayed | | | | Infusion | | Restarted | | Total | Total<br>Volume | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Infusion | Intended | More Than | Date of | | | Interrupte | Interrupted | Infusion | End | Dose | Admini | Volume |
| | | | Given/ | Total | 3 Days/ | Infusion | | Start | d/ | Infusion | Completed/ | Date | Infused | stered | Left |
| Part | Patient ID | Visit | Reason | Dose (mg) | Reason | (Rel Days [ | 1]) | Time | Reason | Restarted | Reason | Time | (mg) | (mL) | (mL) |
| A-200 | PPD | C1D1 | Y | 500 | N | PPD | (1) | 10:55 | N | | | 11:25 | 500 | 100 | 0 |
| A-200 | | C2D1 | Y | 500 | N | | (22) | 09:55 | N | | | 10:25 | 500 | 100 | 0 |
| A-200 | | C3D1 | Y | 500 | N | | (43) | 12:31 | N | | | 13:02 | 500 | 100 | 0 |
| A-200 | | C4D1 | Y | 500 | N | | (64) | 11:20 | N | | | 11:52 | 500 | 100 | 0 |
| A-200 | | C5D1 | Y | 1000 | N | | (85) | 11:44 | N | | | 12:18 | 1000 | 100 | 0 |

[1] Rel Days are calculated as infusion date minus first dose date (plus 1 day if infusion date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Listing 16.2.5.7
Carboplatin Administration (Safety Population)

| | | | | | Delayed | | | | | | | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Intended | More | Date | of | | | Restarted | End | Total | Volume | Total |
| | | | Infusion | Dose | Than | Infus | ion | Infusion | Interrupted | lInfusion | Time | Dose | to | be Volume |
| | Patient | | Given/ | Level | 3 Days | / (Rel | Days Start | Interrupted/ | 'Infusion | Completed/ | of | Infused | d Administer | ed Left |
| Part | ID | Visit | Reason | (AUC) | Reason | [1]) | Time | Reason | Restarted | Reason | Infusion | (mg) | (mL) | (mL) |
| В | PPD | C1D1 | Y | 413 | N | PPD | 09:55 | N | | | 10:55 | 413 | 541 | 0 |
| | | | | | | (1) | | | | | | | | |
| В | | C2D1 | Y | 403 | N | PPD | 11:15 | N | | | 12:15 | 403 | 540 | 0 |
| | | | | | | (22) | | | | | | | | |
| В | | C3D1 | Y | 403 | N | PPD | 12:15 | N | | | 13:15 | 403 | 540 | 0 |
| | | | | | | (43) | | | | | | | | |
| В | | C4D1 | Y | 403 | Y/OTHER- | PPD | 14:46 | N | | | 15:46 | 403 | 540 | 0 |
| | | | | | SCHEDULING | G (75) | | | | | | | | |
| | | | | | CONFLICT | | | | | | | | | |

[1] Rel Days are calculated as infusion date minus first dose date (plus 1 day if infusion date is on or after first dose date)

# PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

 $Part\ F-300:\ TSR-042,\ TSR-022\ (300mg)\ and\ carboplatin-pemetrexed\ combination\ treatment$ 

Listing 16.2.5.8
Paclitaxel Administration (Safety Population)

| | | | | | | | Date of | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Body | Intende | Delayed | Infusio | | | | | Restarted | | | Total | Total |
| | | | Infusio | Surfac | d | More | n | | | Infusion | Interrupte | Infusion | | Total | Volume | Volum |
| | | | n | е | Total | Than | (Rel | Star | Infusion | Interrupted | d | Completed | | Dose | Administere | е |
| Par | Patien | Visi | Given/ | Area | Dose | 3 Days/ | / Days | t | Complete | / | Infusion | / | End | Infuse | d | Left |
| - | t ID | t | Reason | (m2) | (mg) | Reason | [1]) | Time | d | Reason | Restarted | Reason | Time | d (mg) | (mL) | (mL) |
| 3 | PPD | C1D1 | Y | 2.09 | 364 | N | PPD | 11:0 | Y | N | | | 14:0 | 364 | 560 | 0 |
| | | | | | | | (1) | 0 | | | | | 0 | | | |
| 3 | | C2D1 | Y | 2.06 | 360 | N | (22) | 12:3<br>0 | Y | N | | | 15:3<br>0 | 360 | 560 | 0 |
| | | C3D1 | Y | 2.04 | 360 | N | | 13:5<br>0 | Y | N | | | 16:5<br>0 | 360 | 560 | 0 |
| i | | C4D1 | Y | 2.07 | 355 | Y/OTHER-<br>SCHEDULIN<br>G<br>CONFLICT | PPD | 11:4<br>5 | Y | N | | | 14:4<br>5 | 355 | 559 | 0 |

. . .

[1] Rel Days are calculated as infusion date minus first dose date (plus 1 day if infusion date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

# Repeat for

Listing 16.2.5.9 Pemetrexed Administration (Safety Population)

For programmer: add following footnotes

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Listing 16.2.5.11
Bevacizumab Administration (Safety Population)

| Part | Patient ID | Visit. | Infusion<br>Given<br>(15mg/kg)/<br>Reason | Total | d Delayed<br>More Tha<br>3 Days<br>Reason | Date<br>In Infusions/<br>Infusions/<br>Info | | Infusion Interrupted | Interrupted<br>dInfusion<br>Restarted | Completed/ | End<br>Time | Total<br>Dose<br>Infused | Total Volume to be Admini stered (mL) | Total<br>Volume |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | C1D1 | Y | 1274 | N | PPD | 10:28 | | | | 12:03 | , ,, | | 0 |
| | | | | | | (1) | | | | | | | | |
| C-200 | | C2D1 | Y | 1203 | N | PPD | 10:40 | N | | | 11:34 | 1203 | 100 | 0 |
| ~ 000 | | 0251 | | 1170 | | (22)<br><b>PPD</b> | 11 10 | | | | 11 00 | 1170 | 100 | 0 |
| C-200 | | C3D1 | Y | 1172 | N | (43) | 11:10 | N | | | 11:38 | 1172 | 100 | 0 |
| | | | | | | (43) | | | | | | | | |

[1] Rel Days are calculated as infusion date minus first dose date (plus 1 day if infusion date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Listing 16.2.5.12
TSR-022 Administration (Safety Population)

| | | | | | Delayed | dDate o | f | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Intende | ed More | Infusio | n | | | | | Total | Total | Total |
| | | | Infusio | n Total | Than | (Rel | | | Interrupted | d Restarted | End | Dose | Volume | Volume |
| | | | Given/ | Dose | 3 Days/ | / Days | Start | Infusion | Infusion | Infusion | Date | Infuse | d Administer | ed Left |
| Part | Patient ID | Visit | Reason | (mg) | Reason | [1]) | Time | Interrupted/Reason | n Restarted | Completed/Reason | Time | (mg) | (mL) | (mL) |
| F-900 | PPD | C1D1 | Y | 900 | N | PPD | 10:14 | ł N | | | 10:44 | 900 | 250 | 0 |
| F-900 | | C2D1 | Y | 900 | N | (1) | 11:23 | 3 N | | | 11:53 | 900 | 250 | 0 |
| | | | | | | (22)<br><b>PPD</b> | | | | | | | | |
| F-900 | | C3D1 | Y | 900 | N | (42) | 11:31 | L N | | | 12:01 | 900 | 250 | 0 |
| F-900 | | C4D1 | Y | 900 | N | PPD (64) | 11:0 | 7 N | | | 11:37 | 900 | 250 | 0 |
| F-900 | | C5D1 | Y | 900 | N | PPD (85) | 11:38 | N N | | | 12:08 | 684 | 250 | 60 |

[1] Rel Days are calculated as infusion date minus first dose date (plus 1 day if infusion date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

| Part | Patient ID | Did the subject receive at least 5 doses (350 to 1,000 μg oral) of folic acid during the week preceding the first dose of Pemetrexed? | Did the subject receive the dose (1,000 µg intramuscular injection) of Vitamin B-12 during the week preceding the first dose of Pemetrexed? |
|---|---|---|---|
| Part E | | | |
| Part F-300 | | | |
| Part F-900 | | | |
| PROGRAM | I NAME: | | |

PROGRAM NAME: DATE: DDMMYYYY

# Listing 16.2.5.14 Pemetrexed Supplemental Medications (Safety Population)

| Part | Patient ID | Name of Medication | Indication | Dose per administration | Frequency | Route of Administration | Start Date | Ongoing? | End Date |
|---|---|---|---|---|---|---|---|---|---|
| Part E | | | | | Specify other | | unknonw | Y/N | |
| Part F-300<br>Part F-900 | | | | | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment


Listing 16.2.6.1
Tumor Target Lesion Assessment (Safety Population)

| Part | Patient ID | Visit | Any Target<br>Lesions | Lesion<br>Number | Site | Region for<br>Lymph Node | Date of<br>Scan/Assessment (Rel<br>Days [1]) | Method | Lesion<br>Measurement | Lesion<br>Status |
|---|---|---|---|---|---|---|---|---|---|---|
| Part A-200 | | | Y/N | | Specify if other Site | Specify<br>Other | DDMMYYYY (days) | | | |
| Part A-300 | | | 1/11 | | other site | o in cr | DDMM11111 (days) | | | |
| Part B | | | | | | | Not Done | | | |
| Part C-200 | | | | | | | | | | |
| Part C-300 | | | | | | | | | | |
| Part D | | | | | | | | | | |

<sup>[1]</sup> Rel Days are calculated as assessment date minus first dose date (plus 1 day if assessment date is on or after first dose date)

### PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.6.2
Tumor Non-Target Lesion Assessment (Safety Population)

| Part | Patient<br>ID | Visit | Any Non-<br>Target Lesions | Lesion<br>Number | Site | Region for Lymph<br>Node-Other | Date of Scan/Assessment (Rel Days [1]) | Method | Lesion<br>Status |
|---|---|---|---|---|---|---|---|---|---|
| Part A-200<br>Part A-300<br>Part B | | | Y/N | | Specify<br>region for<br>lymph node | | DDMMYYYY (days) | | |
| ••• | | | | | | | | | |

[1] Rel Days are calculated as assessment date minus first dose date (plus 1 day if assessment date is on or after first dose date).

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Listing 16.2.6.3 New Lesion Assessment (Safety Population)

| Part | Patient<br>ID | Visit | Any New<br>Lesions | Lesion<br>Number | Site | Region for Lymph<br>Node-Other | Evaluation Date (Rel Days [1]) | Method | Status |
|---|---|---|---|---|---|---|---|---|---|
| Part A-200<br>Part A-300 | | | Y/N | | Specify region for lymph node | | DDMMYYYY (days) | | |
| Part B | | | | | | | | | |

...

## PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

<sup>[1]</sup> Rel Days are calculated as assessment date minus first dose date (plus 1 day if assessment date is on or after first dose date).

Listing 16.2.6.4
Tumor Response Assessments by RECIST v1.1 (Safety Population)

| | | | | | | | of | Diameters<br>all<br>sions (mm) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Part<br>Patient ID | Visit | Date of<br>Radiological<br>Scan/Asmnt.<br>(Rel Days [1]) | | Sum of Diameters Target of all Lesion(s) target Respon- lesions se (mm) | | New<br>Lesion | Change % Chang<br>from from<br>baseline baselin<br>n (mm) (%) | | Change from smallest sum on study of all measurable lesions (mm) | % Change<br>from<br>Smallest<br>(%) | Non-Target<br>Lesion(s)<br>Response | Overall<br>Respon-<br>se |
| Part A-200 S | SCREENING | PPD | (-6) | | 43.0 | N | | | | | | |
| | | | (81) | CR | 0.0 | N | -43.0 | -100.0 | 0.0 | | Non-CR/Non-PD | PR |
| | | | (166) | CR | 0.0 | N | -43.0 | -100.0 | 0.0 | | Non-CR/Non-PD | PR |
| | | | (250) | | 0.0 | N | -43.0 | -100.0 | 0.0 | | Non-CR/Non-PD | PR |
| | | | (337) | CR | 0.0 | Y | -43.0 | -100.0 | 0.0 | | UNEQUIVOCAL<br>PD | PD |
| Part A-200 S | SCREENING | | (-11) | | 46.0 | N | | | | | | |
| | | | (15) | SD | 45.0 | N | -1.0 | -2.2 | 0.0 | 0.0 | Not<br>Applicable | SD |

<sup>[1]</sup> Rel Days are calculated as assessment date minus first dose date (plus 1 day if assessment date is on or after first dose date).

## PROGRAM NAME: DATE: DDMMYYYY

For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment
TESARO Inc.


Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment

Statistical Analysis Plan

Listing 16.2.6.5.2

Confirmed Best Overall Response and Duration of Response (RECIST v1.1) and Survival (Safety Population)

| Part | Patient<br>ID | Best Overall<br>Response | Date of First<br>CR/PR (Rel Days<br>[1]) | Duration of<br>Response | Disease Progression | Date of PD<br>(Rel Days [1]) | Death | Date of Death<br>(Rel Days [1]) | Date of Last<br>Contact (Rel<br>Days [1]) |
|---|---|---|---|---|---|---|---|---|---|
| Part A- | | | YYYY-MM-DD | | | YYYY-MM- | | YYYY-MM- | YYYY-MM- |
| 200 | | CR | (days) | | Yes/No | DD (days) | Yes/No | DD (days) | DD (days) |
| Part A-<br>300 | | PR | | | | | | | |
| Part B | | SD | | | | | | | |
| Part C-200 | | PD | | | | | | | |
| Part C-300 | | NE | | | | | | | |
| Part D | | | | | | | | | |

[1] Relative to the date of first dose

PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

TESARO Inc. Statistical Analysis Plan
Dated:18SEP2020

## Listing 16.2.6.16 Survival Assessment (Safety Population)

| Part | Patient ID | First Dose<br>Date | Current<br>Patient Status | Date of Contact (Rel<br>Days [1]) | New Malignancy<br>Reported | Diagnosis of New<br>Malignancy |
|---|---|---|---|---|---|---|
| | | DDMMY | | DDMMYYYY | | |
| Part A-200 | | YYY | | (days) | Y/N | |
| | | | | | Not Reported | |
| Part A-300 | | | | | /Unknown | |
| Part B | | | | | | |
| Part C-200 | | | | | | |
| Part C-300 | | | | | | |
| Part D | | | | | | |

<sup>[1]</sup> Rel Days are calculated as contact date minus first dose date (plus 1 day if contact date is on or after first dose date).

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.7.1

Adverse Events for Part A (Safety Population)

| | | System Organ Class/ | | | | | SAE | | Action Taken | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient | Preferred | Start Date/Time | | CTCAE | | Due to | Relationship to | [3] [4] | Trt. or | AESI/ |
| Part | ID | Term/Verbatim Term | (Rel Days [1]) | Stop Date/Time | Grade | TEAE/SAE | [2] | Drug | /Outcome [5] | Medication given | DLT |
| | | | DDMMYYY | | | | | | | | |
| | | | YTHH:MM:S | | | | | | Other Action | | |
| Part A-200 | | | S (days) | | | Y/N | | Niraparib | Taken | Y/N | Y/N |
| Part A-300 | | | | ongoing | | | | TSR-042 | | | |

<sup>[1]</sup> Rel Days are calculated as AE date minus first dose date (plus 1 day if AE date is on or after first dose date).

#### PROGRAM NAME: DATE: DDMMYYYY

#### Repeat for

Listing 16.2.7.2 Adverse Events for Part B (Safety Population)

Listing 16.2.7.3 Adverse Events for Part C (Safety Population)

Listing 16.2.7.4 Adverse Events for Part D (Safety Population)

Listing 16.2.7.5 Adverse Events for Part E (Safety Population)

Listing 16.2.7.6 Adverse Events for Part F (Safety Population)

<sup>[2] 1=</sup>Death, 2=Life Threatening, 3=Requires inpatient hospitalization or prolongation of existing hospitalization, 4=Persistent or Significant Disability or Incapacity,5=Congenital Anomaly or Birth Defect, 6=Other Medically Important Event

<sup>[3]</sup> N=Niraparib, T=TSR-042

<sup>[4] 1=</sup> Dose/Infusion Not Changed; 3= Dose Reduced; 4= Drug/Infusion Interrupted; 5= Infusion Delayed; 6= Drug Withdrawn; 7= Not Applicable;

<sup>[5] 2=</sup> Not Recovered/Not Resolved; 3= Recovered/Resolved; 4= Recovered/Resolved With Sequelae; 5= Recovering/Resolving; 6= Unknown;

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

TESARO Inc.

Statistical Analysis Plan

Dated:18SEP2020

Listing 16.2.8.1 Hematology Results (Safety Population)

| | Patient | | Date of Lab (Rel | | | | Change from | Normal | Out of | Clinically |
|---|---|---|---|---|---|---|---|---|---|---|
| Part | ID | Visit | Days [1]) | Parameter | Result | Unit | Baseline | Range | Range Flag | Significant |
| Part A-200 | | | DDMMYYYY (days) | | | | | | | |
| Part A-300 | | | | | | | | | | |
| art B | | | | | | | | | | |
| Part C-200 | | | | | | | | | | |
| Part C-300 | | | | | | | | | | |
| Part D | | | | | | | | | | |

[1] Rel Days are calculated as lab date minus first dose date (plus 1 day if lab date is on or after first dose date).

PROGRAM NAME: DATE: DDMMYYYY

### Repeat for

Listing 16.2.8.2 Chemistry Results (Safety Population)

Listing 16.2.8.3 Coagulation Results (Safety Population)

Listing 16.2.8.4 Serum tumor markers (Safety Population)

Listing 16.2.8.5 Thyroid Function Results (Safety Population)

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment


TESARO Inc. Statistical Analysis Plan
Dated:18SEP2020

# Listing 16.2.8.6 Pregnancy Test (Safety Population)

| Part | Patient ID | Visit | Test Performed | Test Date (Rel Days [1]) | Test Type | Test Result |
|---|---|---|---|---|---|---|
| Part A-200 | | | Y/N | DDMMMYYYY (days) | Serum | Positive |
| Part A-300 | | | | | Urine | Negative |
| Part B | | | | | | |
| Part C-200 | | | | | | |
| Part D | | | | | | |

[1] Rel Days are calculated as test date minus first dose date (plus 1 day if test date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

## Listing 16.2.8.7 Urinalysis Results (Safety Population)

| Part | Patient ID | Visit | Lab Date (Rel Days [1]) | Parameter | Result |
|---|---|---|---|---|---|
| Part A-200 | | | DDMMYYYY (days) | Glucose | |
| Part A-300 | | | | Ketones | |
| Part B | | | | | |
| Part C-200 | | | | | |
| Part D | | | | | |

<sup>[1]</sup> Rel Days are calculated as lab date minus first dose date (plus 1 day if lab date is on or after first dose date).

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

## Listing 16.2.9 Vital Signs (Safety Population)

| Part | Patient ID | Visit | Assessment Date (Rel Days [1]) | Height (cm) | Weight (kg) | Temperature (°C) | Pulse<br>(beats/min) | Systolic Blood<br>Pressure (mmHg) | Diastolic Blood<br>Pressure (mmHg) |
|---|---|---|---|---|---|---|---|---|---|
| Part A-200 | | | DDMMYYYY (days) | | | | | | |
| Part A-300 | | | | | | | | | |
| Part B | | | | | | | | | |
| Part C-200 | | | | | | | | | |
| Part D | | | | | | | | | |
| ••• | | | | | | | | | |

[1] Rel Days are calculated as assessment date minus first dose date (plus 1 day if assessment date is on or after first dose date).

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment

Part G: TSR-042 and carboplatin-nab-paclitaxel combination treatment

Part H-300: TSR-042, TSR-022 (300mg) and carboplatin-nab-paclitaxel combination treatment

Part H-900: TSR-042, TSR-022 (900mg) and carboplatin-nab-paclitaxel combination treatment

Part I-300: TSR-042, TSR-022 (300mg) and carboplatin-paclitaxe combination treatment

Listing 16.2.10 ECOG Performance Status (Safety Population)

| Part | Patient ID | Visit | ECOG Performance<br>Status Collected | Performance Date (Rel Days [1]) | Performance<br>Status |
|---|---|---|---|---|---|
| Part A-200 | | | Y/N | DDMMYYYY (days) | |
| Part A-300 | | | | | |
| Part B | | | | | |
| Part C-200 | | | | | |
| Part C-300 | | | | | |
| Part D | | | | | |

<sup>[1]</sup> Rel Days are calculated as ECOG performance date minus first dose date (plus 1 day if ECOG performance date is on or after first dose date)

## PROGRAM NAME: DATE: DDMMYYYY

#### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.11
Physical Examination Findings (Safety Population)

| Part | Patient ID | Visit | Date of Examination (Rel<br>Days [1]) | Body System<br>Examined | Examination<br>Result | Description of<br>Abnormal<br>Findings | Symptom Directed Physical Exam Performed |
|---|---|---|---|---|---|---|---|
| Part A-200 | | | DDMMYYYY (days) | | | | Y/N |
| Part A-300 | | | | | | | |
| Part B | | | | | | | |
| Part C-200 | | | | | | | |
| Part C-300 | | | | | | | |
| Part D | | | | | | | |

<sup>[1]</sup> Rel Days are calculated as exam date minus first dose date (plus 1 day if exam date is on or after first dose date)

## PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment  $\,$ 

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment

# Listing 16.2.12.1 ECG - Pre-Post Niraparib Dose (Safety Population)

| _ Part | Patient<br>ID | Visit | ECG<br>Performed | ECG Date and Time<br>(Rel Days [1]) | ECG Timepoint | ECG Test<br>(Unit) | ECG Result | ECG Interpretation |
|---|---|---|---|---|---|---|---|---|
| | | | | YYYY-MM-DDTHH:MM | | | | |
| Part A-200 | | | Y/N | (days) | | | | |
| Part A-300 | | | | | | | | |
| Part B | | | | | | | | |
| Part C-200 | | | | | | | | |
| Part C-300 | | | | | | | | |
| Part D | | | | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment Part F-900: TSR-042, TSR-022 (900mg) and carboplatin-pemetrexed combination treatment


Listing 16.2.12.2 ECG (Safety Population)

| Part | Patient<br>ID | Visit | ECG<br>Performed | ECG Date and Time<br>(Rel Days [1]) | Position of the Subject | ECG Test<br>(Unit) | ECG Result | ECG Interpretation |
|---|---|---|---|---|---|---|---|---|
| | | | | YYYY-MM-DDTHH:MM | • | | | • |
| Part A-200 | | | Y/N | (days) | | | | |
| Part A-300 | | | | | | | | |
| Part B | | | | | | | | |
| Part C-200 | | | | | | | | |
| Part C-300 | | | | | | | | |
| Part D | | | | | | | | |

PROGRAM NAME: DATE: DDMMYYYY

### Repeat for

Listing 16.2.12.3 Notable ECG (Safety Population)

## For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment Part A-300: TSR-042 and niraparib (300mg) combination treatment Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Listing 16.2.13
Subsequent Anticancer Treatment for Primary Cancer (Safety Population)

| | | Any Subsequent | | | | | | | Date of | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Patient | Anticancer | Regimen | | Reason for | Start Date (Rel | | Best | Progression or | Reason for |
| Part | ID | Therapy | Number | Agent Name | administration | Days [1]) | End Date | Response | Recurrence | discontinuation |
| | | | | Specify | | | | | | Specify if |
| | | | | Other Agent | | DDMMYYYY | DDMMY | | | Toxicity or |
| Part A-200 | | Y/N | | Name | Other/Specify | Y (days) | YYYY | | | Other |
| Part A-300 | | | | | | | | | | |
| Part B | | | | | | | Ongoing | | | |
| Part C-200 | | | | | | | | | | |
| Part C-300 | | | | | | | | | | |
| Part D | | | | | | | | | | |

[1] Rel Days are calculated as start date minus first dose date (plus 1 day if start date is on or after first dose date)

PROGRAM NAME: DATE: DDMMYYYY

### For programmer: add following footnotes

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

 $Part\ D:\ TSR-042,\ carboplatin-paclitaxel\ and\ bevacizum ab\ combination\ treatment$ 

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

 $Part\ F-300:\ TSR-042,\ TSR-022\ (300mg)\ and\ carboplatin-pemetrexed\ combination\ treatment$ 

Listing 16.2.14
Listing of COVID19 Assessments and Symptom Assessments for Subjects with COVID19 Adverse Events

Site Id.: PPD

| Treatment | Unique Subject<br>Id./<br>Subject Id. | Adverse<br>Event | AE<br>Start<br>Date | COVID-19<br>Case<br>Diagnosis<br>[1] | COVID-19 Test<br>Performed/<br>Test Date/<br>Results | Assessments and<br>Symptom Assessments | Result |
|---|---|---|---|---|---|---|---|
| Part A-200 | PPD | Coronavirus<br>infection | PPD | Suspected | Y/<br>PPD /<br>Indeterminate | Travel to Location with Community Transmission [2] | N |
| | | | | | | Visited Health Care<br>Facility [2]<br>Contact with COVID-<br>19<br>Confirmed/Probable | N<br>Unknown |
| | | | | | | Case [2] Medication Taken to Treat COVID-19 Fever | Y<br>Y |
| | | | | | | Cough | Y |
| | | | | | | Shortness of Breath | Y |
| | | | | | | Sore Throat | N |
| | | | | | | Loss of Appetite | N |
| | | | | | | Nausea | N |
| | | | | | | Vomiting | N |
| | | | | | | Diarrhea | N |

TESARO Inc.


# Statistical Analysis Plan **Dated:18SEP2020**

| Abdominal Pain | N |
|----------------|---------|
| Fatigue | N |
| Loss of Smell | N |
| Loss of Taste | N |
| Asymptomatic | N |
| Home | Unknown |

Ouarantined/Isolated

PROGRAM NAME: DATE: DDMMYYYY

## For programmer: add following footnotes as applicable

Part A-200: TSR-042 and niraparib (200mg) combination treatment

Part A-300: TSR-042 and niraparib (300mg) combination treatment

Part B: TSR-042 and carboplatin-paclitaxel combination treatment

Part C-200: TSR-042, niraparib (200mg) and bevacizumab combination treatment

Part C-300: TSR-042, niraparib (300mg) and bevacizumab combination treatment

Part D: TSR-042, carboplatin-paclitaxel and bevacizumab combination treatment

Part E: TSR-042 and carboplatin-pemetrexed combination treatment

Part F-300: TSR-042, TSR-022 (300mg) and carboplatin-pemetrexed combination treatment